#### CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

**DMID Protocol: 22-0004** 

# **Study Title:**

Phase 2 Clinical Trial to Optimize Immune Coverage of SARS-CoV-2 Existing and Emerging Variants

COVID-19 VAriant Immunologic Landscape Trial (COVAIL)

NCT05289037

Version 1.0

**DATE: 100CT2023** 

RESTRICTED

# **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 22-0004 |
|---|---|
| <b>Development Phase:</b> | Phase 2 |
| Products: | Moderna [mRNA-1273, mRNA-1273.351, mRNA-1273.529, mRNA-1273.617.2] |
| | Pfizer [BNT162b2 (wildtype), BNT162b2 (B.1.351, Beta), BNT162b2 (B1.1.529, Omicron), BNT162b2 bivalent (wildtype and Omicron BA.1) and BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5)] |
| | Sanofi [CoV2 preS dTM-AS03 [D614] (prototype), CoV2 preS dTM-AS03 [B.1.351] (Beta), and CoV2 preS dTM-AS03 [D614 + B.1.351] (prototype + Beta)] |
| Form/Route: | Injection |
| Indication Studied: | COVID-19 |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | 30MAR2022 |
| Clinical Trial Completion Date: | Ongoing |
| Date of the Analysis Plan: | 10 October 2023 |
| Version Number: | 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | 2 |
|---|---|---|
| TABLE | OF CONTENTS | 3 |
| LIST OF | F ABBREVIATIONS | 6 |
| 1. | PREFACE | 8 |
| 2. | INTRODUCTION | 9 |
| 2.1. | Purpose of the Analyses | 12 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 13 |
| 3.1. | Study Definitions and Derived Variables | 14 |
| 4. | INVESTIGATIONAL PLAN | 15 |
| 4.1. | Overall Study Design and Plan | 15 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 15 |
| 4.3. | Selection of Study Population | 16 |
| 4.4. | Treatments | 18 |
| 4.4.1. | Treatments Administered | 18 |
| 4.4.2. | Identity of Investigational Product(s) | 18 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 19 |
| 4.4.4. | Selection of Doses in the Study | 19 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 20 |
| 4.4.6. | Blinding | 20 |
| 4.4.7. | Prior and Concomitant Therapy | 20 |
| 4.4.8. | Treatment Compliance | 20 |
| 4.5. | Immunogenicity and Safety Variables | 21 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 25 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 26 |
| 6.1. | General Principles | 26 |
| 6.2. | Timing of Analyses | 26 |
| 6.3. | Analysis Populations | 26 |
| 6.3.1. | Modified Intention-to-Treat (mITT) Population | 26 |
| 6.3.2. | Per Protocol Population | 26 |
| 6.3.3. | Safety Population | 26 |

#### **Table of Contents** (continued) 6.4. 6.5. 6.6. Interim Analyses and Data Monitoring .......27 6.7. 6.8. 7. 7 1 7.2. 8. IMMUNOGENICITY EVALUATION .......29 8.1. 8.2. 8.3. 8.3.1. 8.3.2. B-cells 30 8.3.3. 8.3.4. Sequencing Results of Breakthrough Infections.......31 9. SAFETY EVALUATION ......32 9.1. 9.1.1. 9.1.2. Prior and Concomitant Medications 32 9.2. 9.3. Adverse Events 33 9.3.1. 9.3.2. 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events .......34 9.5. Pregnancies 34 9.6. 9.7. Vital Signs and Physical Evaluations ......34 9.8. 9.9. 10. PHARMACOKINETICS ......35

| Table of Contents (continued) | | |
|---|---|---|
| 11. | IMMUNOGENICITY | 36 |
| 12. | OTHER ANALYSES | 37 |
| 13. | REPORTING CONVENTIONS | 38 |
| 14. | TECHNICAL DETAILS | 39 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 40 |
| 16. | REFERENCES | 41 |
| 17. | LISTING OF TABLES, FIGURES, AND LISTINGS | 44 |
| APPENDI | CES | 45 |
| APPENDI | X 1. TABLE MOCK-UPS | 46 |
| APPENDI | X 2. FIGURE MOCK-UPS | 227 |
| APPENDI | X 3. LISTINGS MOCK-UPS | 383 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event |
|--------|--------------------------------------------------|
| CI | Confidence Interval |
| CRF | Case Report Form |
| DMID | Division of Microbiology and Infectious Diseases |
| DSMB | Data and Safety Monitoring Board |
| EDC | Electronic Data Capture |
| ECLIA | Electrochemiluminescence Immunoassay |
| GMT | Geometric Mean Titer |
| FRNT | Focus Reduction Neutralization Assay |
| GMFD | Geometric Mean Fold Drop |
| GMFR | Geometric Mean Fold Rise |
| GMR | Geometric Mean Ratio |
| ICH | International Conference on Harmonisation |
| IRB | Institutional Review Board |
| ITT | Intention to Treat |
| LLOD | Lower Limit of Detection |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intention to Treat |
| N | Number (typically refers to subjects) |
| NIH | National Institutes of Health |
| PI | Principal Investigator |
| PP | Per Protocol |
| PsVNA | Pseudovirus Neutralization Assay |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| SOC | System Organ Class |

# **List of Abbreviations** (continued)

| SOP | Standard Operating Procedures |
|-----|-------------------------------|
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "Phase 2 Clinical Trial to Optimize Immune Coverage of SARS-CoV-2 Existing and Emerging Variants" (DMID Protocol 22-0004) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity and safety outcomes, and (4) a list of proposed tables and figures. Within the table, figure, and listing mock-ups (Appendix 1, Appendix 2, and Appendix 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

The Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) was first detected in Wuhan, Hubei Province, China in December 2019. The corresponding illness designation, coronavirus disease 2019 (COVID-19), was declared as a pandemic respiratory illness in March 2020 [1]. As of 18 August 2022, it has infected close to 600 million people worldwide and resulted in more than 6 million deaths, including close to 1 million in the United States [1, 2].

Six Phase 3 efficacy trials of SARS-CoV-2 vaccine constructs were conducted and are in long-term follow-up in the U.S. The ModernaTX, Inc mRNA-1273 and Pfizer/BioNTech BNT162b2 mRNA platforms encode for the full-length spike (S) protein of SARS-CoV-2, modified to introduce 2 proline residues to stabilize the S protein (S-2P) in a prefusion conformation, derived from the Wuhan-Hu-1 strain (prototype) [3]. The Janssen Pharmaceutical/Johnson & Johnson COVID-19 Vaccine (Ad26.COV.2) is composed of recombinant, replication-incompetent human adenovirus type 26, encoding a prefusion-stabilized SARS-CoV-2 spike antigen [4]. Studies of the Pfizer and Moderna mRNA vaccines demonstrated high efficacy against all symptomatic and severe disease and received Emergency Use Authorization (EUA) on December 12 and 18, 2020, respectively and full FDA approval on August 23, 2021 and January 31, 2022. Similarly, Janssen Pharmaceuticals reported 66% vaccine efficacy with a single dose and high-level protection against severe disease and death. FDA EUA was issued on February 26, 2021. Novavax's NVX-CoV2373, a recombinant nanoparticle vaccine containing the full-length spike protein received FDA EUA on July 13, 2022[5]. AstraZeneca/Oxford's ChAdOx-2, a recombinant, replication-incompetent chimpanzee adenovirus vector that expresses the spike protein, and Sanofi/GSK's adjuvanted recombinant spike protein vaccine are currently not licensed [6, 7]. Despite widespread vaccine distribution and availability, and high coverage among adults in the United States (87.4% of the US population  $\geq$  18 years of age have received at least one dose) [8], ongoing waves of the pandemic continue to cause significant disease burden, notable for increasing incidence of breakthrough infections in fully vaccinated individuals. Studies have suggested that vaccine protection against symptomatic SARS-CoV-2 infection wanes over time though protection against severe COVID-19 outcomes remains relatively intact [9, 10, 11, 12]. However, the evolution of variant strains may favor immune escape or reinfection among previously infected or vaccinated individuals. A variant first identified in late 2020 (B.1.351), is associated with increased transmission, higher viral burden, and possibly increased mortality in infected persons [13]. Another variant identified in December 2020 (B.1.617.2) is associated with increased transmission, higher risk of severe disease and hospitalization than the ancestral strain [14]. B.1.617.2 was the dominant strain worldwide before being replaced by B.1.1.529 in November 2021 which is characterized by a replication advantage, higher re-infection rates and evasion of humoral immunity mediated by more than 30 mutations in the spike protein [15].

Recent data suggest that a booster dose given as either a third dose for most vaccines (mRNA, protein and ChAdOx-2) or a second dose for Janssen improved vaccine effectiveness against new variants in the short term [16, 17, 18]. Data on immunogenicity with booster doses of BNT162b2, mRNA-1273, and AD26.COV2.S demonstrated higher antibody titers to D614G after either homologous and heterologous prime-boost combinations [19]. The result is better neutralizing activity against B.1.351, B.1.617.2 and B.1.1.529 [20, 21, 22]. In an open label phase 2 study of participants who received a single 50 mcg booster dose of mRNA-1273  $\geq$  6 months after a primary series, a 13-fold rise in antibody titers against D614G were noted from pre-boost levels as well as a 17-fold rise in in titers against the B.1.617.2 variant [20]. In another study, participants boosted with 50 mcg of mRNA-1273 demonstrated ID<sub>50</sub> GMTs against the omicron variant 20 times higher than those described 1 month after the second vaccination of the primary series; these titers were 2.9 times lower than titers for the D614G variant [21].

The Sanofi/GSK adjuvanted recombinant prefusion spike protein vaccine (CoV2 preS dTM-AS03 [D614]) was developed from an established, platform used for influenza vaccines. A phase 2 study showed the safety and immunogenicity of a two-dose primary series of CoV2 preS dTM-AS03 [D614] in adults who were SARS-CoV-2 naïve and those who were previously infected [23]. The dose-finding results informed selection of the adjuvanted formulation with 10 mcg antigen as primary dose and the adjuvanted formulation with 5 mcg antigen as boost dose for further evaluation. Neutralizing antibody titers were higher in non-naïve participants after one dose than in naïve participants after two doses. In addition, 5 mcg booster dose increased neutralizing antibody titers when used as a heterologous (18-30 times) or homologous (≥ 84 times) boost compared to pre boost [24]. Interim results from an international phase 3 trial showed 57.9% (95% confidence interval 26.5% to 76.7%) efficacy of the two-dose primary series against any symptomatic disease and 75% efficacy against moderate or severe COVID-19 with an acceptable safety and reactogenicity profile [24].

FDA EUA was subsequently issued for a booster 30 ug dose of Pfizer BNT162b2 on September 24, 2021, 50 ug booster dose of Moderna mRNA-1273 on October 21, 2021, and a 5×10<sup>10</sup> viral particles booster dose of J&J AD26.COV2 on October 21, 2021. This was recommended for adults 18 years of age and older who received a FDA authorized and CDC recommended primary booster series with an mRNA vaccine at least 5 months prior or a primary series with AD26.COV2 at least 2 months prior. The Sanofi/GSK vaccine is currently undergoing regulatory review for approval of their vaccine candidate for the prevention of COVID-19.

Published reports have also provided some early evidence for the safety and immunogenicity of a fourth dose of an mRNA vaccine. An open-label study of healthcare workers in Israel suggests that a fourth dose was well-tolerated and restored neutralizing antibody titers for variants to levels similar to those after a third dose [25]. Notably, this study did not include older adults, and rates of infection with B.1.1.529 (omicron) were similar for the control and Pfizer or Moderna 4<sup>th</sup> dose groups. In a retrospective study conducted by the Israeli Ministry of Health, of 1,138,681 adults aged 60 to 100 years of age, a fourth dose of mRNA was associated with 2 times lower rate of confirmed infection 12 or more days after vaccination compared to those who had only received 3 doses and the rate of severe illness was lower by a factor of 4.3 [26]. However, the added protection of an additional booster shot is small in absolute terms since less than 0.1% mortality was noted after a 3<sup>rd</sup> dose. Additionally, a separate study of adults age 60 or older suggests that vaccine effectiveness of a fourth dose against infection wanes quickly declining from a peak of 64% to 29% within 2 months though effectiveness of >73% was maintained against severe disease [27].

On March 29, 2022, the FDA authorized an additional booster dose of an mRNA vaccine for adults 50 years of age or older, or for those with immunocompromising conditions (12 years and older with immunocompromising conditions could receive a second booster with the Pfizer vaccine and 18 years and older could receive a second booster with the Moderna vaccine). Subsequent to this authorization, the CDC updated vaccination guidance to permit an additional booster dose for these groups in recognition of the increased and ongoing risk for severe disease in these populations.

The emergence of variant strains has raised concerns about the breadth and duration of immunity and protection achieved by the current vaccines. Studies of vaccine immunogenicity for early variants of concern demonstrated those vaccinated to prototype vaccine may have reduced neutralizing activity to the variants [28]. For variants like B.1.351, pivotal studies testing both viral vector and adjuvanted protein technologies had lower efficacy in regions where B.1.351 was known to be circulating [29, 30]. Moreover, sera from individuals vaccinated with mRNA-based vaccines had a 6-to-9-fold reduction in neutralizing activity against a B.1.351-matched pseudovirion relative to a Wuhan-matched pseudovirion [10, 11]. Similarly, sera from

individuals vaccinated with mRNA-1273 had an 8-fold reduction in neutralizing activity against the B.1.617.2 variant compared to titers against the D614G variant [21].

Studies have also demonstrated 6.7 fold reduction in neutralizing activity for Pfizer BNT162b2 against B.1.351 with two doses of Pfizer BNT162b2 [31]. Additionally, in one assessment of sera obtained from individuals vaccinated with Pfizer BNT162b2, obtained one month after the second dose, a 25 fold reduction in neutralizing antibody geometric mean titers against B.1.1.529 was noted compared to the wild-type virus [32]. Neutralizing activity has been shown to be partially restored by vaccination with a third dose of Pfizer BNT162b2. However, even with three doses, neutralizing activity was 4 times lower against B.1.1.529 and 3 times lower against B.1.351 compared to B.1.617.2 and 7-8 times lower compared to wild-type virus [33]. Thus, additional vaccinations, higher doses or variant specific vaccines may improve protection against current and emerging variants of concern.

Vaccine manufacturers have performed some trials of candidate variant vaccines. For example, a phase 2a open label clinical trial to examine the immunological benefit of boosting subjects previously vaccinated 6 months prior with mRNA-1273 with mRNA-1273.351, a B.1.351 strain-specific mRNA construct (50 mcg), or mRNA-1273.211 (50 mcg) showed 61.6 and 33.7 times higher titers against B.1.351 compared to titers from participants one month after the second dose of the primary series, with similar titers against B.1.617.2 [22]. Similar findings were seen from a study of a boost with a bivalent mRNA-1273.213 vaccine (a 1:1 mix of beta and delta variant mRNA) [21].

Similarly, several BNT162b2-based variant vaccines that target these variants are also being developed including BNT162b2 (B.1.617.2), BNT162b2 (B.1.351) and BNT162b2 (B.1.1.529). In addition, Sanofi has developed a SARS-CoV2 prefusion Spike delta TM with AS03 adjuvant (CoV2 preS dTM-AS03 [B.1.351]) monovalent vaccine and a SARS-CoV2 prefusion Spike delta TM with AS03 adjuvant bivalent vaccine (D614/B.1.351 (CoV2 preS dTM-AS03 [D614 + B.1.351]). In a nonhuman primate model, these vaccines used as boosters induced cross-neutralizing antibodies against variants of concern including Delta and Omicron [34].

However, current efforts are directed towards modifying the existing vaccines to include the current circulating Omicron variant, though this may not be the circulating variant during the next wave of COVID-19. It is therefore important to look beyond Omicron, and understand the immunologic landscape and how we can use prototype and variant vaccines alone or in combination to address emerging variants.

For seasonal influenza viruses, the antigenic, viral genetic and epidemiological data guide annual updates of the seasonal influenza virus vaccines. Antigenic cartography is a visualization tool aimed at understanding the relationship among SARS-CoV-2 variants of concern (VOCs) in terms of their ability to induce cross-neutralizing antibodies. A recent study using the antigenic mapping approach showed that Omicron represents the first widely circulating new major SARS-CoV-2 variant [35]. Though the dimensions of the cartography, representing new VOCs that could circulate in the future, remain largely unknown, a better understanding of diverse immune landscape induced by vaccination and natural infection could lead, along with vaccine modification, to more durable and broadly protective immunity. The update in vaccine formulations proposed in this study will still rely on similar platforms, route of administration and dosing, though will include an update of immunogens with VOCs alone or in combination that could result in broadly cross reactive serological and cellular immune responses especially in groups with high risk for mortality (e.g., older adults).

This phase 2 clinical trial will evaluate the safety and immunogenicity of additional doses of vaccine to expand and optimize immune coverage of the existing and emerging antigenic space. Utilizing several prototype and variant specific COVID-19 vaccines based on mRNA and other approved platforms, we propose to evaluate innate, cellular, and humoral immune responses elicited from different vaccine

candidates. As part of an adaptive design, we anticipate adding groups with other variant-lineage spike proteins and other vaccine platforms, subject to availability.

# 2.1. Purpose of the Analyses

These analyses will assess the immunogenicity and safety of additional doses of prototype and variant (alone or in combination) vaccine candidates in previously vaccinated participants with or without prior SARS-CoV-2 infection, and will evaluate innate, cellular, and humoral immune responses to inform on how to shift the immune response to cover new variants as they emerge.

Data may be disseminated to public health officials and partners as needed and included in publications and presentations to inform the global scientific community. Early analyses will include safety and immunogenicity as described in Protocol v5.0 Sections 9.4.6.1, 9.4.6.2, and 9.4.6.3. Further, the protocol team will review data periodically to confirm no halting criteria have been met as described in Protocol v5.0 Section 7.1.1.

# 3. STUDY OBJECTIVES AND ENDPOINTS

**Table 1: Objectives and Endpoints (Outcome Measures)** 

| OBJECTIVES | ENDPOINTS (OUTCOME MEASURES) |
|---|---|
| Primary | |
| To evaluate humoral immune responses of<br>candidate SARS-CoV-2 variant vaccines | Response rate and magnitude of SARS-CoV-<br>2-specific antibody binding and<br>neutralization titers in serum samples as<br>assessed via a range of assays at all<br>timepoints |
| Secondary | |
| To evaluate the safety of candidate SARS-<br>CoV-2 variant vaccines | <ul> <li>Local and systemic solicited Adverse Events<br/>for 7 days following each vaccine dose</li> <li>Unsolicited Adverse Events from Dose 1 to</li> </ul> |
| | 28 days following each vaccine dose |
| | SAEs, MAAEs, NOCMCs, AESIs, and AEs leading to withdrawal from the study from Dose 1 to 12 months after the last vaccine dose |
| Exploratory | |
| To assess, in at least a subset of samples, the B cell immune response of candidate SARS-CoV-2 variant vaccines | Magnitude, phenotype, and percentage of<br>SARS-CoV-2-specific B cells, as measured<br>by flow cytometry and targeted B cell subset<br>analysis at selected time points post-<br>vaccination |
| To assess, in at least a subset of samples, the SARS-CoV-2 spike protein-specific T cell responses of candidate SARS-CoV-2 variant vaccines | Magnitude, phenotype, and percentage of cytokine-producing S protein T cells as measured by flow cytometry at selected time points post-vaccination. |
| To assess, in at least a subset of samples, the magnitude, phenotype, and percentage of innate immune cells with candidate SARS-CoV-2 variant vaccines | Magnitude, phenotype, and percentage of innate immune cells as measured by flow cytometry at D1 and 14 days after each vaccination |
| To assess, in at least a subset of samples, the function potential of SARS-CoV-2 specific antibodies to mediate Fc-effector functions | Characterization of antigen-specific antibody<br>by a) subclass, b) isotype, c) ability to<br>interact with Fc receptors, d) innate immune |

| OBJECTIVES | ENDPOINTS (OUTCOME MEASURES) |
|---|---|
| across candidate SARS-CoV-2 variant vaccines | receptors, e) lectin-like molecules, and f) lectins at different times post-vaccination |
| | Functional Fc effector assessments which may include quantification of antigen-specific antibody-mediated NK cell activation (ADCC-NK) levels, antibody-dependent cellular phagocytosis (ADCP) levels, antibody-dependent complement deposition (ADCD) and/or antibody-dependent neutrophil activation/phagocytosis levels at different times post-vaccination |
| To evaluate breakthrough SARS-CoV-2 infection by sequencing strains for variant spike lineage and assessing antinucleocapsid serology | <ul> <li>Sequence analysis on breakthrough NAAT-confirmed SARS-CoV-2 strains at any time post-vaccination</li> <li>Anti-nucleocapsid immunoassay at different times post-vaccination</li> </ul> |

# 3.1. Study Definitions and Derived Variables

For calculations using the baseline value, the value obtained pre-fourth vaccination (Day 1) will be used.

If a value falls below the lower limit of detection for the immunogenicity assay, the value will be replaced by one-half the lower limit of detection in analyses.

Subjects infected at baseline will be defined as by either self-report or positive for N-antibody.

Major protocol deviations will be defined by the sponsor.

Unless otherwise noted Omicron refers to B.1.1.529/BA.1.

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

This is a Phase 2 randomized, adaptive, open label, non-placebo controlled multi-site, multi-stage clinical trial in individuals, 18 years of age and older, who are in stable state of health, have received a complete authorized/approved vaccine series (primary series + booster either with homologous or heterologous vaccine products) and meet all other eligibility criteria.

Approximately 1500 subjects will be enrolled at up to 30 clinical research sites. At enrollment, subjects will be stratified by i) age (18-64 and  $\geq$  65 years of age) (however arms 16 and 17 or stage 4 will only enroll participants between the ages of 18-49 years) and ii) confirmed prior SARS-CoV-2 infection, and randomly assigned to one of several study arms of variant vaccines. The study will target the enrollment of approximately 45% older adults ( $\geq$  65 years of age) for stages 1, 2, and 3. Additionally, the study will target to enroll approximately 20% of participants with a history of confirmed SARS-CoV-2 infection. It is estimated that another 10-30% will have undiagnosed prior infection. Taken together, we anticipate about 40% of the total enrolled participants will have prior infection. The study team will decide, based on latest epidemiology, if enrollment of participants in any particular groups are slowed in order to ensure good representation of previously infected and not previously infected.

The adaptive design of this study will include additional arms, an increase in sample size, or additional vaccine doses or different dosing and provide rapid information about the immunogenicity and the safety of candidate SARS-CoV-2 variant vaccines to inform near term public health policy. This trial will provide proof of concept on how variant vaccines could shift the immune response to become more specific to the VOCs' antigens or broaden the antigenic landscape for emergent variants.

Screening can occur up to 28 days prior to the first dose of study product or on Day 1 prior to administration of Dose 1. Safety will be assessed during the study and blood will be drawn for immunogenicity assays at enrollment and in-person follow-up visits. Swabs will be self-collected or collected by staff at unscheduled illness visits to evaluate breakthrough SARS-CoV-2 infection (symptomatic infection or asymptomatic infection with a positive SARS-CoV-2 test outside the study). A summary of the four currently planned stages can be found in Table 2.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

This phase 2 study is an open-label study, without administration of a placebo formulation. An open-label study will facilitate the need for rapid review and dissemination of study data for public health reasons. Safety findings are not expected to be dissimilar from Phase 1/2/3 studies conducted for similar vaccine constructs. Randomization will improve comparisons between different arms. Each stage will contain an arm with a monovalent prototype vaccine (except for stage 4).

Selected arms will assess 2 study doses of vaccine candidates to assess if 2 doses provide a more durable and specific response to variant viruses.

An interval of 4 months was chosen since a recent study performed by the investigators showed that an interval of 3 months between primary series and boost had acceptable safety and immunogenicity responses [19].

# 4.3. Selection of Study Population

All participants will have received a complete (primary and booster) US approved/authorized vaccine series. The US population has received either homologous primary series and boost (i.e. Moderna mRNA-1273 for lst dose, second dose, and booster), or heterologous boosters, and some were infected with SARS-CoV-2 either prior to or after vaccination. This trial will enroll this immunologically diverse population, to ensure any findings are applicable to the larger population.

Based on CDC data about use of primary vaccine or boost (https://covid.cdc.gov/covid data-tracker/#vaccinations\_vacc-total-admin-rate-total), it is estimated that of people in the US that have received a primary vaccine series and booster:

- 50% will have received Pfizer primary series and Pfizer boost,
- 37% will have received Moderna primary series and Moderna boost,
- 4% will have received Pfizer primary series and Moderna boost,
- 3% will have received Moderna primary series and Pfizer boost,
- 1% will have received Janssen primary series and Janssen boost,
- 2% will have received Janssen primary series and Moderna boost,
- 2% will have received Janssen primary series and Pfizer boost.

Additionally, approximately 20% of the US population has been infected with SARS-CoV-2, likely higher with asymptomatic infections [36].

It is anticipated the enrollment into this trial will be similar to these proportions.

Subject Inclusion and Exclusion Criteria must be confirmed by a study clinician, licensed to make medical diagnoses and listed on the Form FDA 1572. No exemptions are granted on Subject Inclusion or Exclusion Criteria in DMID-sponsored studies.

#### **Inclusion Criteria**

Participants must meet all the following criteria to be eligible to participate in this study:

- 1. Individuals  $\geq$  18 years of age at the time of consent (18-49 years for stage 4).
- Confirmed receipt of a complete primary and booster COVID-19 vaccine series, either homologous or heterologous, with an FDA authorized/approved vaccine at least 16 weeks prior to study vaccine dose 1
- 3. Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests and other study procedures
- 4. Determined by medical history, targeted physical examination and clinical judgement of the investigator to be in stable state of health

Note: Participants with pre-existing stable chronic medical conditions defined as condition not requiring significant change in therapy or hospitalization for worsening disease within 4 weeks form enrollment, can be included at the discretion of the investigator.

#### **Exclusion Criteria**

Participants meeting any of the following criteria will be excluded from participation in this study:

- 1. Confirmed SARS-CoV-2 infection < 16 weeks prior to any study vaccine dose
- 2. Pregnant and breastfeeding participants
- 3. Prior administration of an investigational coronavirus vaccine at any time or SARS-CoV-2 immunoglobulin, monoclonal antibody or plasma antibody therapy in the preceding 3 months
  - Note: Subjects that participated in clinical trials of products that are now FDA approved/authorized are allowed to participate.
- 4. Current/planned simultaneous patriation in another interventional study or receipt of any investigational study product within 28 days prior to vaccine study dose(s)
- 5. A history of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine, polyethylene glycol (PEG), or nanolipid particles.
- 6. A history of myocarditis or pericarditis at any time prior to enrollment (for subjects in stages 1, 2 and 4).
- 7. Received or plans to receive a vaccine within 28 days prior to or after any dose of study vaccine.
  - Note: Receipt of seasonal influenza vaccine is allowed at any time
- 8. Bleeding disorder diagnosed by a healthcare provider (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or bleeding difficulties with intramuscular injections or blood draws.
- 9. Current or previous diagnosis of an immunocompromising condition or other immunosuppressive condition.
- 10. Advanced liver or kidney diseases.
- 11. Advanced (CD4 count < 200) and/or untreated HIV, untreated Hepatitis B or untreated Hepatitis C.
- 12. Received oral, intramuscular or intravenous systemic immunosuppressants, or immune-modifying drugs for >14 days in total within 6 months prior to any study vaccine dose (for corticosteroids  $\geq$  20 mg/day of prednisone equivalent).
  - Note: Topical medications are allowed.
- 13. Received immunoglobulin or blood-derived products, within 3 months prior any study vaccine dose.
- 14. Received chemotherapy, immunotherapy or radiation therapy within 6 months prior to any study vaccine dose.
- 15. Study personnel or an immediate family member or household member of study personnel.
- 16. Is acutely ill or febrile 72 hours prior to or at vaccine dosing (fever defined as  $\geq 38.0^{\circ}\text{C}/100.4^{\circ}\text{F}$ ). Participants meeting this criterion may be rescheduled within the relevant window periods.
  - Note: Afebrile participants with minor illnesses can be enrolled at the discretion of the Investigator, as long as the illness is not suggestive of COVID-19.
- 17. Plan to receive a COVID-19 booster vaccine outside of the study within the next 180 days. (for subjects in Stage 4 only)

#### **Exclusion of Specific Populations**

The effects of SARS-CoV-2 vaccines on the developing fetus are not known, though there are data to suggest that mRNA vaccines are safe. Pregnant subjects will not be eligible for the trial as the immune responses to vaccines can be different than non-pregnant subjects. Children will not be included in this trial as presently there are limited safety data in adults for the variant strains.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

Seventeen treatment arms administer various combinations of COVID-19 vaccines (Table 2).

#### 4.4.2. Identity of Investigational Product(s)

# <u>Products: mRNA-1273 (Prototype), mRNA-1273.351 (Beta), mRNA-1273.617.2 (Delta), and mRNA-1273.529 (Omicron)</u>

mRNA-1273 (0.2 mg/mL) is an LNP dispersion containing an mRNA that encodes for the pre-fusion stabilized S protein of the Wuhan-Hu-1 strain of SARS-CoV-2. mRNA-1273 consists of an mRNA Drug Substance that is manufactured into LNPs composed of the proprietary ionizable lipid, SM-102, and 3 commercially available lipids, cholesterol, 1,2-distearoyl-sn-glycero-3-phosphocholine (DSPC), and PEG2000 DMG.

mRNA-1273.351 (0.1 mg/mL) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 (Beta) variant SARS-CoV-2 strain.

mRNA-1273.617.2 (0.2 mg/mL) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the B.1.617.2 (Delta) variant SARS-CoV-2 strain.

mRNA-1273.529 (0.2 mg/mL) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.

# BNT162b2 (wildtype), BNT162b2 (B.1.351, Beta), BNT162b2 (B1.1.529, Omicron), BNT162b2 bivalent (wildtype and Omicron BA.1) and BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5)

BNT162b2 (500 mcg/mL for stage 2) is a preservative-free, sterile dispersion of RNA formulated in LNP in aqueous cryoprotectant buffer. mRNA encodes for the pre fusion stabilized S protein of the ancestral strain of SARS-CoV-2.

BNT162b2 (B.1.351) (500 mcg/mL for stage 2) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the B.1.351 (Beta) variant SARS-CoV-2 strain.

BNT162b2 (B.1.1.529)(500 mcg/mL for stage 2) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the B.1.1.529 (Omicron) variant SARS-CoV-2 strain.

BNT162b2 bivalent (wildtype and Omicron BA.1 100mcg/mL for stage 4) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the Omicron BA.1 variant SARS-CoV-2 strain and the ancestral strain of SARS-CoV-2..

BNT162b2 bivalent (wildtype and Omicron BA.4/BA.5 100mcg/mL for stage 4) is formulated in the same way but contains mRNA that encodes for the prefusion stabilized S protein of the Omicron BA.4/BA.5 variant SARS-CoV-2 strain and the ancestral strain of SARS-CoV-2.

# <u>CoV2 preS dTM-AS03 [D614] (prototype), CoV2 preS dTM-AS03 [B.1.351] (Beta), and CoV2 preS dTM-AS03 [D614 + B.1.351] (prototype + Beta)</u>

CoV2 preS dTM-AS03 [D614] (Recombinant COVID-19 Vaccine 20 mcg/mL + AS03) is a liquid formulation made of recombinant protein placed in a formulation buffer and to be mixed with equal volumes of AS03 adjuvant (supplied separately) at the study site before administration. The antigen solution contains the Spike protein sequence of the ancestral strain of SARS-CoV-2. AS03 is an adjuvant system containing α-tocopherol and squalene in an oil/water emulsion. For this formulation, the antigen and AS03 vials are not packaged in a carton box together but are supplied as individual vials.

CoV2 preS dTM-AS03 [B.1.351] (Recombinant COVID-19 Vaccine B1.351 20 mcg/mL+ AS03) is formulated in the same way but contains the Spike protein sequence of the B.1.351 (Beta) variant SARS-CoV-2 strain. Both antigen and AS03 vials are packaged in a carton box.

CoV2 preS dTM-AS03 [D614 + B.1.351] (Recombinant COVID-19 Bivalent Vaccine 10/10 mcg/mL + AS03) is formulated in the same way but contains the Spike protein sequences of the ancestral and B.1.351 (Beta) variant SARS-CoV-2 strains. Both antigen and AS03 vials are packaged in a carton box.

#### **Diluent: 0.9% NaCl for injection, USP**

The USP grade 0.9% NaCl or normal saline for injection is a sterile, nonpyrogenic, isotonicsolution; each mL contains NaCl 9 mg. It contains no bacteriostatic agent, antimicrobial agent, preservatives, or added buffer and is supplied only in single-dose containers. This product should be used to dilute the vaccine to the desired concentration.

#### 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

Subjects will be randomized to study intervention in an equal allocation ratio within each stage. The study will be open label and study sites will administer product to a subject according to which study arm the subject has been assigned. Sites will be asked to recruit for all arms within a stage.

#### 4.4.4. Selection of Doses in the Study

The dosages of mRNA vaccines selected are those authorized for booster doses under EUA, and previously shown in prior studies to elicit good immune responses with no major safety concerns.

In an open label study of participants in the Moderna Phase 3 clinical trial who received a single 50 mcg booster dose of mRNA-1273 ≥ 6 months after a primary series, a 13 fold rise in antibody titers against D614G was noted from pre-boost levels as well as a 17-fold rise in in titers against the B.1.617.2 variant [20]. This is now the CDC recommended dose for booster vaccinations with the Moderna mRNA-1273 product in immunocompetent adults, to be given at least 5 months from the last inoculation in the primary series [37]. Similarly, in a recent study, boosting with a 50 mcg total antigen dose of a bivalent mRNA-1273.213 vaccine (a 1:1 mix of beta and delta variant mRNA) produced only modestly lower antibody titers than using a 100 mcg booster dose [21]. A separate study evaluating safety and immunogenicity of multiple boost strategies suggests that a heterologous boost strategy generates antibody and neutralizing responses and that 100 mcg of mRNA-1273 (the authorized dose at the time) is likely higher than needed for a booster dose after primary mRNA series [38]. In addition, surveillance data indicate that following an mRNA boost, local and systemic reactions are less common and myocarditis is rarely reported, suggesting that the currently authorized doses are safe [39]. These findings support the evaluation of mRNA-1273, mRNA-1273.351, mRNA-1273.617.2 and mRNA-1273.529 at total dosages of 50 mcg per vaccination.

For BNT162b2, the dose is the same for primary or booster doses in adults. In an open-label clinical study, immunogenicity and safety of a fourth dose of either 30 mcg of BNT162b2 (Pfizer–BioNTech) or 50 mcg of mRNA-1273 (Moderna) administered 4 months after the third dose was assessed in 154 and 120 health care workers, respectively [25]. After the fourth dose, both messenger RNA (mRNA) vaccines increased neutralizing antibody titers to D614G, B.1.617.2 and B.1.1.529 by a factor of 9 to 10 and were slightly higher than those achieved after the third dose [25]. There were no significant adverse events with only mild system and local reactogenicity reported which was comparable with previous doses of mRNA vaccines. The bivalent booster of BNT162b2 was authorized by the FDA based on pre-clinical data (Omicron BA.4/BA.5 + prototype) [40].

For CoV2 preS dTM-AS03 vaccines, none are currently approved. The dose used for booster vaccination is as established in the phase 2 trial and is the adjuvanted formulation with 5 mcg for any variant vaccine candidate in stage 3 [24]. That booster dose increased neutralizing antibody titers when used as a heterologous (18-30 times) or homologous (≥ 84 times) boost [24]. However, no data exist on CoV2 preS dTM-AS03 vaccines as a second boost after primary series with mRNA or adenoviral vectored vaccines.

#### 4.4.5. Selection and Timing of Dose for Each Subject

Subjects will be randomly assigned to a study intervention. Subjects assigned to the arm receiving 2 doses will receive dose 2 eight weeks after dose 1.

#### 4.4.6. Blinding

This study is unblinded.

#### 4.4.7. Prior and Concomitant Therapy

Concomitant medications include prescription medications and vaccinations taken within 28 days of screening or Day 1. Topical, ophthalmic and OTC medications, herbal supplements and vitamins will not be collected. This information is asked to assess eligibility. Only COVID-19 vaccination received at any time in the past will be captured in the trial database. After enrollment, immunosuppressant drugs, COVID-19 vaccines received outside of the study as well as COVID-19 related treatment and prophylaxis should be reported at any time during study participation and captured in the trial database. At each study visit, if there are new SAEs, concomitant medications should be recorded on the appropriate DCF and not included in the database unless these are immunosuppressant drugs, COVID-19 vaccines received outside of the study or COVID-19 related treatment and prophylaxis.

#### 4.4.8. Treatment Compliance

Subjects in all treatment arms except for treatment arm 3 will receive a single dose of study product administered in the clinic. Subjects in treatment arm 3 will receive 2 total doses (Days 1 and 57) of study product administered in the clinic.

# 4.5. Immunogenicity and Safety Variables

#### **Immunogenicity**

#### **Humoral Immunogenicity Assays**:

The following humoral immunogenicity assays may be performed:

- IgG ELISA or Multiplex MSD antibody binding assays to SARS-CoV-2 proteins (may include nucleocapsid protein, and multiple variant Receptor Binding Domains (RBD) and variant spike proteins).
- Neutralization assays using SARS-CoV-2 variant specific S-pseudotyped viruses.
- Neutralization assays using different strains of live SARS-CoV-2.
- Characterization of antigen-specific antibody by a) subclass, b) isotype, c) ability to interact with Fc receptors, d) innate immune receptors, e) lectin-like molecules and f) lectins at different times post-vaccination.
- Functional Fc effector assays which may include quantification of antigen specific antibody-mediated NK cell activation (ADCC-NK) levels, antibody-dependent cellular phagocytosis (ADCP) activity, Antibody-dependent complement deposition (ADCD) and/or Antibody-dependent neutrophil activation/phagocytosis activity.

#### Cellular Immunology Assays:

This trial may also investigate innate, B and T cell immune responses using multiparametric flow cytometry. Refer to the protocol-specific immune monitoring plan for details.

#### Safety

All safety endpoints for this trial are obtained by reporting of adverse events.

- New symptoms will be queried with broad open-ended questions at the Day 8 telephone call and by specifically asking about symptoms of chest pain, shortness of breath or palpitations that may represent myocarditis and/or pericarditis.
- Data on new medical conditions, doctors' office visits (outside of routine care), emergency room visits, and hospitalizations will be collected.
- Memory Aid: All subjects will complete a Memory Aid from the time of each vaccination through 7 days after each vaccination. Subjects will be asked to confirm completion of the Memory Aid and will be queried on the presence of any grade 3 symptoms. Based on the information provided, subjects may be asked to return to the clinic for evaluation. Fourteen days after each vaccination, Memory Aids are reviewed thoroughly with the subject and confirmed data recorded in the CRF.

As these vaccines are similar to licensed vaccines, there are no laboratory assessments for safety that will be done for this trial.

#### Adverse Events

AE means any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related [21 CFR 312.32 (a)]. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of medicinal (investigational) product.

Any medical condition that is present at the time that the subject is screened will be considered as baseline and not reported as an AE. However, if the severity of any pre-existing medical condition increases, it should be recorded as an AE.

AEs can be further divided into solicited AEs and unsolicited AEs. Solicited AEs are those that are described in the package insert as local or systemic reactogenicity occurring in the first 7 days after vaccination. Unsolicited AEs are those events that the subject reports occurring without being queried about the specific event.

AEs will be assessed for severity and relationship to study intervention. Reporting of all AEs, solicited and unsolicited, will occur during the period from study product administration on Day 1 through 28 days after each vaccination. After 28 days post last vaccination through the end of study, only SAEs, Protocol Specified AESIs, MAAEs, NOCMCs, and AEs leading to withdrawal from the study will be reported.

All AEs, solicited and unsolicited, will be captured on the appropriate DCF. Solicited AEs will be regarded as related to the study product and will not require separate entry into the AE log. Information to be collected for unsolicited AEs includes event description, date of onset, assessment of severity, relationship to study product and alternate etiology (assessed only by those with the training and authority to make a diagnosis and listed on the Form FDA 1572 as the participating site PI or appropriate sub-investigator), date of resolution, seriousness, and outcome. AEs occurring during the study-collection and reporting period will be documented appropriately regardless of relationship.

AEs will be followed to resolution or stabilization.

#### Solicited Adverse Events

Solicited AEs are anticipated local and systemic AEs for which consistent collection of information is desired. Study clinicians will follow and collect resolution information for any reactogenicity symptoms that are not resolved within 7 days.

Solicited AEs (i.e., reactogenicity) will be collected using a memory aid and confirmed data recorded on the appropriate DCF from the time of each vaccination through 7 days post each vaccination.

For this study, solicited AEs will be:

- Injection site Pain
- Injection site Erythema
- Injection site Edema/Induration
- Headache
- Fatigue
- Myalgia
- Arthralgia
- Nausea
- Fever
- Chills

#### **Unsolicited Adverse Events**

All AEs spontaneously reported by the subject and/or in response to an open question from study staff or revealed by observation, physical examination or other diagnostic procedures must be recorded on the appropriate DCF.

Unsolicited AEs of all severities will be reported from the time of study product administration through 28 days post each vaccination.

After 28 days post last vaccination through the end of study, only SAEs, AESIs, NOCMCs, MAAEs, and AEs leading to withdrawal from the study will be reported.

#### Serious Adverse Events

An SAE is defined in 21 CFR 312.32 as follows: "An AE or suspected adverse reaction is considered serious if, in the view of either the participating site PI or appropriate sub-investigator or the sponsor, it results in any of the following outcomes:

- Death,
- a life-threatening AE,
- inpatient hospitalization or prolongation of existing hospitalization,
- a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions,
- or a congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse."

"Life-threatening" refers to an AE that at occurrence represents an immediate risk of death to a subject. An event that may cause death if it occurs in a more severe form is not considered life-threatening. Similarly, a hospital admission for an elective procedure is not considered an SAE.

All SAEs, as with any AE, will be assessed for severity and relationship to study intervention.

All SAEs will be recorded on the appropriate SAE DCF.

All SAEs will be followed through resolution or stabilization by a study clinician, licensed to make medical diagnoses and listed on the Form FDA 1572 as the participating site PI or appropriate sub-investigator.

All SAEs will be reviewed and evaluated by DMID and will be sent to the DSMB (for periodic review unless related) and IRB/IEC as needed.

#### Adverse Events of Special Interest (AESIs)

AESIs represent any events for which additional data (besides the standard AE data) are desired. An adverse event of special interest (serious or nonserious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor is required. Such an event may require further investigation in order to characterize and understand it. Depending on the nature of the event, rapid communication by the trial sponsor to other parties (e.g., regulators) may also be required. These may be at the request of the regulatory agency, industry partner or DMID, and driven by a regulatory requirement, or known or potential risk from the product or class.

Protocol Specified AESIs are listed in Appendix A of the protocol. In addition, for stage 3, AESIs will also include a list of pIMD.

#### Potential immune-mediated diseases (pIMDs)

pIMDs are a subset of AESIs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. AESIs that need to be recorded and reported as pIMDs for Stage 3 participants are listed in Appendix A of the protocol.

However, the investigator will exercise their medical and scientific judgement in deciding whether other diseases have an autoimmune origin (that is pathophysiology involving systemic or organspecific pathogenic autoantibodies) and should also be recorded as a pIMD.

When there is enough evidence to make any of the diagnoses mentioned in Appendix A of the protocol, the AESI must be reported as a pIMD. Symptoms, signs or conditions which might (or might not) represent the above diagnoses, should be recorded and reported as AEs but not as pIMDs until the final or definitive diagnosis has been determined, and alternative diagnoses have been eliminated or shown to be less likely.

#### New Onset of Chronic Medical Conditions (NOCMCs)

NOCMCs are defined as any new ICD diagnosis (per current International Statistical Classification of Diseases and Related Health Problems) that is applied to the subject during the course of the study, after receipt of the study agent, that is expected to continue for at least 3 months and requires continued health care intervention.

#### Medically Attended Adverse Events (MAAEs)

MAAEs are defined as a hospitalization < 24 hours, emergency room visit or an otherwise unscheduled visit to or from medical personnel for any reason; and considered related or possibly related to study product.

# Time Period and Frequency for Event Assessment and Follow-Up

For this study:

- Solicited Adverse Events will be collected for 7 days following each vaccine dose.
- Unsolicited AEs will be collected until 28 days after each vaccination.
- AESIs, NOCMCs, MAAEs, SAEs, and AEs leading to withdrawal from the study will be collected from Day 1 through the end of the study.

#### SARS-CoV-2 infection

Confirmed SARS-CoV-2 infection at any time during the study defined as a positive RT-PCR test performed by the site or using a non-site testing method (RT-PCT or antigen test), will be documented. While this event would occur on study, it is not typical AE and therefore captured as an exploratory efficacy assessment.

#### 5. SAMPLE SIZE CONSIDERATIONS

#### Sample Size Calculations for the Safety Endpoints

Rare AEs are not demonstrable in a clinical study of this size; however, the probabilities of observing one or more AEs given various true event rates are presented in Table 5. With the assumption that all enrolled subjects will likely complete immunizations and safety visits in this relatively short study duration, the following statistical considerations apply. With approximately 100 subjects there is a greater than 99.9% chance of observing at least one AE of probability 10%. With approximately 50 subjects, there is a 99.5% chance of observing at least one AE of probability 10%. With approximately 25 subjects, there is a 92.8% chance of observing at least one AE of probability 10%. Finally, with approximately 15 subjects, there is a 79.4% chance of observing at least one AE of probability 10%. Therefore, if no AEs of a given type occur in a group (or strata/subgroup), we can be relatively confident that they will occur in fewer than 10% of people if the vaccine is implemented.

#### Sample Size Calculations for the Immunogenicity Endpoints

The primary objective of this study is to evaluate the magnitude and durability of SARS-CoV-2 specific antibody titers in serum samples. This objective is descriptive in nature and will be accomplished by estimating 95% confidence intervals (CI) for the geometric mean titer (GMT) at each timepoint when samples are collected.

The precision with which the GMT can be estimated from observed data depends on the standard deviation (SD) of the measurements, on the logarithmic scale, and the sample size. Table 6 displays two-sided 95% confidence intervals for the GMT for several values of the observed antibody titer.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

Unless otherwise noted, continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum, and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by vaccine arm and subject, and when appropriate by visit number within subject. Summary tables will be structured with a column for each variant and will be annotated with the total population size relevant to that table/cohort, including any missing observations.

# **6.2.** Timing of Analyses

Interim analyses will occur as needed. Statistical analyses of immunogenicity endpoints, by vaccine arm, may be performed when subjects have completed key immunogenicity visits.

# 6.3. Analysis Populations

A tabular listing of all subjects, visits, and observations excluded from the immunogenicity analysis will be provided in the CSR (Listing 5).

#### 6.3.1. Modified Intention-to-Treat (mITT) Population

The modified intention-to-treat (mITT) population includes all subjects who received at least one dose of vaccine and contributed both pre- and at least one post-vaccination venous blood sample for immunogenicity testing for which valid results were reported.

#### **6.3.2.** Per Protocol Population

In the final analysis, protocol deviations will be reviewed to determine which protocol deviations may affect the analysis. The per protocol (PP) population will then be defined. The PP population will, at minimum, exclude the following from the mITT Population:

- Data from all available visits for subjects found to be ineligible at baseline.
- Data from all visits subsequent to the protocol deviations that are considered to affect the science.
- Data from any visit that occurs substantially out of window.

#### 6.3.3. Safety Population

The safety analysis population includes all enrolled subjects who received at least one dose of study vaccine. This population will be summarized according to the actual study vaccine received, not necessarily the vaccine to which a subject was randomized.

# 6.4. Covariates and Subgroups

Subgroup analyses, by age group and infection status, will be completed. Analyses for each subgroup will include descriptive summaries and confidence intervals but no formal hypothesis testing, following recommendations for subgroup analyses that may inflate false positive conclusion rates and lack statistical power. Additional exploratory subgroup analyses may be performed as required.

# 6.5. Missing Data

There are no imputations planned for missing data.

For immunogenicity assays, any values below the lower limit of detection will be imputed as one-half of the lower limit of detection for analysis purposes. Any such imputations will be noted in the corresponding analysis.

# 6.6. Interim Analyses and Data Monitoring

Cumulative safety information, study status, and primary endpoint results may be published, presented at a public forum, or presented as summaries aggregated by vaccination group at the discretion of the sponsor while the study is ongoing. None of the interim analyses will include any formal statistical hypothesis testing; therefore, p-value adjustment will not be made to any analyses.

#### 6.7. Multicenter Studies

Data will be pooled across all clinical sites. Center effects are not anticipated because the sites are using standardized procedures for vaccination and assessment of solicited and unsolicited adverse events, and the study relies on central laboratories for the assessment of immunogenicity endpoints.

### 6.8. Multiple Comparisons/Multiplicity

No hypothesis testing will be conducted, therefore, there are no p-value adjustments planned for multiple comparisons. Confidence intervals may be adjusted as appropriate.

#### 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

Table 11 will present a summary of the reasons that subjects were screened but not enrolled.

The composition of analysis populations, including reasons for subject exclusion, by vaccination arm, is presented in Table 10.

The disposition of subjects in the study will be tabulated by vaccination group (Table 9). The table shows the total number of subjects screened, enrolled, receiving at least 1 dose, receiving 2 doses (if applicable), discontinued dosing or terminated from study follow-up and the number completing the study.

A flowchart showing the disposition of study subjects, adapted from the Consort Statement [41] will be included (Figure 1). This figure will present the number of subjects screened, enrolled, lost to follow-up, and analyzed, by vaccination arm.

A listing of subjects who discontinued dosing or terminated from study follow-up and the reason will be included in Listing 1.

#### 7.2. Protocol Deviations

A summary of subject-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and vaccination group for all subjects (Table 7) as well as similar summaries for major subject-specific protocol deviations that may affect analyses (Table 8). All subject-specific protocol deviations and non-subject specific protocol deviations will be included in Appendix 3 as data listings (Listing 2 and Listing 3, respectively).

#### 8. IMMUNOGENICITY EVALUATION

# 8.1. Primary Immunogenicity Analyses

Descriptive summaries of immunogenicity data will be presented for the mITT population. If there are protocol deviations which may affect the analysis, an analysis of the per-protocol (PP) population may also be performed.

The results of three immunological assays will be analyzed. The 10-plex (ECLIA) assay is a fit-for-purpose assay that reports antibody concentrations as arbitrary units (AU) interpolated from ECL signal of internal standards or reports as area under the curve (AUC) and is used to assess antibody binding for variants of concern. The results of the 10-plex ECLIA assay will be summarized for each group at each timepoint by the geometric mean (GM), geometric mean fold rise (GMFR) from baseline (Day 1), geometric mean ratio (GMR) against D614G, and geometric mean fold drop (GMFD) from Day 29 (and Day 85 for 2 dose group) along with corresponding 95% confidence intervals (CIs). GMFR is defined as the ratio of the result at a timepoint divided by the result at Day 1. GMR is defined as the ratio of the result for a variant of concern to D614G (e.g. Beta to D614G). GMFD is defined as the ratio of the result at Day 29 (or day 85) divided by the result at a timepoint following day Day 29 (or Day 85). Seropositive rate is the proportion of subjects with a result above the lower limit of detection. The lower limit of detection will be annotated in the tables and figures where applicable. Summaries of the 10-plex ECLIA results are shown starting with Table 15 and ending with Table 122. Graphical displays will include geometric mean over time (starting with Figure 2 and ending with Figure 109), and distribution of responses over time (starting with Table 326 and ending with Table 433).

The SARS-CoV-2 pseudovirus neutralization assay (PsVNA) and focus reduction neutralization test (FRNT) will be run using serial dilutions against available variants (*e.g.* Beta, Delta, Omicron). From these assays, ID<sub>50</sub>, which estimates the amount of antibodies required for a neutralization rate of 50%, will be reported. Neutralization titers will be summarized by the GM, GMFR, GMR, GMFD, and seropositive rate with corresponding 95% CIs, for each group at each timepoint. The summaries of PsVNA results are shown starting with Table 123 and ending with Table 230, and the summaries of FRNT results are shown starting with Table 231 and ending with Table 338. Graphical displays for PsVNA and FRNT will include geometric mean over time (starting with Figure 110 and ending with Figure 325) and distributions of responses over time (starting with Figure 434 and ending with Figure 649).

The immunogenicity timepoints for single-dose arms are Study Days 1, 15, 29, 91, 181, 271, and 366. The timepoints for the two-dose arm are Study Days 1, 15, 29, 57, 71, 85, 147, 237, 327, and 422. CIs for GM, GMFR, GMR, and GMFD will be calculated using the Student's t-distribution and CIs for seropositive rates will be calculated using the Clopper-Pearson binomial method. If additional immunological assays are determined to be necessary, then the results will be summarized in a similar manner to that of the assays described above.

The ELISA SARS-CoV-2 Nucleoprotein IgG (N-Protein) assay will be used to test for antibodies to the N-protein as an indicator of previous COVID-19 infection during the course of the study. This assay will return a result of negative or positive for previous COVID-19 infection. The result may be used in subgroup analyses.

For the pseudovirus neutralization assay, an ANCOVA model will be implemented to obtain estimates of the treatment group effect adjusted for prior infection status (determined by the N-Protein assay or self-report),  $log_{10}$  of baseline antibody titers, and age group. A  $log_{10}$  transformation will be applied to the dependent variable, which will be antibody titers, to obtain the treatment effect estimates as ratios of each treatment

group relative to the prototype treatment arm. The ANCOVA model will be applied to all immunogenicity study time points in single dose arms. Estimates and 95% CIs will be reported for the treatment group effects, and a Bonferroni adjustment will be applied to adjust the CIs for the number of treatment group comparisons. The model will be estimated for the mITT population as well as the subsample of the mITT population of subjects who do not have a history of COVID-19 infection, as determined by the N-Protein assay or self report. When the model is applied to the sample of uninfected subjects, prior infection status will not be included as a covariate (Table 339, Table 340, Table 341, and Table 342).

Correlations between the results from samples tested at different labs (e.g. PsVNA) may be calculated to evaluate the consistency of results across testing facilities.

Individual immunogenicity responses are shown in Listing 8.

# 8.2. Secondary Immunogenicity Analyses

See Section 9 for safety analyses which are the secondary endpoints of this study.

# 8.3. Exploratory Immunogenicity/Efficacy Analyses

#### **8.3.1.** T-cells

The magnitude, phenotype and percentage of cytokine expressing S protein specific T cells will be summarized at selected timepoints by vaccination group. Mean percentages of CD4 and CD8 T cells expressing cytokines and proportions of responders with 95% CI, along with median, minimum, and maximum, will be presented by peptide pool stimulation (starting with Table 343 and ending with Table 414). Distributions of T cell percentages will be graphically displayed (starting with Figure 650 and ending with Figure 757).

Individual T-cell responses are shown in Listing 9.

#### 8.3.2. B-cells

Antigen-specific memory B cells were defined as CD3, CD8, CD14, CD16, and CD56 negative, but CD19, CD20, CD27, IgG or IgA (both on the same color) positive, and positive for one or more of WT or SA RBD, NTD (both variants on a single color) or S-2P. Longitudinal timepoints from each study participant were analyzed as a unit to mitigate batch effects and allow internal normalization to each individual's baseline sample. Median percentages of antigen specific B-cells along with min, max, median fold rise, and min and max of fold rise will be presented by probe (starting with Table 415 and ending with Table 450). Distributions of B cell percentages will be graphically displayed (starting with Figure 758 and ending with Figure 1009.

Individual B-cell responses are shown in Listing 10.

#### 8.3.3. Breakthrough Infections

Confirmed SARS-CoV-2 infection at any time during the study, defined as a positive RT-PCR test performed by the site or using a non-site testing method (RT-PCR or antigen test) or N-antibody positive at a visit, will be documented as an exploratory efficacy assessment. Kaplan-Meier curves and 95% confidence intervals of infection free survival will be calculated (starting with Figure 1010 and ending with Figure 1018). Time to infection restricted mean survival time analyses will also be reported (starting with Table 451 and ending with Table 459).

#### 8.3.4. Sequencing Results of Breakthrough Infections

The Simon and Bakel labs at the Icahn School of Medicine at Mount Sinai will analyze nasopharyngeal swab specimens collected from participants who experienced a SARS-CoV-2 breakthrough infection. The analysis aims to provide data on SARS-CoV-2 copy numbers and SARS-CoV-2 genotype/lineage.

The SARS-CoV-2 breakthrough positive nasopharyngeal specimens will be provided either as a dry swab or resuspended in viral transport media (both specimen types cryo-preserved at –80C). Biospecimen will be accessioned and processed according to the SOPs developed in collaboration with Dr. Greninger [42]. Briefly, each specimen undergoesRNA extraction, Reverse Transcriptase quantitative real time PCR (RT qPCR) and cDNA synthesis, whole-genome amplification followed by library preparation and next generation Illumina sequencing if the amount of SARS-CoV-2 passes the minimum requirements (e.g., less than threshold cycle 32). SARS-CoV-2 genomes will be assembled and subjected to quality control using the lab's custom vRAPID pipeline [43]. Genomes with at least 95% coverage and 100X depth across all regions will be considered complete. Genotypic analysis and clade/lineage assignment of complete genomes will be performed using the Nextclade CLI (v2.13.1), pangolin (v2.4) and pangoLEARN (v1.19) pipelines. Samples will be traced to their ancestral lineage assignments by obtaining the first letter and first numerical character of the lineage aliases provided by Nextclade.

A summary of variant PANGO calls are provided starting at Table 460 and ending at Table 468. A visual summary is provided starting at Figure 1019 and ending at Figure 1024.

Individual sequencing results are shown in Listing 11.

Further details on the analyses of exploratory endpoints will be described in an addendum to the Statistical Analysis Plan.

#### 9. SAFETY EVALUATION

Summaries and analysis of safety data will be presented for the Safety Analysis Population.

Solicited non serious AEs will be collected from the time of each vaccination until 7 days after. Solicited AEs will be summarized by severity for each day post each vaccination and as the maximum severity over all 8 days. Additionally, solicited AEs will be analyzed using standard techniques, such as 95% CIs (using the Clopper-Pearson method), to summarize the proportion of subjects reporting each symptom, any application site symptom, and any systemic symptom.

Unsolicited non-serious AEs will be collected from the time of first vaccination through 28 days after each vaccination. Unsolicited AEs will be coded by MedDRA for preferred term and system organ class (SOC). SAEs, MAAEs, NOCMCs, AESIs, and AEs leading to withdrawal from the study will be collected from the time of first vaccination through 12 months after the last vaccine dose. The numbers of SAEs, MAAEs, NOCMCS, AESIs, and AEs leading to withdrawal from the study will be reported by detailed listings showing the event description, MedDRA preferred term and SOC, relevant dates (vaccinations and AEs), severity, relatedness, and outcome for each event. Non-serious unsolicited AEs will be summarized as number and percentage of subjects reporting at least one event in each MedDRA preferred term and SOC, cross tabulated by severity and relationship to study product. Additionally, the proportion of subjects and 95% CIs of AEs in aggregate and by MedDRA categories will be computed.

#### 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, race, time from first booster, time since covid infection, time since 1<sup>st</sup> booster or covid infection, and prior infection status (by self-report, N-Protein, either) will be presented by vaccination group (Table 12 and Table 13). Ethnicity is categorized as Hispanic or LatinX, or not Hispanic and not LatinX. In accordance with NIH reporting policy, subjects may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option.

Individual subject listings (Appendix 3) will be presented for all demographics (Listing 6).

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 23.0 or higher.

Summaries of subjects' pre-existing medical conditions will be presented by vaccination group (Table 14). Individual subject listings will be presented for all medical conditions (Listing 7).

#### 9.1.2. Prior and Concomitant Medications

Summaries of medications that were started prior to dosing and continuing at the time of dosing will be presented by WHO Drug Terms 2 and 3 and treatment group (Table 486).

Individual subject listings will be presented for all concomitant medications (Listing 17).

# 9.2. Measurements of Treatment Compliance

All subjects are to receive one or two doses of study product administered in the clinic. The number of subjects receiving each dose will be summarized as part of the subject disposition table (Table 9).

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per subject basis), each subject will only be counted once and any repetitions of adverse events within a subject will be ignored; the denominator will be the total population size. All adverse events reported will be included in the summaries and analyses.

#### 9.3.1. Solicited Events and Symptoms

Systemic solicited adverse events were collected pre-vaccination, and systemic and local solicited adverse events were collected 30 minutes post-vaccination and then daily for 7 days after each vaccination and graded on a scale of 0 (absent), 1 (mild), 2 (moderate) and 3 (severe). Systemic events include fatigue, headache, myalgia, and fever. Local events include pain at injection site, erythema, and induration.

The proportion of subjects reporting at least one solicited adverse event will be summarized for each solicited adverse event, any systemic symptom, any local symptom, and any symptoms. The 95% CI will be calculated using the Clopper-Pearson method (Table 470, Table 471, Table 472, Figure 1025, and Figure 1026).

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the Safety population. The number and percentage of subjects reporting each event will be summarized by the maximum severity and treatment group, separately for each vaccination and over all vaccinations. For each event the denominator is the number of subjects with non-missing data for the specific event (Table 471, Table 472, Figure 1025, and Figure 1026).

The number of subjects reporting a solicited adverse event will be summarized for each day post vaccination for each vaccination and for all vaccinations combined both in a summary table (Table 473, Table 474, Table 475, Table 476, Table 477, Table 478) and graphically in a bar chart (Figure 1027 and Figure 1028).

The mean, standard deviation, median, minimum, and maximum duration of solicited events will be summarized (Table 479). Day of solicited symptom onset will be summarized graphically (Figure 1029, Figure 1030, Figure 1031, Figure 1032)

Solicited adverse events by subject will be presented in Listing 9 and Listing 10, and graphically starting with Figure 1033 and ending with Figure 1044.

#### 9.3.2. Unsolicited Adverse Events

Unsolicited AEs will be collected until 28 days after each vaccination. The proportion of subjects reporting at least one unsolicited adverse event will be summarized by MedDRA system organ class and preferred term for each vaccination and over all vaccinations. Denominators for percentages are the number of subjects who received the vaccination being summarized.

Adverse events by subject will be presented in Listing 14.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, vaccination, and treatment group:

- Summary of severity and relationship to study product (Table 480, Table 481, and Table 482);
- Subject listing of non-serious adverse events of moderate or greater severity (Table 484);
- Bar charts of incidence and frequency of adverse events by severity and MedDRA system organ class (Figure 1045 and Figure 1046).

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Subject ID, Age (years) Adverse Event Description, Adverse Event Onset Date/End Date, Last Dose Received/Days Post Dose, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 483);
- Adverse Events of Special Interest (Table 485);
- New Onset Chronic Medical Conditions and Medically Attended Adverse Events (Table 485).

### 9.5. Pregnancies

For any subjects in the Safety population who became pregnant during the study, every attempt was made to follow these subjects to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. In addition, a listing of pregnancies and outcomes will be presented (Listing 18, Listing 19, Listing 20, Listing 21, and Listing 22).

#### 9.6. Clinical Laboratory Evaluations

Not applicable.

# 9.7. Vital Signs and Physical Evaluations

Vital sign measurements included systolic blood pressure, diastolic blood pressure and oral temperature. Vital signs were assessed at screening visit and Day 1 (Listing 15).

Physical Examinations performed at screening visit and Day 1 (Listing 16).

There are no planned vital sign measurements or physical examinations for follow-up visits. No tabulations will be made.

#### 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-subject listing of concomitant medication use will be presented (Listing 17). The use of concomitant medications during the study will be summarized by ATC1, ATC2 code and treatment group for the Safety population (Table 486).

# 9.9. Other Safety Measures

Not applicable.

# 10. PHARMACOKINETICS

Not applicable.

# 11. IMMUNOGENICITY

See Section 8.
#### **12. OTHER ANALYSES**

Not applicable.

#### 13. REPORTING CONVENTIONS

The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

### 14. TECHNICAL DETAILS

SAS version 9.4 and R 3.6.2 or above will be used to generate all tables, figures, and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

ANCOVA models were added to compare vaccination groups to prototype.

An analysis of breakthrough infections was also added that includes Kaplan-Meier Curves and restricted mean survival time.

An analysis of geometric mean fold drop was added.

#### 16. REFERENCES

- 1. WHO. World Health Organization, Weekly Operational Update on COVID-19.
- 2. JHU. JHU. -19 Dashboard, Center for Systems Science and Engineering (CCSE) at Johns Hopkins University (JHU).
- 3. Corbett KS, Edwards DK, Leist SR, et al. SARS-CoV-2 mRNA vaccine design enabled by prototype pathogen preparedness. Nature 2020;586:567-71.
- 4. Bos R, Rutten L, van der Lubbe JEM, et al. Ad26 vector-based COVID-19 vaccine encoding a prefusion-stabilized SARS-CoV-2 Spike immunogen induces potent humoral and cellular immune responses. NPJ Vaccines 2020;5:91.
- 5. Dunkle LM, Kotloff KL, Gay CL, et al. Efficacy and Safety of NVX-CoV2373 in Adults in the United States and Mexico. N Engl J Med 2022;386:531-43.
- 6. Heath PT, Galiza EP, Baxter DN, et al. Safety and Efficacy of NVX-CoV2373 Covid-19 Vaccine. N Engl J Med 2021;385:1172-83.
- 7. Falsey AR, Sobieszczyk ME, Hirsch I, et al. Phase 3 Safety and Efficacy of AZD1222 (ChAdOx1 nCoV-19) Covid-19 Vaccine. N Engl J Med 2021;385:2348-60.
- 8. CDC. COVID Vaccine Tracker. https://covidcdcgov/covid-data-tracker/#vaccinations\_vacc-total-admin-rate-total;Accessed February 13, 2022.
- 9. Britton A, Jacobs Slifka KM, Edens C, et al. Effectiveness of the Pfizer-BioNTech COVID-19 Vaccine Among Residents of Two Skilled Nursing Facilities Experiencing COVID-19 Outbreaks Connecticut, December 2020-February 2021. MMWR Morb Mortal Wkly Rep 2021;70(11):396-401. DOI: 10.15585/mmwr.mm7011e3
- 10. Chemaitelly H, Tang P, Hasan MR, et al. Waning of BNT162b2 Vaccine Protection against SARS-CoV-2 Infection in Qatar. N Engl J Med 2021;385:e83.
- 11. Israel A, Merzon E, Schaffer AA, et al. Elapsed time since BNT162b2 vaccine and risk of SARS-CoV-2 infection: test negative design study. BMJ 2021;375:e067873.
- 12. Goldberg Y, Mandel M, Bar-On YM, et al. Waning Immunity after the BNT162b2 Vaccine in Israel. N Engl J Med 2021;385:e85.
- 13. Tegally H, Wilkinson E, Giovanetti M, et al. Detection of a SARS-CoV-2 variant of concern in South Africa. Nature 2021;592:438-43.
- 14. Di Giacomo S, Mercatelli D, Rakhimov A, Giorgi FM. Preliminary report on severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) Spike mutation T478K. J Med Virol 2021;93:5638-43.
- 15. Organization WH. Enhancing Readiness for Omicron (B.1.1.529): Technical Brief and Priority Actions for Member States. December 10, 2021.
- 16. Barda N, Dagan N, Cohen C, et al. Effectiveness of a third dose of the BNT162b2 mRNA COVID-19 vaccine for preventing severe outcomes in Israel: an observational study. Lancet 2021;398:2093-100.
- 17. Bar-On YM, Goldberg Y, Mandel M, et al. Protection against Covid-19 by BNT162b2 Booster across Age Groups. N Engl J Med 2021;385:2421-30.

- 18. Patalon T, Gazit S, Pitzer VE, Prunas O, Warren JL, Weinberger DM. Odds of Testing Positive for SARS-CoV-2 Following Receipt of 3 vs 2 Doses of the BNT162b2 mRNA Vaccine. JAMA Intern Med 2022;182:179-84.
- 19. Atmar RL, Lyke KE, Deming ME, et al. Homologous and Heterologous Covid-19 Booster Vaccinations. N Engl J Med 2022.
- 20. Miller J. Safety and Immunogenicity of a 50 μg Booster Dose of Moderna COVID-19 Vaccine. Presented at the ACIP Oct 21, 2021. .
- 21. Pajon R, Doria-Rose NA, Shen X, et al. SARS-CoV-2 Omicron Variant Neutralization after mRNA-1273 Booster Vaccination. N Engl J Med 2022.
- 22. Choi A, Koch M, Wu K, et al. Safety and immunogenicity of SARS-CoV-2 variant mRNA vaccine boosters in healthy adults: an interim analysis. Nat Med 2021;27:2025-31.
- 23. Sridhar S, Joaquin A, Bonaparte MI, et al. Safety and immunogenicity of an AS03-adjuvanted SARS-CoV-2 recombinant protein vaccine (CoV2 preS dTM) in healthy adults: interim findings from a phase 2, randomised, dose-finding, multicentre study. Lancet Infect Dis 2022;22(5):636-648. DOI: 10.1016/S1473-3099(21)00764-7.
- 24. Sanofi/GSK. Sanofi and GSK to seek regulatory authorization for COVID-19 vaccine. 2022.
- 25. Regev-Yochay G, Gonen T, Gilboa M, et al. Efficacy of a Fourth Dose of Covid-19 mRNA Vaccine against Omicron. N Engl J Med 2022.
- 26. Arbel R, Sergienko R, Friger M, Peretz A. Second Booster Vaccine and Covid-19 Mortality in Adults 60 to 100 Years Old. Research Square2022.
- 27. Gazit S, Saciuk Y, Perez G, Peretz A, Pitzer V, Patalon T. Relative Effectiveness of Four Doses Compared to Three Dose of the BNT162b2 Vaccine in Israel. medRxiv2022.
- 28. Shen X, Tang H, McDanal C, et al. SARS-CoV-2 variant B.1.1.7 is susceptible to neutralizing antibodies elicited by ancestral Spike vaccines. bioRxiv 2021.
- 29. Callaway E, Mallapaty S. Novavax offers first evidence that COVID vaccines protect people against variants. Nature 2021;590:17.
- 30. Wang P, Nair MS, Liu L, et al. Antibody resistance of SARS-CoV-2 variants B.1.351 and B.1.1.7. Nature 2021;593:130-5.
- 31. Muik A, Lui BG, Wallisch AK, et al. Neutralization of SARS-CoV-2 Omicron by BNT162b2 mRNA vaccine-elicited human sera. Science 2022;375:678-80.
- 32. Cele S, Jackson L, Khoury DS, et al. Omicron extensively but incompletely escapes Pfizer BNT162b2 neutralization. Nature 2022;602:654-6.
- 33. Nemet I, Kliker L, Lustig Y, et al. Third BNT162b2 Vaccination Neutralization of SARSCoV-2 Omicron Infection. N Engl J Med 2022;386(5):492-494. DOI:10.1056/NEJMc2119358
- 34. Pavot V, Berry C, Kishko M, et al. Protein-based SARS-CoV-2 spike vaccine booster increases cross-neutralization against SARS-CoV-2 variants of concern in non-human primates. Nat Commun 2022;13(1):1699. DOI: 10.1038/s41467-022-29219-2.
- 35. van der Straten K, Guerra D, van Gils MJ, et al. Mapping the antigenic diversification of SARS-CoV-2. medRxiv 2022:2022.01.03.21268582. DOI: 10.1101/2022.01.03.21268582.

- 36. Jones JM, Stone M, Sulaeman H, et al. Estimated US Infection- and Vaccine-Induced SARSCoV-2 Seroprevalence Based on Blood Donations, July 2020-May 2021. JAMA 2021;326(14):1400-1409. DOI: 10.1001/jama.2021.15161.
- 37. Guidelines CCVB. https://www.cdc.gov/coronavirus/2019-ncov/vaccines/boostershot.html?s\_cid=11737:cdc covid booster shot guidelines:sem.ga:p:RG:GM:gen:PTN:FY22.Accessed February 13, 2022.
- 38. Munro APS, Janani L, Cornelius V, et al. Safety and immunogenicity of seven COVID-19 vaccines as a third dose (booster) following two doses of ChAdOx1 nCov-19 or BNT162b2 in the UK (COV-BOOST): a blinded, multicentre, randomised, controlled, phase 2 trial. Lancet 2021;398(10318):2258-2276. DOI: 10.1016/S0140-6736(21)02717-3
- 39. Hause AM, Baggs J, Marquez P, Myers TR. Safety Monitoring of COVID-19 Vaccine Booster Doses Among Adults United States, September 22, 2021–February 6, 2022. MMWR Morb Mortal Wkly Rep 2022. DOI: http://dx.doi.org/10.15585/mmwr.mm7107e1.
- 40. Pfizer asks FDA to greenlight new omicron booster shots, which could arrive this fall. NPR. (https://www.npr.org/sections/health-shots/2022/08/22/1118788439/vaccine-maker-asks-fdato-greenlight-updated-omicron-booster-shot).
- 41. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.
- 42. "Polyester nasal swabs collected in a dry tube are a robust and inexpensive, minimal self-collection kit for SARS-CoV-2 testing." Padgett LR, Kennington LA, Ahls CL, Samarasinghe DK *et al.* PLoS One. 2021 Apr 14;16(4):e0245423. doi: 10.1371/journal.pone.0245423. eCollection 2021. PMID: 33852576
- 43. "vRAPID: Virus Reference-based Assembly Pipeline and IDentification" Zain Khalil, Mitch Sullivan, Ana S. Gonzalez-Reiche, Ajay Obla *et al.* (1.0.0) Zenodo. 2023 https://doi.org/10.5281/zenodo.7829342

## 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3. Note, shells are shown only for stage 1 as examples. Tables, figures and listings will be presented for each stage in the CSRs.

## **APPENDICES**

## APPENDIX 1. TABLE MOCK-UPS

## LIST OF TABLES

| Table 1: | Objectives and Endpoints (Outcome Measures) | 13 |
|---|---|---|
| Table 2: | Study Design | 81 |
| Table 3: | Schedule of Study Procedures - Single Dose | 82 |
| Table 4: | Schedule of Study Procedures - 2 Doses | 84 |
| Table 5: | Probability of observing one or more Adverse Events for various event rates in one vaccine group (or strata) | 87 |
| Table 6: | Two-sided 95% confidence intervals based on observing a particular average log <sub>e</sub> -antibody titer in subjects' vaccine groups and potential strata sizes | 87 |
| Table 7: | Distribution of Protocol Deviations by Category, Type, and Treatment Group | 89 |
| Table 8: | Distribution of Major Protocol Deviations by Category, Type, and Treatment Group | 90 |
| Table 9: | Subject Disposition by Treatment Group | 93 |
| Table 10: | Analysis Populations by Treatment Group | 94 |
| Table 11: | Ineligibility Summary of Screen Failures | 95 |
| Table 12: | Summary of Categorical Demographic and Baseline Characteristics by<br>Treatment Group, All Enrolled Subjects | 96 |
| Table 13: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects | 98 |
| Table 14: | Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group | 100 |
| Table 15: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Overall – mITT Population | 101 |
| Table 16: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Overall – Per<br>Protocol Population | 103 |
| Table 17: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Younger<br>Cohort – mITT Population | 103 |
| Table 18: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Younger<br>Cohort – Per Protocol Population | 103 |
| Table 19: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Summary Results by Time Point and Variant, Prototype, Older Cohort – mITT Population | 103 |

| Table 20: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Older Cohort<br>– Per Protocol Population | .103 |
|---|---|---|
| Table 21: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Infected (by<br>Self-Report or N-protein) Cohort – mITT Population | .103 |
| Table 22: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Infected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population | .103 |
| Table 23: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Uninfected (by<br>Self-Report or N-protein) Cohort – mITT Population | .104 |
| Table 24: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Uninfected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population | .104 |
| Table 25: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Younger<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | .104 |
| Table 26: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Younger<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .104 |
| Table 27: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .104 |
| Table 28: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .104 |
| Table 29: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Older Infected<br>(by Self-Report or N-protein) Cohort – mITT Population | .104 |
| Table 30: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Older Infected<br>(by Self-Report or N-protein) Cohort – Per Protocol Population | .104 |
| Table 31: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Older<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .104 |
| Table 32: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Prototype, Older<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .104 |

| Table 33: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Overall – mITT Population | 104 |
|---|---|---|
| Table 34: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Overall – Per Protocol Population | 104 |
| Table 35: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Cohort – mITT Population | 104 |
| Table 36: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Cohort – Per Protocol Population | 104 |
| Table 37: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Older Cohort – mITT Population | 105 |
| Table 38: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Older Cohort – Per Protocol Population | 105 |
| Table 39: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 105 |
| Table 40: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 105 |
| Table 41: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 105 |
| Table 42: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 105 |
| Table 43: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 105 |
| Table 44: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 105 |
| Table 45: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – mITT<br>Population | 105 |

| Table 46: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 105 |
|---|---|---|
| Table 47: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Older Infected (by Self-Report or N-protein) Cohort – mITT Population | |
| Table 48: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 105 |
| Table 49: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 105 |
| Table 50: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron,<br>Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 106 |
| Table 51: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Overall<br>– mITT Population | 106 |
| Table 52: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Overall<br>- Per Protocol Population | 106 |
| Table 53: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron,<br>Younger Cohort – mITT Population | 106 |
| Table 54: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron,<br>Younger Cohort – Per Protocol Population | 106 |
| Table 55: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Older<br>Cohort – mITT Population | 106 |
| Table 56: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Older<br>Cohort – Per Protocol Population | 106 |
| Table 57: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | |

| Table 58: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population106 |
|---|---|
| Table 59: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron,<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 60: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population106 |
| Table 61: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population106 |
| Table 62: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population |
| Table 63: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 64: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population |
| Table 65: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Older<br>Infected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 66: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Older<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population107 |
| Table 67: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 68: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Delta + Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population107 |
| Table 69: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Summary Results by Time Point and Variant, Omicron, Overall–mITT Population |

| Table 70: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Overall – Per<br>Protocol Population |
|---|---|
| Table 71: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Younger<br>Cohort – mITT Population |
| Table 72: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Younger<br>Cohort – Per Protocol Population |
| Table 73: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Older Cohort –<br>mITT Population |
| Table 74: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Older Cohort –<br>Per Protocol Population |
| Table 75: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Infected (by<br>Self-Report or N-protein) Cohort – mITT Population |
| Table 76: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Infected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population |
| Table 77: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Uninfected (by<br>Self-Report or N-protein) Cohort – mITT Population |
| Table 78: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Uninfected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population |
| Table 79: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Younger<br>Infected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 80: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Younger<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population108 |
| Table 81: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population108 |
| Table 82: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population108 |

| Table 83: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 108 |
|---|---|---|
| Table 84: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 108 |
| Table 85: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 108 |
| Table 86: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 108 |
| Table 87: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Overall– mITT Population | 108 |
| Table 88: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Overall– Per Protocol Population | 108 |
| Table 89: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Younger Cohort – mITT Population | |
| Table 90: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Younger Cohort – Per Protocol Population | 108 |
| Table 91: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Older Cohort – mITT Population | 108 |
| Table 92: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Older Cohort – Per Protocol Population | 108 |
| Table 93: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 109 |
| Table 94: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 109 |
| Table 95: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |

| Table 96: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 109 |
|---|---|---|
| Table 97: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 109 |
| Table 98: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 109 |
| Table 99: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – mITT<br>Population | 109 |
| Table 100: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 109 |
| Table 101: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 109 |
| Table 102: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, Omicron + Prototype,<br>Older Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 109 |
| Table 103: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 109 |
| Table 104: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 109 |
| Table 105: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Overall – mITT Population | 110 |
| Table 106: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Overall– Per Protocol Population | 113 |
| Table 107: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population | 113 |

| Table 108: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Cohort – Per Protocol Population |
|---|---|
| Table 109: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Older Cohort – mITT Population |
| Table 110: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Older Cohort – Per Protocol Population |
| Table 111: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 112: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population113 |
| Table 113: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population114 |
| Table 114: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population114 |
| Table 115: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population114 |
| Table 116: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population |
| Table 117: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – mITT<br>Population |
| Table 118: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population |
| Table 119: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Older Infected (by Self-Report or N-protein) Cohort – mITT Population114 |
| Table 120: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, |

| | Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 114 |
|---|---|---|
| Table 121: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 114 |
| Table 122: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron,<br>Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 114 |
| Table 123: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall – mITT Population | 115 |
| Table 124: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall – Per Protocol Population | 117 |
| Table 125: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort – mITT Population | 117 |
| Table 126: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort – Per Protocol Population | 117 |
| Table 127: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort – mITT Population | 117 |
| Table 128: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort – Per Protocol Population | 117 |
| Table 129: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 117 |
| Table 130: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 117 |
| Table 131: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 118 |
| Table 132: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 118 |
| Table 133: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 118 |
| Table 134: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |

| Table 135: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 118 |
|---|---|---|
| Table 136: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 118 |
| Table 137: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population. | 118 |
| Table 138: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 118 |
| Table 139: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 118 |
| Table 140: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 118 |
| Table 141: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall– mITT Population | 118 |
| Table 142: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population | 118 |
| Table 143: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – mITT Population | 118 |
| Table 144: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 118 |
| Table 145: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – mITT Population | 118 |
| Table 146: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 118 |
| Table 147: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 118 |
| Table 148: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 119 |
| Table 149: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 119 |

| Table 150: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 119 |
|---|---|---|
| Table 151: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 119 |
| Table 152: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 119 |
| Table 153: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 119 |
| Table 154: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 119 |
| Table 155: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 119 |
| Table 156: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 119 |
| Table 157: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 119 |
| Table 158: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 119 |
| Table 159: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall– mITT Population | |
| Table 160: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall – Per Protocol Population | 119 |
| Table 161: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort – mITT Population | 119 |
| Table 162: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort – Per Protocol Population | 119 |
| Table 163: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort – mITT Population | 120 |
| Table 164: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort – Per Protocol Population | 120 |

| Table 165: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 120 |
|---|---|---|
| Table 166: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 120 |
| Table 167: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 120 |
| Table 168: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 120 |
| Table 169: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 120 |
| Table 170: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 120 |
| Table 171: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 120 |
| Table 172: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 120 |
| Table 173: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 120 |
| Table 174: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 120 |
| Table 175: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 120 |
| Table 176: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 120 |
| Table 177: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Overall– mITT Population | 120 |
| Table 178: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Overall – Per Protocol Population | 121 |

| Table 179: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort – mITT Population | 121 |
|---|---|---|
| Table 180: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort – Per Protocol Population | 121 |
| Table 181: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort – mITT Population | 121 |
| Table 182: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort – Per Protocol Population | 121 |
| Table 183: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 121 |
| Table 184: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 121 |
| Table 185: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 121 |
| Table 186: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 121 |
| Table 187: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 121 |
| Table 188: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 121 |
| Table 189: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 121 |
| Table 190: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 121 |
| Table 191: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 121 |
| Table 192: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 121 |

| Table 193: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 121 |
|---|---|---|
| Table 194: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 121 |
| Table 195: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall – mITT Population | 121 |
| Table 196: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall – Per Protocol Population | 122 |
| Table 197: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort – mITT Population | 122 |
| Table 198: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort – Per Protocol Population | 122 |
| Table 199: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population | 122 |
| Table 200: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort – Per Protocol Population | 122 |
| Table 201: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 122 |
| Table 202: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 122 |
| Table 203: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 122 |
| Table 204: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 122 |
| Table 205: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 122 |
| Table 206: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Table 207: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 122 |

| Table 208: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .122 |
|---|---|---|
| Table 209: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | .122 |
| Table 210: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .122 |
| Table 211: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .123 |
| Table 212: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .123 |
| Table 213: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population | .124 |
| Table 214: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population | .127 |
| Table 215: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population | .127 |
| Table 216: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | .127 |
| Table 217: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population | .127 |
| Table 218: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population | .127 |
| Table 219: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | .127 |
| Table 220: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .127 |
| Table 221: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .128 |
| Table 222: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .128 |

| Table 223: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 128 |
|---|---|---|
| Table 224: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 128 |
| Table 225: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 128 |
| Table 226: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 128 |
| Table 227: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 128 |
| Table 228: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 128 |
| Table 229: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 128 |
| Table 230: | Pseudovirus Neutralization Assay ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 128 |
| Table 231: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall – mITT Population | 129 |
| Table 232: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall–Per Protocol Population | 131 |
| Table 233: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort – mITT Population | 131 |
| Table 234: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort – Per Protocol Population | 131 |
| Table 235: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort – mITT Population | 131 |
| Table 236: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort – Per Protocol Population | 131 |
| Table 237: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 131 |

| Table 238: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 131 |
|---|---|---|
| Table 239: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 131 |
| Table 240: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 131 |
| Table 241: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 131 |
| Table 242: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 132 |
| Table 243: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 132 |
| Table 244: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 132 |
| Table 245: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 132 |
| Table 246: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 132 |
| | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 132 |
| Table 248: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 132 |
| Table 249: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall – mITT Population | 132 |
| Table 250: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall – Per Protocol Population | 132 |
| Table 251: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – mITT Population | 132 |

| Table 252: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 132 |
|---|---|---|
| Table 253: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – mITT Population | 132 |
| Table 254: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 132 |
| Table 255: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 132 |
| Table 256: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 132 |
| Table 257: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 132 |
| Table 258: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 133 |
| Table 259: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 133 |
| Table 260: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 133 |
| Table 261: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 133 |
| Table 262: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 133 |
| Table 263: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 133 |
| Table 264: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |

| Table 265: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 133 |
|---|---|---|
| Table 266: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 133 |
| Table 267: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall – mITT Population | 133 |
| Table 268: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall – Per Protocol Population | 133 |
| Table 269: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort – mITT Population | 133 |
| Table 270: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort – Per Protocol Population | 133 |
| Table 271: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort – mITT Population | 133 |
| Table 272: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort – Per Protocol Population | 133 |
| Table 273: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 134 |
| Table 274: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 134 |
| Table 275: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 134 |
| Table 276: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 134 |
| Table 277: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 134 |
| Table 278: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 134 |
| Table 279: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 134 |

| Table 280: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 134 |
|---|---|---|
| Table 281: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 134 |
| Table 282: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 134 |
| Table 283: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 134 |
| Table 284: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 134 |
| Table 285: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Overall – mITT Population | 134 |
| Table 286: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Overall – Per Protocol Population | 134 |
| Table 287: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort – mITT Population | 134 |
| Table 288: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort – Per Protocol Population | 135 |
| Table 289: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort – mITT Population | 135 |
| Table 290: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort – Per Protocol Population | 135 |
| Table 291: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 135 |
| Table 292: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 135 |
| Table 293: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 135 |
| Table 294: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 135 |

| Table 295: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 135 |
|---|---|---|
| Table 296: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 135 |
| Table 297: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 135 |
| Table 298: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 135 |
| Table 299: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 135 |
| Table 300: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 135 |
| Table 301: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 135 |
| Table 302: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 135 |
| Table 303: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall – mITT Population | 135 |
| Table 304: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall – Per Protocol Population | 135 |
| Table 305: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort – mITT Population | 135 |
| Table 306: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort – Per Protocol Population | 136 |
| Table 307: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population | 136 |
| Table 308: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort – Per Protocol Population | 136 |
| Table 309: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 136 |

| Table 310: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 136 |
|---|---|---|
| Table 311: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 136 |
| Table 312: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 136 |
| Table 313: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 136 |
| Table 314: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 136 |
| Table 315: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 136 |
| Table 316: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 136 |
| Table 317: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 136 |
| Table 318: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 136 |
| Table 319: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Table 320: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 136 |
| Table 321: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population | |
| Table 322: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population | 140 |
| Table 323: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population | 140 |

| Table 324: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 140 |
|---|---|---|
| Table 325: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population | 140 |
| Table 326: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 140 |
| Table 327: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 140 |
| Table 328: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 140 |
| Table 329: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 140 |
| Table 330: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 141 |
| Table 331: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 141 |
| Table 332: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 141 |
| Table 333: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 141 |
| Table 334: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 141 |
| Table 335: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 141 |
| Table 336: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |

| Table 337: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 141 |
|---|---|---|
| Table 338: | Focus Reduction Neutralization Test ID <sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 141 |
| <b>Table 339</b> : | Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Overall – mITT Population. | 142 |
| <b>Table 340</b> : | Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Overall – Per Protocol Population | 143 |
| <b>Table 341</b> : | Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Uninfected (by Self-Report or N-Protein) Cohort – mITT Population | 143 |
| <b>Table 342</b> : | Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Uninfected (by Self-Report or N-Protein) Cohort – Per Protocol Population | 143 |
| Table 343: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Overall – mITT Population | 144 |
| Table 344: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1<br>Dose Groups, Overall – Per Protocol Population | 152 |
| Table 345: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1<br>Dose Groups, Older Cohort – mITT Population | 152 |
| Table 346: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1<br>Dose Groups, Older Cohort – Per Protocol Population | 152 |
| Table 347: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1<br>Dose Groups, Younger Cohort – mITT Population | 152 |
| Table 348: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Cohort – Per Protocol Population | 152 |
| Table 349: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein) Cohort – mITT Population | 153 |
| Table 350: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 153 |
| Table 351: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 153 |

| Table 352: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 153 |
|---|---|---|
| Table 353: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1<br>Dose Groups, Older Infected (by Self-Report or N-protein) Cohort – mITT<br>Population | 153 |
| Table 354: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 153 |
| Table 355: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 153 |
| Table 356: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 153 |
| Table 357: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 153 |
| Table 358: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 153 |
| Table 359: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 153 |
| Table 360: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 153 |
| Table 361: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall – mITT Population | 154 |
| Table 362: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall – Per Protocol Population | 161 |
| Table 363: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort – mITT Population | 161 |
| Table 364: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort – Per Protocol Population | 161 |
| Table 365: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort – mITT Population | 161 |
| Table 366: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort – Per Protocol Population | 161 |
| Table 367: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein) Cohort – mITT Population | 161 |
|---|---|---|
| Table 368: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 161 |
| Table 369: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 161 |
| Table 370: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 161 |
| Table 371: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 162 |
| Table 372: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 162 |
| Table 373: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 162 |
| Table 374: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 162 |
| Table 375: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 162 |
| Table 376: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 162 |
| Table 377: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 162 |
| Table 378: | Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 162 |
| Table 379: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Overall – mITT Population | 163 |
| Table 380: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Overall – Per Protocol Population | 170 |

| Table 381: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Cohort – mITT Population | 170 |
|---|---|---|
| Table 382: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Cohort – Per Protocol Population | 170 |
| Table 383: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Cohort – mITT Population | 170 |
| Table 384: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Cohort – Per Protocol Population | 170 |
| Table 385: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein) Cohort – mITT Population | 170 |
| Table 386: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 170 |
| Table 387: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 170 |
| Table 388: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 170 |
| Table 389: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 170 |
| Table 390: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 170 |
| Table 391: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 170 |
| Table 392: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 170 |
| Table 393: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report) Cohort – mITT Population | 170 |
| Table 394: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 170 |
| Table 395: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 171 |

| Table 396: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 171 |
|---|---|---|
| Table 397: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall – mITT Population | 172 |
| Table 398: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall – Per Protocol Population | 178 |
| Table 399: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort – mITT Population | 178 |
| Table 400: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort – Per Protocol Population | 178 |
| Table 401: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort – mITT Population | 178 |
| Table 402: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort – Per Protocol Population | 178 |
| Table 403: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein) Cohort – mITT Population | 178 |
| Table 404: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 178 |
| Table 405: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 178 |
| Table 406: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 178 |
| Table 407: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 178 |
| Table 408: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 178 |
| Table 409: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 178 |
| Table 410: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 178 |

| Table 411: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 178 |
|---|---|---|
| Table 412: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 178 |
| Table 413: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 179 |
| Table 414: | Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 179 |
| Table 415: | Percent of Total B-cells by timepoint and Vaccination arm, Overall – mITT Population | 180 |
| Table 416: | Percent of Total B-cells by timepoint and Vaccination arm, Overall – Per Protocol Population | 180 |
| Table 417: | Percent of Total B-cells by timepoint and Vaccination arm, Older Cohort – mITT Population | 180 |
| Table 418: | Percent of Total B-cells by timepoint and Vaccination arm, Older Cohort – Per Protocol Population | 180 |
| Table 419: | Percent of Total B-cells by timepoint and Vaccination arm, Younger Cohort – mITT Population | 180 |
| Table 420: | Percent of Total B-cells by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population | 180 |
| Table 421: | Percent of Total B-cells by timepoint and Vaccination arm, Infected (by Self-Report or N-protein) Cohort – mITT Population | 180 |
| Table 422: | Percent of Total B-cells by timepoint and Vaccination arm, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 180 |
| Table 423: | Percent of Total B-cells by timepoint and Vaccination arm, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 181 |
| Table 424: | Percent of Total B-cells by timepoint and Vaccination arm, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 181 |
| Table 425: | Percent of Total B-cells by timepoint and Vaccination arm, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 181 |
| Table 426: | Percent of Total B-cells by timepoint and Vaccination arm, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 181 |
| Table 427: | Percent of Total B-cells by timepoint and Vaccination arm, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |

| Table 428: | Percent of Total B-cells by timepoint and Vaccination arm, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population181 |
|---|---|
| Table 429: | Percent of Total B-cells by timepoint and Vaccination arm, Younger<br>Infected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 430: | Percent of Total B-cells by timepoint and Vaccination arm, Younger<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population181 |
| Table 431: | Percent of Total B-cells by timepoint and Vaccination arm, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population181 |
| Table 432: | Percent of Total B-cells by timepoint and Vaccination arm, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population181 |
| Table 433: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Overall – mITT Population |
| Table 434: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Overall – Per Protocol Population |
| Table 435: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Cohort – mITT Population |
| Table 436: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Cohort – Per Protocol Population |
| Table 437: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Younger Cohort – mITT Population |
| Table 438: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Younger Cohort – Per Protocol Population |
| Table 439: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Infected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 440: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population182 |
| Table 441: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population182 |
| Table 442: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population183 |
| Table 443: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Older Infected (by Self-Report or N-protein) Cohort – mITT Population |
| Table 444: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population |
| Table 445: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population183 |

| Table 446: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 183 |
|---|---|---|
| Table 447: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 183 |
| Table 448: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 183 |
| Table 449: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 183 |
| Table 450: | Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 183 |
| Table 451: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Overall – mITT Population | 184 |
| Table 452: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group,<br>Younger Cohort– mITT Population | 184 |
| Table 453: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Older Cohort – mITT Population | 184 |
| Table 454: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group,<br>Infected Cohort (By Self-Report or N-protein) – mITT Population | 184 |
| Table 455: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group,<br>Uninfected Cohort (By Self Report or N-protein) – mITT Population | 185 |
| Table 456: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group,<br>Younger Infected Cohort (By Self-Report or N-protein)—mITT Population | 185 |
| Table 457: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group,<br>Younger Uninfected Cohort (By Self-Report or N-protein)— mITT<br>Population | 185 |
| Table 458: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group,<br>Older Infected Cohort (By Self-Report or N-protein)—mITT Population | 185 |
| Table 459: | Time to Infection Restricted Mean Survival Analysis by Vaccination Group,<br>Older Uninfected Cohort (By Self-Report or N-protein)—mITT Population | 185 |
| Table 460: | Number of Breakthrough Infections by PANGO Call and Treatment Group, Overall – Safety Population | 186 |
| Table 461: | Breakthrough Infections by PANGO Call and Treatment Group, Older Cohort – Safety Population | 188 |
| Table 462: | Breakthrough Infections by PANGO Call and Treatment Group, Younger Cohort – Safety Population | 188 |

| Table 463: | Breakthrough Infections by PANGO Call and Treatment Group, Infected (by Self-Report or N-protein) Cohort – Safety Population | 188 |
|---|---|---|
| Table 464: | Breakthrough Infections by PANGO Call and Treatment Group, Uninfected (by Self-Report or N-protein) Cohort – Safety Population | 188 |
| Table 465: | Breakthrough Infections by PANGO Call and Treatment Group, Older Infected (by Self-Report or N-protein) Cohort – Safety Population | 188 |
| Table 466: | Breakthrough Infections by PANGO Call and Treatment Group, Older Uninfected (by Self-Report or N-protein) Cohort – Safety Population | 188 |
| Table 467: | Breakthrough Infections by PANGO Call and Treatment Group, Younger Infected (by Self-Report) Cohort – Safety Population | 188 |
| Table 468: | Breakthrough Infections by PANGO Call and Treatment Group, Younger Uninfected (by Self-Report or N-protein) Cohort – Safety Population | 188 |
| Table 469: | Overall Summary of Adverse Events by Treatment Group – All Subjects | 189 |
| Table 470: | Serious Adverse Events and Non-Serious Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Safety Population | 191 |
| Table 471: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Post Dose 1 | 192 |
| Table 472: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Two Dose Treatment Group | 195 |
| Table 473: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Prototype | 198 |
| Table 474: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Beta + Omicron | 201 |
| Table 475: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Delta + Omicron | 201 |
| Table 476: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Omicron | 201 |
| Table 477: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Omicron + Prototype | 201 |
| Table 478: | Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Beta+Omicron | 202 |
| Table 479: | Summary of Duration of Solicited Symptoms by Treatment Group - All Subjects | 208 |
| Table 480: | All Adverse Events Cross-Classified by MedDRA System Organ Class,<br>Severity, Relationship to Study Treatment, and Treatment Group | 212 |

| Table 481: | Summary of All Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group | 215 |
|---|---|---|
| Table 482: | Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group | 217 |
| Table 483: | Listing of Serious Adverse Events | 219 |
| Table 484: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 220 |
| Table 485: | Listing of AESIs, MAAEs and NOCMCs | 221 |
| Table 486: | Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group | 226 |

### 9.1 Overall Study Design and Plan Description

**Table 2:** Study Design

| Arms | Vaccine<br>Platform | Samp<br>le<br>Size | Vaccine Candidate | Interval (weeks)* | Timing of First Dose | Timing of<br>Second Dose |
|---|---|---|---|---|---|---|
| | | 100 | Prototype | ≥16 | Dosc<br>D1 | NA |
| | 73 | 100 | Beta + Omicron | <u>≥16</u><br>≥16 | D1 | NA |
| | Moderna<br>RNA-127 | 100 | Beta + Omicron | <u>≥</u> 16 | D1 | D57 |
| | ode<br>VA: | 100 | Delta + Omicron | <u>≥16</u> | D1 | NA |
| | Moderna<br>mRNA-1273 | 100 | Omicron | <u>≥16</u> | D1 | NA |
| | Ξ Ξ | 100 | Omicron + Prototype | <u>≥</u> 16 | D1 | NA |
| | | 50 | W'11 (D + + + ) | >16 | D1 | »T A |
| | . 61 | 50 | Wildtype (Prototype) | ≥16 | D1 | NA |
| | Pfizer/<br>BioNTech<br>BNT162b2 | 50 | Beta + Omicron | ≥16 | D1 | NA |
| | Zel<br>VTC<br>16 | 50 | Omicron | ≥16 | D1 | NA |
| - | F (5) F | 50 | Beta | ≥16 | D1 | NA |
| - | B B | 50 | Beta + Wildtype | ≥16 | D1 | NA |
| | | 50 | Omicron + Wildtype | ≥16 | D1 | NA |
| | eS<br>103 | 50 | Prototype | ≥16 | D1 | NA |
| | fi<br>2 pr<br>-AS | 50 | Beta | ≥16 | D1 | NA |
| | Sanofi<br>CoV2 preS<br>dTM-AS03 | 50 | Beta+ Prototype | ≥16 | D1 | NA |
| | | 100 | Omicron BA.1 + | >16 | D1 | NIA |
| | cer/<br>Tech<br>62b2<br>lent | 100 | Wildtype (Prototype) | ≥16 | וע | NA |
| | Pfizer/<br>BioNTech<br>BNT162b2<br>bivalent | 100 | Omicron BA.4/BA.5 + Wildtype (Prototype) | ≥16 | D1 | NA |

## Two age strata:

- 18-64 years
- $\geq$  65 years (~45% in  $\geq$  65 years).

### Two infection strata:

- Confirmed prior SARS-CoV-2 infection (~20%)
- No known history of prior infection.

<sup>^</sup>For arms 16 and 17 or stage 4, only participants between the ages of 18 to 49 years will be enrolled.

<sup>\*</sup>interval (in weeks) since last exposure to SARS-CoV-2 infection or vaccination

## 9.5.1 Immunogenicity and Safety Measurements Assessed and Flow Chart

**Table 3:** Schedule of Study Procedures - Single Dose

| Study Day | D-28<br>to<br>D-1 | 1 | 4 | 8 <sup>b</sup> | 15 | 29 | 91 | 181 | 271 | 366 | Illness/<br>Unscheduled<br>Visit <sup>k,m</sup> | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 00 <sup>a</sup> | 1 | 1A | 2 | 3 | 4 | 5 | 6 | 7 | 8 | | |
| Window (+/-) | | 0 | 1 | 1 | 2 | 2 | 7 <sup>m</sup> | 14 <sup>m</sup> | 14 <sup>m</sup> | 28 <sup>m</sup> | | |
| Informed Consent <sup>a</sup> | X | | | | | | | | | | | |
| Eligibility Criteria | X | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | |
| Vaccination | | X | | | | | | | | | | |
| Concomitant Meds | X | X | $X^{j}$ | $X^{j}$ | $X^{j}$ | $\mathbf{X}^{\mathrm{j}}$ | $X^{j}$ | $X^{j}$ | X <sup>j</sup> | $X^{j}$ | $X^{j}$ | X <sup>j</sup> |
| Interim History | | X | X | X | X | X | X | X | X | X | X | X |
| Physical Exam <sup>c</sup> - Targeted | X | X | | | | | | | | | (X) | |
| Vital Signs <sup>c</sup> | X | X | | | | | | | | | (X) | |
| Height/Weight (BMI) <sup>a</sup> | X | | | | | | | | | | | |
| Urine β-HCG <sup>d</sup> | X | X | | | | | | | | | | |
| Memory Aid <sup>e</sup> | | X | X | X | | | | | | | | |
| Solicited AEs | | X | X | X | | | | | | | | |
| Unsolicited AEs | | X | X | X | X | X | | | | | | |
| MAAEs, SAEs, NOCMCs, AEs leading to withdrawal from the study and AESIs | | X | X | X | X | X | X | X | X | X | X | X |
| Nasal swab for PCR & Sequencing <sup>f</sup> | | | | | | | | | | | (X) | |
| Assays | | | | | | | | - | | | | |
| Serum for Serological Immunogenicity<br>Assays <sup>g</sup> and Biomarker Testing <sup>1</sup> | | 34 <sup>1</sup> | 4 <sup>1</sup> | | 34 | 34 | 34 | 34 | 34 | 34 | 4 <sup>l</sup> -34 <sup>m</sup> | 34 |
| PBMC Cellular Assays & Plasma <sup>g,h</sup> (select sites only) | | 64-70 | | | 64-70 | | 64-70 | 64-70 | 64-70 | | 64-70 <sup>m</sup> | 64-70 |
| Daily Volume (mL) <sup>g,i</sup> | | 98-<br>104 | 4 | | 98-<br>104 | 34 | 98-<br>104 | 98-<br>104 | 98-<br>104 | 34 | 4-104 | 98-104 |

| Cumulative Volume (mL) over 56 day- | 98- | 102- | 200- | 234- | 132- | 98- | 98- | 132- |
|---|---|---|---|---|---|---|---|---|
| period <sup>g,i</sup> | 104 | 108 | 212 | 246 | 138 | 104 | 104 | 138 |
| | 98- | 102- | 200- | 234- | 332- | 430- | 528- | 562- |
| Total Cumulative Volume (mL) <sup>g,i</sup> | 104 | 108 | 212 | 246 | 350 | 454 | 558 | 592 |

<sup>&</sup>lt;sup>a</sup> Optional screening visit – informed consent and screening activities can be a separate visit or combined with Day 1.

<sup>f</sup>Collect nasal swab for PCR (1-2). Swabs can be self-collected and visit done by phone. Sequencing will be performed on all Illness visit-confirmed SARS-CoV-2 specimens.

mIf a participant is planning to receive a COVID-19 booster outside the study, an unscheduled visit will be performed where safety and immunogenicity (collection of sera, plasma and PBMC) assessments will be performed. However, if that planned visit falls within twice the window for an upcoming visit (e.g +/- 14 days for D 91, +/-28 days for D 181 and D 271, +/- 56 days for D 366) then it will occur and be documented as out of window for the planned upcoming scheduled visit (refer to MOP for more guidance).

<sup>&</sup>lt;sup>b</sup> Telephone visit

<sup>&</sup>lt;sup>c</sup> Vital signs and targeted physical exam will be performed on screening and before vaccination otherwise, only as clinically indicated or based on interim medical history.

<sup>&</sup>lt;sup>d</sup> For subjects of childbearing potential, a urine pregnancy will be performed at screening. If enrollment occurs on a separate day, a repeat urine pregnancy test will be done within 24 hours of study vaccine administration and negative results confirmed prior to dosing.

<sup>&</sup>lt;sup>e</sup> The memory aid will be distributed at the Day 1 visit, queried for completion at the Day 8 telephone call and reviewed during an interview with the subject at the D15 visit and confirmed data recorded on the DCF.

g Inability (e.g., failure of venipuncture) to collect all baseline samples on Day 1 will not exclude the subject from further participation in this study as long as a minimum of baseline blood volume is collected (refer to the MOP for the protocol defined minimum number of required aliquots). Blood volume for PBMC varies depending on the type of tubes used for blood collection (refer to the MOP).

<sup>&</sup>lt;sup>h</sup> Selected sites will perform PBMC separation on selected subjects (refer to MOP for more guidance).

<sup>&</sup>lt;sup>i</sup>Blood volumes for early termination visit are not included in the blood volume totals.

<sup>&</sup>lt;sup>j</sup> After vaccination on Day 1, immunosuppressant drugs, COVID-19 related prophylaxis and therapies as well as vaccines will be recorded. For any SAE occurring at any time during the study, all medications will be recorded.

<sup>&</sup>lt;sup>k</sup> If an unscheduled visit is performed to evaluate an adverse event, vital signs and targeted physical exam will be performed, as indicated. If, in the judgement of the site investigator, the event, occurring within 4 weeks after vaccination, is a case of suspected myocarditis and/or pericarditis, the site will coordinate an appropriate diagnostic workup to make a determination of probable or confirmed myocarditis and/or pericarditis which may include, but is not limited to, an ECG, cardiac troponin testing and referral to a cardiologist (directly, or through the emergency department or primary care clinic). The suspected myocarditis and/or pericarditis case should be reported to the DMID Medical Monitor within 24 hours of site awareness. <sup>l</sup>Serum for biomarker testing will be collected on Day 4 and stored for potential biomarker testing at a central laboratory and compared to testing of an aliquot from serum obtained on Day 1. If an unscheduled visit is related to a concern for myocarditis and/or pericarditis within 4 weeks after vaccination, a 4 mL SST will be collected and stored for potential biomarker testing at a central laboratory.

**Table 4:** Schedule of Study Procedures - 2 Doses

| Study Day | D-<br>28<br>to | 1 | 4 | 8 <sup>b</sup> | 15 | 29 | 57 | 60 | 64 <sup>b</sup> | 71 | 85 | 147 | 237 | 327 | 422 | Illness/<br>Unscheduled<br>Visit <sup>k,m</sup> | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <b>D-</b> 1 | | | | | | | | | | | | | | | | |
| Visit Number | 00a | 1 | 1A | 2 | 3 | 4 | 5 | 5A | 6 | 7 | 8 | 9 | 10 | 11 | 12 | | |
| Window (+/-) | | 0 | 1 | 1 | 2 | 2 | 3 | 1 | 1 | 2 | 2 | 7 <sup>m</sup> | 14 <sup>m</sup> | 14 <sup>m</sup> | 28 <sup>m</sup> | | |
| Informed Consent <sup>a</sup> | X | | | | | | | | | | | | | | | | |
| Eligibility Criteria | X | | | | | | X | | | | | | | | | | |
| Medical History | X | | | | | | X | | | | | | | | | | |
| Vaccination | | X | | | | | X | | | | | | | | | | |
| Concomitant Meds | X | X | X <sup>j</sup> | X <sup>j</sup> | $X^{j}$ | $X^{j}$ | $X^{j}$ | X <sup>j</sup> | X <sup>j</sup> | $X^{j}$ | X <sup>j</sup> | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ | $X^{j}$ |
| Interim History | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical Exam <sup>c</sup> –<br>Targeted | X | X | | | | | X | | | | | | | | | (X) | |
| Vital Signs <sup>c</sup> | X | X | | | | | X | | | | | | | | | (X) | |
| Height/Weight (BMI) <sup>a</sup> | X | | | | | | | | | | | | | | | | |
| Urine β-HCG <sup>d</sup> | X | X | | | | | X | | | | | | | | | | |
| Memory Aid <sup>e</sup> | | X | X | X | | | X | X | X | | | | | | | | |
| Solicited AEs | | X | X | X | | | X | X | X | | | | | | | | |
| Unsolicited AEs | | X | X | X | X | X | X | X | X | X | X | | | | | | |
| MAAEs, SAEs,<br>NOCMCs, AEs leading<br>to withdrawal from the<br>study and AESIs | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Nasal swab for PCR & Sequencing <sup>f</sup> | | | | | | | | | | | | | | | | (X) | |
| Assays | | | | | | | | | | | | | | | | | |
| Serum for Serological<br>Immunogenicity | | 34 <sup>1</sup> | 4 <sup>1</sup> | | 34 | 34 | 34 <sup>1</sup> | 4 <sup>1</sup> | | 34 | 34 | 34 | 34 | 34 | 34 | 4 <sup>1</sup> -34 <sup>m</sup> | 34 |

| Study Day | D-<br>28<br>to<br>D-<br>1 | 1 | 4 | 8 <sup>b</sup> | 15 | 29 | 57 | 60 | 64 <sup>b</sup> | 71 | 85 | 147 | 237 | 327 | 422 | Illness/<br>Unscheduled<br>Visit <sup>k,m</sup> | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Number | 00a | 1 | 1A | 2 | 3 | 4 | 5 | 5A | 6 | 7 | 8 | 9 | 10 | 11 | 12 | | |
| Window (+/-) | | 0 | 1 | 1 | 2 | 2 | 3 | 1 | 1 | 2 | 2 | 7 <sup>m</sup> | 14 <sup>m</sup> | 14 <sup>m</sup> | 28 <sup>m</sup> | | |
| Assays <sup>g</sup> and Biomarker<br>Testing <sup>l</sup> | | | | | | | | | | | | | | | | | |
| PBMC Cellular Assays<br>& Plasma <sup>g,h</sup><br>(select sites only) | | 64-<br>70 | | | 64-<br>70 | | 64-<br>70 | | | 64-<br>70 | | 64-<br>70 | 64-<br>70 | 64-<br>70 | | 64-70 <sup>m</sup> | 64-70 |
| Daily Volume (mL) <sup>g,i</sup> | | 98-<br>104 | 4 | | 98-<br>104 | 34 | 98-<br>104 | 4 | | 98-<br>104 | 34 | 98-<br>104 | 98-<br>104 | 98-<br>104 | 34 | 4-104 | 98-104 |
| Cumulative Volume (mL) over 56 day-period <sup>g,i</sup> | | 98-<br>104 | 102-<br>108 | | 200-<br>212 | 234-<br>246 | 332-<br>350 | 238-<br>250 | | 336-<br>354 | 268-<br>280 | 132-<br>138 | 98-<br>104 | 98-<br>104 | 132-<br>138 | | |
| Total Cumulative<br>Volume (mL) <sup>g,i</sup> | | 98-<br>104 | 102-<br>108 | | 200-<br>212 | 234-<br>246 | 332-<br>350 | 336-<br>354 | | 434-<br>458 | 468-<br>492 | 566-<br>596 | 664-<br>700 | 762-<br>804 | 796-<br>838 | | |

<sup>&</sup>lt;sup>a</sup> Optional screening visit – informed consent and screening activities can be a separate visit or combined with Day 1.

<sup>&</sup>lt;sup>b</sup> Telephone visit

<sup>&</sup>lt;sup>c</sup> Vital signs and targeted physical exam will be performed on screening and before vaccination otherwise, only as clinically indicated or based on interim medical history.

<sup>&</sup>lt;sup>d</sup> For subjects of childbearing potential, a urine pregnancy test will be performed at screening. If enrollment occurs on a separate day as screening, a repeat urine pregnancy test will be done within 24 hours of first study vaccine administration and repeated on day 57 prior to second study vaccine administration. Negative results must be confirmed prior to each dosing. <sup>e</sup> The memory aid will be distributed at the Day 1 and Day 57 visits, queried for completion at the Day 8 and Day 64 telephone calls and reviewed during an interview with the subject at the D15 and Day 71 visits and confirmed data recorded on the DCF.

<sup>&</sup>lt;sup>f</sup>Collect nasal swab for PCR (1-2). Swabs can be self-collected and visit done by phone. Sequencing will be performed on all Illness visit-confirmed SARS-CoV-2 specimens.

g Inability (e.g., failure of venipuncture) to collect all baseline samples on Day 1 will not exclude the subject from further participation in this study as long as a minimum of baseline blood volume is collected (refer to the MOP for the protocol defined minimum number of required aliquots). Blood volume for PBMC varies depending on the type of tubes used for the blood collection (refer to the MOP).

<sup>&</sup>lt;sup>h</sup> Selected sites will perform PBMC separation on selected subjects (refer to MOP for more guidance).

<sup>&</sup>lt;sup>i</sup>Blood volumes for early termination visit are not included in the blood volume totals.

<sup>&</sup>lt;sup>j</sup> After vaccination on Day 1, immunosuppressant drugs, COVID-19 related prophylaxis and therapies as well as vaccines will be recorded. For any SAE occurring at any time during the study, all medications will be recorded.

<sup>k</sup> If an unscheduled visit is performed to evaluate an adverse event, vital signs and targeted physical exam will be performed, as indicated. If, in the judgement of the site investigator, the event, occurring within 4 weeks after each vaccination, is a case of suspected myocarditis and/or pericarditis, the site will coordinate an appropriate diagnostic workup to make a determination of probable or confirmed myocarditis and/or pericarditis which may include, but is not limited to, an ECG, cardiac troponin testing and referral to a cardiologist (directly, or through the emergency department or primary care clinic). The suspected myocarditis and/or pericarditis case should be reported to the DMID Medical Monitor within 24 hours of site awareness.

Serum for biomarker testing will be collected on Days 4 and 60 and stored for potential biomarker testing at a central laboratory and compared to testing of an aliquot of serum obtained on Days 1 and 57, respectively. If an unscheduled visit is related to a concern for myocarditis and/or pericarditis within 4 weeks after vaccination, a 4 mL SST will be collected and stored for potential biomarker testing at a central laboratory.

mIf a participant is planning to receive a COVID-19 booster outside the study, an unscheduled visit will be performed where safety and immunogenicity (collection of sera, plasma and PBMC) assessments will be performed. However, if that planned visit falls within twice the window for an upcoming visit (e.g +/- 14 days for D 147, +/-28 days for D 237 and D 327, +/- 56 days for D 422) then it will occur and be documented as out of window for the planned upcoming scheduled visit (refer to MOP for more guidance).

Note Windows for subsequent visits should be based off the preceding vaccination visit.

If intercurrent SARS- CoV-2 infection occurs between the first and prior to the planned second study dose or if a COVID-19 vaccine is given outside the study between the first and prior to the planned second study dose, no second vaccination will be given. Participants who do not receive a second dose will revert to the schedule of activities for single dose participants.

## 9.7.1 Sample Size

Table 5: Probability of observing one or more Adverse Events for various event rates in one vaccine group (or strata)

| <u>N</u> | "True" Event<br>Rate | Probability of Observing ≥ 1<br>events (%) | <u>N</u> | "True" Event Rate | Probability of Observing ≥ 1<br>events (%) |
|---|---|---|---|---|---|
| 100 | 0.1% | 9.5 | <u>50</u> | 0.1% | 4.9 |
| | 0.5% | 39.4 | | 0.5% | 22.2 |
| | 1.0% | 63.4 | | 1.0% | 39.5 |
| | 2.0% | 86.7 | | 2.0% | 63.6 |
| | 3.0% | 95.2 | | 3.0% | 78.2 |
| | 4.0% | 98.3 | | 4.0% | 87 |
| | <u>5.0%</u> | 99.4 | | 5.0% | 92.3 |
| | 10.0% | <u>&gt;99.9</u> | | 10.0% | 99.5 |
| | <u>15.0%</u> | <u>&gt;99.9</u> | | <u>15.0%</u> | <u>&gt;99.9</u> |
| | 20.0% | <u>&gt;99.9</u> | | 20.0% | <u>&gt;99.9</u> |
| | 30.0% | <u>&gt;99.9</u> | | 30.0% | <u>&gt;99.9</u> |
| <u>25</u> | 0.1% | <u>2.5</u> | <u>15</u> | 0.1% | 1.5 |
| | 0.5% | <u>11.8</u> | | 0.5% | 7.2 |
| | <u>1.0%</u> | <u>22.2</u> | | 1.0% | 14 |
| | 2.0% | <u>39.7</u> | | 2.0% | 26.1 |
| | 3.0% | <u>53.3</u> | | 3.0% | 36.7 |
| | 4.0% | <u>64.0</u> | | 4.0% | 45.8 |
| | <u>5.0%</u> | <u>72.3</u> | | 5.0% | 53.7 |
| | 10.0% | <u>92.8</u> | | 10.0% | 79.4 |
| | <u>15.0%</u> | <u>98.3</u> | | <u>15.0%</u> | 91.3 |
| | 20.0% | <u>99.6</u> | | 20.0% | 96.5 |
| | 30.0% | <u>&gt;99.9</u> | | 30.0% | 99.5 |

Table 6: Two-sided 95% confidence intervals based on observing a particular average loge-antibody titer in subjects' vaccine groups and potential strata sizes

| Observed<br>average loge<br>antibody titer | SD of loge<br>antibody<br>titer | | 95% confidenc<br>GMT in vaccine gr | | |
|---|---|---|---|---|---|
| antibody titer | titer | N = 100 | N = 50 | N = 25 | N = 15 |
| log <sub>e</sub> (5) | 0.5 | (4.5, 5.5) | (4.3, 5.8) | (4.1, 6.1) | (3.8, 6.6) |
| log <sub>e</sub> (20) | | (18.1, 22.1) | (17.4, 23.1) | (16.3, 24.6) | (15.2, 26.4) |
| log <sub>e</sub> (50) | | (45.3, 55.2) | (43.4, 57.6) | (40.7, 61.5) | (37.9, 66) |
| log <sub>e</sub> (100) | | (90.6, 110.4) | (86.8, 115.3) | (81.4, 122.9) | (75.8, 131.9) |

| Observed<br>average loge | SD of loge<br>antibody<br>titer | | 95% confidenc<br>GMT in vaccine gr | | |
|---|---|---|---|---|---|
| antibody titer | utter | N = 100 | N = 50 | N = 25 | N = 15 |
| log <sub>e</sub> (250) | | (226.4, 276.1) | (216.9, 288.2) | (203.4, 307.3) | (189.5, 329.8) |
| log <sub>e</sub> (500) | | (452.8, 552.1) | (433.8, 576.3) | (406.8, 614.6) | (379.1, 659.5) |
| log <sub>e</sub> (1000) | | (905.6, 1104.3) | (867.5, 1152.7) | (813.5, 1229.2) | (758.1, 1319) |
| log <sub>e</sub> (5) | 1.0 | (4.1, 6.1) | (3.8, 6.6) | (3.3, 7.6) | (2.9, 8.7) |
| log <sub>e</sub> (20) | | (16.4, 24.4) | (15.1, 26.6) | (13.2, 30.2) | (11.5, 34.8) |
| log <sub>e</sub> (50) | | (41, 61) | (37.6, 66.4) | (33.1, 75.6) | (28.7, 87) |
| log <sub>e</sub> (100) | | (82, 121.9) | (75.3, 132.9) | (66.2, 151.1) | (57.5, 174) |
| log <sub>e</sub> (250) | | (205, 304.9) | (188.2, 332.2) | (165.5, 377.8) | (143.7, 435) |
| log <sub>e</sub> (500) | | (410, 609.7) | (376.3, 664.3) | (330.9, 755.5) | (287.4, 869.9) |
| log <sub>e</sub> (1000) | | (820, 1219.5) | (752.6, 1328.7) | (661.8, 1511) | (574.8, 1739.8) |

## **10.2** Protocol Deviations

## Table 7: Distribution of Protocol Deviations by Category, Type, and Treatment Group

[Implementation Note: Only display deviations that have occurred in at least one treatment group.]

| | | | otype<br>=X) | (B.1.3<br>Omi<br>(B.1.3 | eta<br>351) +<br>icron<br>1.529)<br>=X) | (B.1.3<br>Omi<br>(B.1.1<br>[two o | eta<br>351) +<br>(cron<br>1.529)<br>doses]<br>=X) | (B.1.0<br>+ Om<br>(B.1.1 | elta<br>617.2)<br>nicron<br>1.529)<br>=X) | (B.1. | eron<br>1.529)<br>=X) | (B.1.1<br>Prote | cron<br>1.529)<br>+<br>otype<br>=X) | Sub | .ll<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. |
| Eligibility/enrollment | Any type | Subj | Berr | Subj | Dev. | Subj | Dev. | Subj | Dev. | Subj | Dev. | Subj | Dev. | Subj | Dev. |
| | Did not meet inclusion criterion | x | x | x | x | x | x | x | x | x | x | x | x | x | x |
| | Met exclusion criterion | | | | | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | | | |
| | Missed treatment administration | | | | | | | | | | | | | | |
| | Delayed treatment administration | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | | | | | | | |
| | Blood not collected | | | | | | | | | | | | | | |
| | COVID-19 test swab not collected | | | | | | | | | | | | | | |
| | Other specimen not collected | | | | | | | | | | | | | | |

| | | | otype<br>=X) | (B.1.3<br>Omi<br>(B.1.1 | eta<br>351) +<br>cron<br>1.529)<br>=X) | (B.1.3<br>Omi<br>(B.1.1<br>[two | eta<br>351) +<br>(cron<br>1.529)<br>doses]<br>=X) | (B.1.0<br>+ Om<br>(B.1.1 | elta<br>617.2)<br>nicron<br>1.529)<br>=X) | Omicron (B.1.1.529) (N=X) No. No. | | B.1.1.529) Prototypo<br>(N=X) (N=X) | | Sub | .ll<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. | No.<br>of<br>Subj | No.<br>of<br>Dev. |
| | Too few aliquots obtained | | | | | | | | | | | | | | |
| | Specimen result not obtained | | | | | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | | | | | |
| | Specimen temperature excursion | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Treatment administration | Any type | | | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | |
| Note: N=Number o | f subjects in the Safety | Popula | ation. | | | 1 | 1 | | | | | | | • | |

Table with similar format:

Table 8: Distribution of Major Protocol Deviations by Category, Type, and Treatment Group

## 12.2.2 Displays of Adverse Events

The toxicity grading scales in the FDA "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" will be used.

# 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

Not applicable.

## 14.1 Description of Study Subjects

## 14.1.1 Disposition of Subjects

**Table 9:** Subject Disposition by Treatment Group

| Subject<br>Disposition | | otype<br>=X) | (B.1.3<br>Omi<br>(B.1.3 | eta<br>351) +<br>icron<br>1.529)<br>=X) | (B.1.3<br>Omi<br>(B.1.3<br>(2 D | eta<br>351) +<br>(cron<br>1.529)<br>oses)<br>=X) | (B.1.6<br>Omi<br>(B.1.2 | elta<br>17.2) +<br>icron<br>1.529)<br>=X) | (B.1.) | cron<br>1.529)<br>=X) | (B.1.1<br>Prot | Omicron<br>(B.1.1.529) +<br>Prototype<br>(N=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | | | | | | | | | | | | | X | |
| Enrolled/Randomized | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 | X | 100 |
| Received First<br>Vaccination | Х | XX | Х | xx | х | xx | х | XX | Х | XX | х | XX | Х | XX |
| Received Second<br>Vaccination | NA | NA | х | xx | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA |
| Completed Final<br>Blood Draw | | | | | | | | | | | | | | |
| Completed Follow-up <sup>a</sup> | | | | | | | | | | | | | | |
| Completed Per<br>Protocol <sup>b</sup> | | | | | | | | | | | | | | |

Note: N=Number of subjects enrolled in the study.

<sup>&</sup>lt;sup>a</sup> Refer to Listing 2 for reasons subjects discontinued or terminated early.

<sup>&</sup>lt;sup>b</sup> Refer to Listing 5 for reasons subjects are excluded from the Analysis populations.

**Table 10:** Analysis Populations by Treatment Group

| Analysis<br>Populations | Reason Subjects<br>Excluded | | otype<br>=X) | (B.1<br>Om<br>(B.1. | eta<br>.351)<br>+<br>icron<br>1.529)<br>=X) | (B.1<br>Omi<br>(B.1.<br>(2 D | eta<br>.351)<br>+<br>icron<br>1.529)<br>oses)<br>=X) | (B.1.<br>Om<br>(B.1. | elta<br>617.2)<br>+<br>icron<br>1.529)<br>=X) | Omicron<br>(B.1.1.529)<br>(N=X) | | (B.1. | icron<br>1.529)<br>+<br>otype<br>=X) | Sub | All<br>jects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | % | n |
| mITT Population | Any Reason | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | [Reason 1, for<br>example: Did not meet<br>eligibility criteria] | | | | | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | | | | | |
| | [Reason 4] | | | | | | | | | | | | | | |
| Per Protocol<br>Population | Any Reason | | | | | | | | | | | | | | |
| | [Reason 1] | | | | | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | | | | | |
| Safety<br>Population | Any Reason | | | | | | | | | | | | | | |
| | [Reason 1] | | | | | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | | | | | |

**Table 11:** Ineligibility Summary of Screen Failures

[Implementation Note: See section 4.3 for inclusion and exclusion criteria.]

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | X | 100 |
| Inclusion | Any inclusion criterion | X | XX |
| | [inclusion criterion 1] | X | XX |
| | [inclusion criterion 2] | X | XX |
| | [inclusion criterion 3] | X | XX |
| Exclusion | Any exclusion criterion | X | XX |
| | [exclusion criterion 1] | X | XX |
| | [exclusion criterion 2] | X | xx |
| | [exclusion criterion 3] | X | XX |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.

<sup>&</sup>lt;sup>b</sup> Denominator for percentages is the total number of screen failures.

## 14.1.2 Demographic Data by Study Group

Table 12: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects

| Variable | Characteristic | | otype<br>=X) | Om<br>(B.1. | 1.351) +<br>icron<br>1.529)<br>=X) | Omi<br>(B.1.<br>(2 D | .1.351) +<br>icron<br>1.529)<br>oses)<br>=X) | + On<br>(B.1. | 3.1.617.2)<br>nicron<br>1.529)<br>=X) | (B.1. | Omicron<br>(B.1.1.529)<br>(N=X) | | icron<br>.529) +<br>otype<br>=X) | | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | Х | XX | X | XX | X | XX | Х | XX | X | XX | X | XX | Х | XX |
| | Female | | | | | | | | | | | | | | |
| Ethnicity | Not Hispanic or LatinX | Х | XX | x | xx | X | xx | Х | xx | X | XX | x | XX | Х | XX |
| | Hispanic or LatinX | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Race | American Indian or Alaska<br>Native | Х | XX | Х | xx | X | xx | х | xx | X | xx | Х | xx | х | xx |
| | Asian | | | | | | | | | | | | | | |
| | Native Hawaiian or Other<br>Pacific Islander | | | | | | | | | | | | | | |
| | Black or African American | | | | | | | | | | | | | | |
| | White | | | | | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | |
| Age Group | 18-64 years | | | | | | | | | | | | | | |
| | >= 65 years | | | | | | | | | | | | | | |
| Prior Infection | Yes | | | | | | | | | | | | | | |
| (Self Report) | No | | | | | | | | | | | | | | |

| Variable | Characteristic | | otype<br>=X) | Om<br>(B.1. | .1.351) +<br>icron<br>1.529)<br>=X) | Omi<br>(B.1.1 | 1.351) +<br>cron<br>1.529)<br>oses)<br>=X) | + On<br>(B.1. | 3.1.617.2)<br>nicron<br>1.529)<br>=X) | (B.1.) | cron<br>1.529)<br>=X) | (B.1.1 | cron<br>.529) +<br>otype<br>=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Prior Infection | Yes | | | | | | | | | | | | | | |
| (Positive<br>Nuclear<br>Protein Antibody<br>or Self-Report) | No | | | | | | | | | | | | | | |
| SARS-COV-2<br>Vaccination | mRNA Primary, mRNA<br>Boost | | | | | | | | | | | | | | |
| Regimen | Ad26 Primary, mRNA<br>Boost | | | | | | | | | | | | | | |
| | Ad26 Primary, Ad26 Boost | | | | | | | | | | | | | | |

Note: N=Number of subjects in the Safety Population.

Table 13: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group, All Enrolled Subjects

| Variable | Statistic | Prototype<br>(N=X) | Beta (B.1.351)<br>+ Omicron<br>(B.1.1.529)<br>(N=X) | Beta<br>(B.1.351) +<br>Omicron<br>(B.1.1.529)<br>(2 Doses)<br>(N=X) | Delta<br>(B.1.617.2)<br>+ Omicron<br>(B.1.1.529)<br>(N=X) | Omicron<br>(B.1.1.529)<br>(N=X) | Omicron<br>(B.1.1.529)<br>+<br>Prototype<br>(N=X) | All<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Age (Years) | Mean | XX | xx | xx | xx | xx | XX | xx |
| | Standard<br>Deviation | XX | XX | XX | XX | XX | XX | xx |
| | Median | Х | x | X | X | X | X | Х |
| | Minimum | Х | x | X | X | X | X | Х |
| | Maximum | Х | х | x | х | x | X | Х |
| Height (cm) | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Weight (kg) | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| BMI (kg/m²) | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Days since | Mean | | | | | | | |
| most recent<br>COVID19<br>Vaccine | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Days since | n | | | | | | | |
| most recent self-reported | Mean | | | | | | | |
| COVID19<br>infection | Standard<br>Deviation | | | | | | | |

| Variable | Statistic | Prototype<br>(N=X) | Beta (B.1.351)<br>+ Omicron<br>(B.1.1.529)<br>(N=X) | Beta<br>(B.1.351) +<br>Omicron<br>(B.1.1.529)<br>(2 Doses)<br>(N=X) | Delta<br>(B.1.617.2)<br>+ Omicron<br>(B.1.1.529)<br>(N=X) | Omicron<br>(B.1.1.529)<br>(N=X) | Omicron<br>(B.1.1.529)<br>+<br>Prototype<br>(N=X) | All<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Days since | Mean | | | | | | | |
| most recent<br>self-reported<br>COVID19 | Standard<br>Deviation | | | | | | | |
| infection or<br>COVID19<br>Vaccination | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |

Note: N=Number of subjects in the Safety Population

### 14.1.3 Prior and Concurrent Medical Conditions

Table 14: Summary of Subjects with Pre-Existing Medical Conditions by MedDRA System Organ Class and Treatment Group

| MedDRA System Organ Class | | otype<br>-X) | Om<br>(B.1. | .1.351) +<br>icron<br>1.529)<br>=X) | Omi<br>(B.1.<br>(2 D | 1.351) +<br>icron<br>1.529)<br>oses)<br>=X) | Delta (B.1.617.2)<br>+ Omicron<br>(B.1.1.529)<br>(N=X) | | Omicron<br>(B.1.1.529)<br>(N=X) | | Omicron<br>(B.1.1.529) +<br>Prototype<br>(N=X) | | All Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | х | XX | Х | XX | X | XX | X | xx | X | XX | X | xx | X | XX |
| [SOC 1] | | | | | | | | | | | | | | |
| [SOC 2] | | | | | | | | | | | | | | |

Note: N=Number of subjects in the Safety Population; n = Number of subjects reporting medical history within the specified SOC.

A subject is only counted once per SOC.

## 14.2 Immunogenicity Data

Table 15: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Overall – mITT Population

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.5/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 1 | n | х | Х | X | X | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 15 | n | X | X | X | X | X | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 29 | n | X | X | X | X | Х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 91 | n | х | Х | X | X | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.5/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMR <sub>D614G</sub><br>(95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 181 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 271 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 366 | n | X | X | X | X | Х | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.5/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |

Note: N=Number of subjects in the mITT Population.

n=Number of subjects with results available at time point.

GM=Geometric Mean, GMR<sub>D614G</sub>=Geometric Mean Ratio to D614G variant, GMFR=Geometric Mean Fold Rise, GMFD=Geometric Mean Fold Drop.

Confidence intervals of the GM, GMR, GMFR, and GMFD were calculated with the Student's t distribution on log-transformed data. Confidence intervals of the Seropositive rate were calculated with the Clopper-Pearson method.

### Implementation notes:

Extra variant columns may be added for additional variants.

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

Add a note to indicate the lower limit of detection for the assay used to calculate the seropositive rate.

#### Tables with Similar Format:

- Table 16: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Overall Per Protocol Population
- Table 17: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Table 18: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- Table 19: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Older Cohort mITT Population
- Table 20: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Older Cohort Per Protocol Population
- Table 21: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 22: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein)

  Cohort Per Protocol Population

- Table 23: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 24: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 25: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 26: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 27: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 28: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 29: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 30: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 31: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 32: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 33: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall mITT Population
- Table 34: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall Per Protocol Population
- Table 35: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort mITT Population
- Table 36: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort Per Protocol Population

- Table 37: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort mITT Population
- Table 38: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Table 39: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 40: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 41: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 42: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 43: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 44: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 45: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 46: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 47: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 48: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 49: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Table 50: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 51: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Overall mITT Population
- Table 52: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Table 53: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort mITT Population
- Table 54: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort Per Protocol Population
- Table 55: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Table 56: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol Population
- Table 57: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 58: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 59: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 60: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 61: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 62: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 63: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Table 64: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 65: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 66: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 67: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 68: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 69: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Overall—mITT Population
- Table 70: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Overall Per Protocol Population
- Table 71: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Younger Cohort mITT Population
- Table 72: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- Table 73: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Cohort mITT Population
- Table 74: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Cohort Per Protocol Population
- Table 75: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein)

  Cohort mITT Population
- Table 76: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein)

  Cohort Per Protocol Population
- Table 77: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 78: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

- Table 79: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 80: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 81: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 82: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 83: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 84: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 85: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 86: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 87: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Overall– mITT Population
- Table 88: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Overall– Per Protocol Population
- Table 89: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT Population
- Table 90: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort Per Protocol Population
- Table 91: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort mITT Population
- Table 92: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- Table 93: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 94: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 95: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 96: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 97: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 98: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 99: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 100: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 101: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 102: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 103: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 104: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 105: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 1 | n | X | X | x | x | X | X |
| | GMT (95% | X.X | X.X | X.X | X.X | X.X | X.X |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | X.X | X.X | X.X | X.X | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 15 | n | X | X | X | X | X | X |
| | GMT (95% | X.X | X.X | X.X | X.X | x.x | X.X |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFR<br>(95% CI) | X.X | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (9376 CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 29 | n | X | X | X | X | X | X |
| | GMT (95% | X.X | X.X | X.X | X.X | X.X | X.X |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFR<br>(95% CI) | x.x | x.x | x.x | X.X | X.X | X.X |
| | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (9370 C1) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 57 | n | X | X | X | X | X | X |
| | GMT (95%<br>CI) | x.x | X.X | x.x | x.x | x.x | X.X |
| | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median (Min,Max) | x.x | X.X | x.x | X.X | X.X | X.X |
| | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x | X.X | x.x | x.x | X.X |
| | (9370 CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 71 | n | Х | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 85 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 147 | n | х | X | X | X | х | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub><br>(95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMFD | X.X | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 237 | n | X | X | X | X | X | X |
| | GMT (95% | X.X | X.X | X.X | X.X | X.X | X.X |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x | x.x | X.X | X.X | X.X |
| | | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFR<br>(95% CI) | X.X | X.X | X.X | X.X | X.X | x.x |
| | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD<br>(95% CI) | X.X | X.X | (x.x, x.x) | X.X | X.X | X.X<br>(v.v.v.v.) |
| | | (x.x, x.x)<br>0.0X | (x.x, x.x)<br>0.0X | 0.0X | (x.x, x.x)<br>0.0X | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | (0.x,0.x) | (0.x,0.x) | (0.x) | (0.x,0.x) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 327 | n | X | X | X | X | X | X |
| Day 327 | GMT (95% | | | | | | |
| | CI) | (x.x, x.x) | x.x<br>(x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median | X.X | X.X | X.X | X.X | X.X | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFR | X.X | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | X.X | X.X | x.x | X.X | X.X | X.X |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 422 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | X.X | x.x | x.x | x.x | X.X |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median (Min May) | X.X | X.X | X.X | X.X | X.X | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x | x.x | X.X | x.x | x.x |
| | ` ' | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFR<br>(95% CI) | x.x | x.x | X.X | X.X | x.x | X.X |
| | ` ' | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD<br>(95% CI) | X.X | X.X | X.X | X.X | X.X | X.X |
| | (20,001) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |

n=Number of subjects with results available at time point.

GM=Geometric Mean, GMR<sub>D614G</sub>=Geometric Mean Ratio to D614G variant, GMFR=Geometric Mean Fold Rise, GMFD=Geometric Mean Fold Drop.

Confidence intervals of the GM, GMR, GMFR, and GMFD were calculated with the Student's t distribution on log-transformed data. Confidence intervals of the Seropositive rate were calculated with the Clopper-Pearson method.

# Implementation notes:

Extra variant columns may be added for additional variants.

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

Add a note to indicate the lower limit of detection for the assay used to calculate the seropositive rate.

- Table 106: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall– Per Protocol Population
- Table 107: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort mITT Population
- Table 108: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Table 109: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort mITT Population
- Table 110: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Table 111: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 112: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population

- Table 113: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 114: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 115: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 116: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 117: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 118: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 119: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 120: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 121: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 122: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 123: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall – mITT Population

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 1 | n | x | х | x | x | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub><br>(95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 15 | n | X | X | х | х | Х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 29 | n | x | X | x | х | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 91 | n | х | X | х | X | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 181 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 271 | n | X | X | X | х | Х | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 366 | n | х | X | X | х | х | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFD<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |

n=Number of subjects with results available at time point.

GM=Geometric Mean, GMR<sub>D614G</sub>=Geometric Mean Ratio to D614G variant, GMFR=Geometric Mean Fold Rise,

GMFD=Geometric Mean Fold Drop.

Confidence intervals of the GM, GMR, GMFR, and GMFD were calculated with the Student's t distribution on log-transformed data. Confidence intervals of the Seropositive rate were calculated with the Clopper-Pearson method.

# Implementation notes:

Extra variant columns included as placeholders may not be needed.

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

Add a note to indicate the lower limit of detection for the assay used to calculate the seropositive rate.

- Table 124: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall Per Protocol Population
- Table 125: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Table 126: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- Table 127: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort mITT Population
- **Table 128:** Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort Per Protocol Population
- Table 129: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 130: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population

- Table 131: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 132: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 133: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 134: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 135: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 136: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 137: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 138: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 139: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 140: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 141: Pseudovirus Neutralization Assay ID50 Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Overall—mITT Population
- Table 142: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population
- Table 143: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Cohort mITT Population
- Table 144: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Table 145: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort mITT Population
- Table 146: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population
- Table 147: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population

- Table 148: Pseudovirus Neutralization Assay ID50 Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Table 149: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Table 150: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Table 151: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT
  Population
- Table 152: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Table 153: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Table 154: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Table 155: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT
  Population
- Table 156: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Table 157: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Table 158: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 1
  Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Table 159: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall– mITT Population
- Table 160: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Table 161: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort mITT Population
- Table 162: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort Per Protocol Population

- Table 163: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Table 164: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol Population
- Table 165: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 166: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 167: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 168: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 169: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 170: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant,
  Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Table 171: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 172: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 173: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 174: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 175: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 176: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant,
  Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Table 177: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Overall– mITT Population

- Table 178: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Overall Per Protocol Population
- Table 179: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort mITT Population
- **Table 180:** Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- Table 181: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort mITT Population
- Table 182: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort Per Protocol Population
- Table 183: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 184: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 185: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 186: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 187: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 188: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 189: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 190: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 191: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 192: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 193: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 194: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 195: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall mITT Population

- Table 196: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall Per Protocol Population
- Table 197: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT Population
- Table 198: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort Per Protocol Population
- Table 199: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort mITT Population
- Table 200: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- Table 201: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population
- Table 202: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 203: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 204: Pseudovirus Neutralization Assay ID50 Summary Results by Time Point and Variant,
  Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Table 205: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 206: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 207: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Table 208: Pseudovirus Neutralization Assay ID50 Summary Results by Time Point and Variant,
  Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Table 209: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 210: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population

- Table 211: Pseudovirus Neutralization Assay ID50 Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 212: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 213: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 1 | n | X | X | X | X | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 15 | n | X | X | X | X | Х | Х |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 29 | n | X | X | X | X | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub><br>(95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 57 | n | х | Х | X | X | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 71 | n | X | Х | X | х | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 85 | n | X | X | X | х | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 147 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 237 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 327 | n | X | Х | X | х | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 422 | n | x | X | X | X | x | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMR <sub>D614G</sub><br>(95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFD<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |

n=Number of subjects with results available at time point.

GM=Geometric Mean, GMR<sub>D614G</sub>=Geometric Mean Ratio to D614G variant, GMFR=Geometric Mean Fold Rise,

GMFD=Geometric Mean Fold Drop.

Confidence intervals of the GM, GMR, GMFR, and GMFD were calculated with the Student's t distribution on log-transformed data. Confidence intervals of the Seropositive rate were calculated with the Clopper-Pearson method.

## Implementation notes:

Extra variant columns may be added for additional variants.

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

Add a note to indicate the lower limit of detection for the assay used to calculate the seropositive rate.

- Table 214: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population
- Table 215: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort mITT Population
- Table 216: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population
- Table 217: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population
- Table 218: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population
- Table 219: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2
  Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 220: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2
  Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol
  Population

- Table 221: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Table 222: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Table 223: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT
  Population
- Table 224: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Table 225: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Table 226: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Table 227: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population
- Table 228: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Table 229: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Table 230: Pseudovirus Neutralization Assay ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population

Table 231: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall – mITT Population

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1<br>(N=X) | BA.2.12.1(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 1 | n | x | X | X | x | Х | Х |
| | GMT (95% | X.X | X.X | X.X | X.X | X.X | X.X |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | X.X | X.X | X.X | X.X | x.x | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | X.X | x.x | x.x | x.x |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 15 | n | X | X | X | X | Х | X |
| | GMT (95% | X.X | X.X | X.X | X.X | x.x | X.X |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | X.X | X.X | X.X | X.X | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | X.X | x.x | x.x | X.X |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFR | X.X | X.X | X.X | X.X | x.x | X.X |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 29 | n | X | X | X | X | X | X |
| | GMT (95% | X.X | X.X | X.X | X.X | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | X.X | X.X | X.X | X.X | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | X.X | x.x | x.x | X.X |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFR | X.X | X.X | X.X | X.X | X.X | X.X |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (93% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 91 | n | X | X | X | X | X | X |
| | GMT (95% | X.X | X.X | X.X | X.X | X.X | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | X.X | x.x | x.x | X.X | X.X |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> | NA | X.X | x.x | x.x | X.X | X.X |
| | (95% CI) | | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1<br>(N=X) | BA.2.12.1(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 181 | n | x | x | x | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 271 | n | х | х | х | х | х | Х |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| | n | X | X | X | X | X | Х |
| Day 366 | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1<br>(N=X) | BA.2.12.1(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |

n=Number of subjects with results available at time point.

GM=Geometric Mean, GMR<sub>D614G</sub>=Geometric Mean Ratio to D614G variant, GMFR=Geometric Mean Fold Rise, GMFD=Geometric Mean Fold Drop.

Confidence intervals of the GM, GMR, GMFR, and GMFD were calculated with the Student's t distribution on log-transformed data. Confidence intervals of the Seropositive rate were calculated with the Clopper-Pearson method.

# Implementation notes:

Extra variant columns may be added for additional variants.

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

- **Table 232:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Overall– Per Protocol Population
- **Table 233:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort mITT Population
- **Table 234:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- **Table 235:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort mITT Population
- **Table 236:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Cohort Per Protocol Population
- **Table 237:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- **Table 238:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 239: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- **Table 240:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- **Table 241:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population

- Table 242: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 243: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 244: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 245: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 246: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 247: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 248: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 249: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall mITT Population
- **Table 250:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Overall Per Protocol Population
- **Table 251:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort mITT Population
- Table 252: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Table 253: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort mITT Population
- Table 254: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Table 255: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 256: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 257: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Table 258: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 259: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 260: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 261: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 262: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 263: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 264: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 265: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 266: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 267: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall mITT Population
- **Table 268:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- **Table 269:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort mITT Population
- **Table 270:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Cohort Per Protocol Population
- **Table 271:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Table 272: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol Population

- **Table 273:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 274: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- **Table 275:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 276: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 277: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 278: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 279: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 280: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 281: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 282: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 283: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 284: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- **Table 285:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Overall mITT Population
- Table 286: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, Omicron, Overall Per Protocol Population
- **Table 287:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort mITT Population

- Table 288: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- **Table 289:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort mITT Population
- **Table 290:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Cohort Per Protocol Population
- Table 291: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 292: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 293: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 294: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- **Table 295:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 296: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 297: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 298: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 299: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 300: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 301: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 302: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 303: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall mITT Population
- **Table 304:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Overall Per Protocol Population
- **Table 305:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT Population

- **Table 306:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Cohort Per Protocol Population
- Table 307: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort mITT Population
- Table 308: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- **Table 309:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 310: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 311: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 312: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 313: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 314: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 315: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 316: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 317: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 318: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 319: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 320: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 321: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 1 | n | х | х | x | x | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x | X.X | x.x | x.x | X.X |
| | GMR <sub>D614G</sub> (95% CI) | NA NA | (x.x, x.x)<br>x.x<br>(x.x, x.x) | (x.x, x.x)<br>x.x<br>(x.x, x.x) | (x.x, x.x)<br>x.x<br>(x.x, x.x) | (x.x, x.x)<br>x.x<br>(x.x, x.x) | (x.x, x.x)<br>x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 15 | n | х | X | х | х | х | Х |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub><br>(95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 29 | n | X | X | X | X | х | X |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFD<br>(95% CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 57 | n | х | X | х | х | х | Х |
| | GMT (95%<br>CI) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | Median<br>(Min,Max) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | X.X<br>(X.X, X.X) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 71 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 85 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | X.X<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 147 | n | х | X | х | X | Х | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 237 | n | X | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | X.X | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |
| Day 327 | n | Х | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub> (95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive (95% CI) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) | 0.0X<br>(0.xx,0.xx) |
| Day 422 | n | х | X | X | X | X | X |
| | GMT (95% | x.x | x.x | x.x | x.x | x.x | x.x |
| | CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x |
| | (Min,Max) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | GMR <sub>D614G</sub><br>(95% CI) | NA | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) | x.x<br>(x.x, x.x) |
| | GMFR | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |

| Time Point | Statistic | D614G<br>(N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | BA.1 (N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | GMFD | x.x | x.x | x.x | x.x | x.x | x.x |
| | (95% CI) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) | (x.x, x.x) |
| | Seropositive | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X | 0.0X |
| | (95% CI) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) | (0.xx,0.xx) |

n=Number of subjects with results available at time point.

GM=Geometric Mean, GMR<sub>D614G</sub>=Geometric Mean Ratio to D614G variant, GMFR=Geometric Mean Fold Rise, GMFD=Geometric Mean Fold Drop.

Confidence intervals of the GM, GMR, GMFR, and GMFD were calculated with the Student's t distribution on log-transformed data. Confidence intervals of the Seropositive rate were calculated with the Clopper-Pearson method.

## Implementation notes:

Extra variant columns may be added for additional variants.

For tables using the PP population, update footnote to read: "Notes: N=Number of subjects in the Per Protocol population."

Add a note to indicate the lower limit of detection for the assay used to calculate the seropositive rate.

- Table 322: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Overall Per Protocol Population
- Table 323: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort mITT Population
- Table 324: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Table 325: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort mITT Population
- **Table 326:** Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Table 327: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 328: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 329: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Table 330: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 331: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 332: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 333: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 334: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 335: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 336: Focus Reduction Neutralization Test ID50 Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 337: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 338: Focus Reduction Neutralization Test ID<sub>50</sub> Summary Results by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 339: Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Overall – mITT Population

| Study Day | Treatment<br>Group | D614G (N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | B.1.1.529<br>(N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| Day 15 | Beta +<br>Omicron | | | | | | |
| | Delta +<br>Omicron | | | | | | |
| | Omicron | | | | | | |
| | Omicron +<br>Prototype | | | | | | |
| Day 29 | Beta +<br>Omicron | | | | | | |
| | Delta +<br>Omicron | | | | | | |
| | Omicron | | | | | | |
| | Omicron +<br>Prototype | | | | | | |
| Day 91 | Beta +<br>Omicron | | | | | | |
| | Delta +<br>Omicron | | | | | | |
| | Omicron | | | | | | |
| | Omicron +<br>Prototype | | | | | | |
| Day 181 | Beta +<br>Omicron | | | | | | |
| | Delta +<br>Omicron | | | | | | |
| | Omicron | | | | | | |
| | Omicron +<br>Prototype | | | | | | |
| Day 271 | Beta +<br>Omicron | | | | | | |
| | Delta +<br>Omicron | | | | | | |
| | Omicron | | | | | | |
| | Omicron +<br>Prototype | | | | | | |
| Day 366 | Beta +<br>Omicron | | | | | | |
| | Delta +<br>Omicron | | | | | | |
| | Omicron | | | | | | |

| Study Day | Treatment<br>Group | D614G (N=X) | B.1.351<br>(N=X) | B.1.617.2<br>(N=X) | B.1.1.529<br>(N=X) | BA.2.12.1<br>(N=X) | BA.4/BA.5<br>(N=X) |
|---|---|---|---|---|---|---|---|
| | Omicron +<br>Prototype | | | | | | |
| Effect estima<br>an ANCOVA | tes are ratios rela<br>model adjusted | n the mITT Popular<br>tive to the Prototyp<br>for prior infection,<br>A Bonferroni adjus | e treatment grou<br>log <sub>10</sub> of baseline | antibody titers, ago | | | |

- Table 340: Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Overall Per Protocol Population
- Table 341: Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Uninfected (by Self-Report or N-Protein) Cohort mITT Population
- Table 342: Pseudovirus Neutralization Treatment Group Effects as Ratios Relative to the Prototype Arm from ANCOVA model, Uninfected (by Self-Report or N-Protein) Cohort Per Protocol Population

Table 343: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Overall – mITT Population

[Implementation Note: Tables should include rows for median, min, max, GMFR and 95% CI of GMFR. Column order should be Peptide Pool, Cytokine and Time Point.]

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Day 1, Pre-Booster Dose | Beta Mutations | IFNγ | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | IFNγ or IL-2/N | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/TD | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 and<br>154 | n | | | | | | |
| | | 134 | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 or 154 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 or<br>154/C | n | | | | | | |
| | | 134/€ | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 or<br>154/E | n | | | | | | |
| | | 154/E | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 or<br>154/N | n | | | | | | |
| | | 154/IN | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 or<br>154/T | n | | | | | | |
| | | 134/1 | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IL-17a | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IL-4 and 154 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IL-4 IL-5 IL-13 and<br>154 | n | | | | | | |
| | | 134 | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | TNFα | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | Beta S | IFNγ | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | | | | Repeat for all cyto | okines | | | |
| | Conserved S1 | IFNγ | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | | | | Repeat for all cyte | okines | | | |
| | Conserved S2 | IFNγ | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | | | | Repeat for all cyto | okines | | | |
| | Original | IFNγ | n | | | | | | |
| | Matched | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | | | | Repeat for all cyto | okines | | | |
| | Original S | IFNγ | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta<br>+ Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | | • | • | Repeat for all cyto | okines | | • | |

Repeat for all study days

Note: N=Number of Subjects.

n=Number of subjects with results available at time point.

NE=Not Estimable

# Tables with Similar Format:

Table 344: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Overall – Per Protocol Population

Table 345: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Cohort – mITT Population

Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Cohort – Per Protocol Population

Table 347: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Cohort – mITT Population

Table 348: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Cohort – Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

N-protein) Cohort – Per Protocol Population

Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein) **Table 349: Cohort – mITT Population** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein) **Table 350: Cohort – Per Protocol Population Table 351:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) **Cohort – mITT Population Table 352:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) **Cohort – Per Protocol Population Table 353:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Infected (by Self-Report or N-protein) Cohort – mITT Population **Table 354:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or **Table 355:** N-protein) Cohort – mITT Population **Table 356:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population **Table 357:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report or **Table 358:** N-protein) Cohort – Per Protocol Population Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or **Table 359:** N-protein) Cohort – mITT Population Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or **Table 360:** 

Table 361: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall – mITT Population

[Implementation Note: Tables should include rows for median, min, max, GMFR and 95% CI of GMFR. Column order should be Peptide Pool, Cytokine and Time Point.]

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| Day 1, Pre-Booster Dose | Beta Mutations | ΙΕΝγ | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/TD | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 and 154 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 or 154 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 or 154/C | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 or 154/E | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 or 154/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 or 154/T | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IL-17a | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IL-4 and 154 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | IL-4 IL-5 IL-13 and 154 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | TNFα | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | Beta S | ΙΓΝγ | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | Conserved S1 | ΙΕΝγ | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | Conserved S2 | ΙΕΝγ | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | IFNγ or IL-2/CM | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | | | - 1 |
| | Original Matched | IFNγ | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | | , | 1 |
| | Original S | ΙΓΝγ | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |

### Tables with Similar Format:

Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall – Per Protocol Population **Table 362: Table 363:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort – mITT Population Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort – Per Protocol Population **Table 364:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort – mITT Population **Table 365:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort – Per Protocol Population **Table 366: Table 367:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein) **Cohort – mITT Population Table 368:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein) **Cohort – Per Protocol Population** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) **Table 369: Cohort – mITT Population Table 370:** Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) **Cohort – Per Protocol Population** 

- Table 371: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 372: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 373: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 374: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 375: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 376: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 377: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 378: Mean Percentages of CD4 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 379: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Overall – mITT Population

[Implementation Note: Tables should include rows for median, min, max, GMFR and 95% CI of GMFR. Column order should be Peptide Pool, Cytokine and Time Point.]

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Day 1, Pre-Booster Dose | Beta Mutations | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/N | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | IFNγ or IL-2/TD | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | Beta S | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/N | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/TD | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | Conserved S1 | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | IFNγ or IL-2/N | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/TD | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | Conserved S2 | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/N | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/TD | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | Original<br>Matched | IFNγ or IL-2 | n | | | | | | |
| | Matched | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/N | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/TD | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | Original S | IFNγ or IL-2 | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/CM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |

| Time Point | Peptide Pool | Cytokine | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/EM | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/N | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |
| | | IFNγ or IL-2/TD | n | | | | | | |
| | | | Mean | | | | | | |
| | | | 95% CI <sup>a</sup> | | | | | | |
| | | | Response<br>Rate | | | | | | |
| | | | 95% CI <sup>b</sup> | | | | | | |

Repeat for all study days

Note: N=Number of Subjects.

n=Number of subjects with results available at time point.

NE=Not Estimable

<sup>a</sup> Confidence interval calculated based on the Student's t-distribution

<sup>&</sup>lt;sup>b</sup> Exact binomial confidence interval calculated using the Clopper-Pearson methodology.

#### Tables with Similar Format:

- Table 380: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Overall Per Protocol Population
- Table 381: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Cohort mITT Population
- Table 382: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Cohort Per Protocol Population
- Table 383: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Cohort mITT Population
- Table 384: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Cohort Per Protocol Population
- Table 385: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 386: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Infected (by Self-Report or N-protein)
  Cohort Per Protocol Population
- Table 387: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 388: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 389: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 390: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 391: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 392: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 393: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report) Cohort mITT Population
- Table 394: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population

- Table 395: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 396: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 1 Dose Groups, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 397: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall – mITT Population

[Implementation Note: Tables should include rows for median, min, max, GMFR and 95% CI of GMFR. Column order should be Peptide Pool, Cytokine and Time Point.]

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| Day 1, Pre-Booster Dose | Beta Mutations | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/TD | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | Beta S | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/TD | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | | 95% CI <sup>b</sup> | |
| | Conserved S1 | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/TD | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | Conserved S2 | IFNγ or IL-2 | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/TD | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | Original Matched | IFNγ or IL-2 | n | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/TD | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | Original S | IFNy or IL-2 | n | |
| | | | Mean | |

| Time Point | Peptide Pool | Cytokine | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|---|
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/CM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/EM | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/N | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |
| | | IFNγ or IL-2/TD | n | |
| | | | Mean | |
| | | | 95% CI <sup>a</sup> | |
| | | | Response Rate | |
| | | | 95% CI <sup>b</sup> | |

#### Tables with Similar Format:

- Table 398: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Overall Per Protocol Population
- Table 399: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort mITT Population
- Table 400: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Cohort Per Protocol Population
- Table 401: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort mITT Population
- Table 402: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Cohort Per Protocol Population
- Table 403: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein)
  Cohort mITT Population
- Table 404: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Infected (by Self-Report or N-protein)
  Cohort Per Protocol Population
- Table 405: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 406: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 407: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 408: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 409: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 410: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 411: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 412: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population

- Table 413: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 414: Mean Percentages of CD8 T Cells Expressing Cytokines with 95% CI, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 415: Percent of Total B-cells by timepoint and Vaccination arm, Overall – mITT Population

| Probe | Time Point | Statistic | Prototype<br>(N=X) | 1 Dose Beta +<br>Omicron<br>(N=X) | Delta + Omicron<br>(N=X) | Omicron (N=X) | Omicron +<br>Prototype (N=X) | All 1 Dose<br>Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| NTD WT_SA+ | Day 1 | n | XX | xx | xx | XX | XX | XX |
| | | Median (%) | XX.X | xx.x | XX.X | XX.X | xx.x | XX.X |
| | | Min, Max (%) | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| | | n | XX | xx | xx | XX | xx | XX |
| | | Median (%) | XX.X | xx.x | XX.X | XX.X | xx.x | XX.X |
| | | Min, Max (%) | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X |
| | | Median Fold<br>Rise | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Min, Max Fold<br>Rise | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |

Repeat for probes for RBD WT+, RBD WT+ SA+, S2P SA+, S2P WT+, S2P WT+ SA+, Any probe. Include all available time points.

N=number of subjects in group.

n=number of subjects with data available at visit.

## Tables with Similar Format:

- Table 416: Percent of Total B-cells by timepoint and Vaccination arm, Overall Per Protocol Population
- Table 417: Percent of Total B-cells by timepoint and Vaccination arm, Older Cohort mITT Population
- Table 418: Percent of Total B-cells by timepoint and Vaccination arm, Older Cohort Per Protocol Population
- Table 419: Percent of Total B-cells by timepoint and Vaccination arm, Younger Cohort mITT Population
- Table 420: Percent of Total B-cells by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Table 421: Percent of Total B-cells by timepoint and Vaccination arm, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 422: Percent of Total B-cells by timepoint and Vaccination arm, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
N-protein) Cohort – mITT Population

- Percent of Total B-cells by timepoint and Vaccination arm, Uninfected (by Self-Report or N-protein) Cohort mITT Population **Table 423:** Percent of Total B-cells by timepoint and Vaccination arm, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol **Table 424: Population Table 425:** Percent of Total B-cells by timepoint and Vaccination arm, Older Infected (by Self-Report or N-protein) Cohort – mITT Population Percent of Total B-cells by timepoint and Vaccination arm, Older Infected (by Self-Report or **Table 426:** N-protein) Cohort - Per Protocol Population Percent of Total B-cells by timepoint and Vaccination arm, Older Uninfected (by Self-Report or **Table 427:** N-protein) Cohort – mITT Population Percent of Total B-cells by timepoint and Vaccination arm, Older Uninfected (by Self-Report or **Table 428:** N-protein) Cohort – Per Protocol Population Percent of Total B-cells by timepoint and Vaccination arm, Younger Infected (by Self-Report or **Table 429:**
- Table 430: Percent of Total B-cells by timepoint and Vaccination arm, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 431: Percent of Total B-cells by timepoint and Vaccination arm, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 432: Percent of Total B-cells by timepoint and Vaccination arm, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 433: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Overall – mITT Population

| Probe | Time Point | Statistic | 2 Dose Beta + Omicron<br>(N=X) |
|---|---|---|---|
| NTD WT_SA+ | Day 1 | n | xx |
| | | Median (%) | xx.x |
| | | Min, Max (%) | xx.x, xx.x |
| | Day 15 | n | xx |
| | | Median (%) | xx.x |
| | | Min, Max (%) | xx.x, xx.x |
| | | Median Fold Rise | xx.x |
| | | Min, Max Fold Rise | XX.X, XX.X |

Repeat for probes for RBD WT+, RBD WT+ SA+, S2P SA+, S2P WT+, S2P WT+ SA+, Any probe. Include all available time points.

N=number of subjects in group.

n=number of subjects with data available at visit.

#### Tables with Similar Format:

- Table 434: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Overall Per Protocol Population
- Table 435: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Cohort mITT Population
- Table 436: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Cohort Per Protocol Population
- Table 437: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Cohort mITT Population
- Table 438: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Cohort Per Protocol Population
- Table 439: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 440: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 441: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Table 442: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 443: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 444: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 445: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 446: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 447: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Table 448: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Table 449: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Table 450: Percent of Total B-cells by timepoint and Vaccination arm, 2 Dose Group, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

Table 451: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Overall – mITT Population

| | Total Number | Proportion | Proportion | Proportion | Tau <sup>a</sup> | Restricted Mean I | nfection Time (Days) |
|---|---|---|---|---|---|---|---|
| Vaccination Group | Subjects with COVID-19 Infection | Infected at Day 29<br>(95% CI) <sup>b</sup> | Infected at Day 91 (95% CI) <sup>b,c</sup> | Infected at Day<br>181 (95% CI) <sup>b,c</sup> | | Estimate | 95% CI |
| Prototype | X | | | | | X.X | X.X, X.X |
| 1 Dose<br>Beta+Omicron | Х | | | | | x.x | x.x, x.x |
| 2 Dose<br>Beta+Omicron | X | | | | | x.x | x.x, x.x |
| Delta+Omicron | X | | | | | X.X | X.X, X.X |
| Omicron | X | | | | | X.X | X.X, X.X |
| Omicron+Prototype | X | | | | | X.X | X.X, X.X |

N= Number of subjects in the specified vaccination group.

## **Programming Notes:**

### Within a subgroup:

```
proc lifetest data=dat plots=(rmst) method=breslow rmst(cl);
by subgroup;
time infday * Censor(1);
strata trtcode /diff=all;
ods output rmst=rmst;
run;
```

## Tables with Similar Formatting:

- Table 452: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Younger Cohort- mITT Population
- Table 453: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Older Cohort mITT Population
- Table 454: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Infected Cohort (By Self-Report or N-protein) mITT Population

<sup>&</sup>lt;sup>a</sup> Tau is the truncation time point for the Restricted Mean Survival Time analysis and is equal to the minimum of the largest observed times in each group

<sup>&</sup>lt;sup>b</sup>Kaplan-Meier Estimate and 95% confidence interval.

c91/181 days after last vaccination.

- Table 455: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Uninfected Cohort (By Self Report or N-protein) mITT Population
   Table 456: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Younger Infected Cohort (By Self-Report or
- Table 456: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Younger Infected Cohort (By Self-Report or N-protein)— mITT Population
- Table 457: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Younger Uninfected Cohort (By Self-Report or N-protein)—mITT Population
- Table 458: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Older Infected Cohort (By Self-Report or N-protein)—mITT Population
- Table 459: Time to Infection Restricted Mean Survival Analysis by Vaccination Group, Older Uninfected Cohort (By Self-Report or N-protein)—mITT Population

Table 460: Number of Breakthrough Infections by PANGO Call and Treatment Group, Overall – Safety Population

[Implementation Note: Listed variants are examples only, the sequenced variants will be included in the table. Percentages are based on the number of sequenced samples available during the interval.]

| Interval | Variant | Prototype<br>(N=X) | Beta +<br>Omicron<br>(N=X) | Beta + Omicron (Second Dose) (N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Day 1 to Day 8 (n=x) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 9 to Day 15 (n=x) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 16 to Day 29 (n=x) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 30 to Day 91 (n=x) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

| Interval | Variant | Prototype<br>(N=X) | Beta +<br>Omicron<br>(N=X) | Beta + Omicron (Second Dose) (N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 92 to Day 181 (n=x) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 182 to Day 271 (n=x) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Day 272 to Day 366 (n=x) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Any Time Point ( <b>n=x</b> ) | D614G | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Beta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | Delta | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

| Interval | Variant | Prototype<br>(N=X) | Beta +<br>Omicron<br>(N=X) | Beta + Omicron (Second Dose) (N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | BA.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | BA.4/5 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| | XBB.1 | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Note: N=Number of subjects in Safety F | opulation with seq | uencing done. | | | | | | |
| n=number of subjects with reported infe | ctions and sequenc | ing available at | a given visit. | | | | | |

### Tables with Similar Format:

- Table 461: Breakthrough Infections by PANGO Call and Treatment Group, Older Cohort Safety Population
- Table 462: Breakthrough Infections by PANGO Call and Treatment Group, Younger Cohort Safety Population
- Table 463: Breakthrough Infections by PANGO Call and Treatment Group, Infected (by Self-Report or N-protein) Cohort Safety Population
- Table 464: Breakthrough Infections by PANGO Call and Treatment Group, Uninfected (by Self-Report or N-protein) Cohort Safety Population
- Table 465: Breakthrough Infections by PANGO Call and Treatment Group, Older Infected (by Self-Report or N-protein) Cohort Safety Population
- Table 466: Breakthrough Infections by PANGO Call and Treatment Group, Older Uninfected (by Self-Report or N-protein) Cohort Safety Population
- Table 467: Breakthrough Infections by PANGO Call and Treatment Group, Younger Infected (by Self-Report) Cohort Safety Population
- Table 468: Breakthrough Infections by PANGO Call and Treatment Group, Younger Uninfected (by Self-Report or N-protein) Cohort Safety Population

# 14.3 Safety Data

# 14.3.1 Displays of Adverse Events

**Table 469:** Overall Summary of Adverse Events by Treatment Group – All Subjects

| Subjects <sup>a</sup> with | | | otype<br>=X) | | Omicron<br>=X) | (2 D | Omicron<br>loses)<br>=X) | Omi | ta +<br>icron<br>=X) | | icron<br>=X) | Prot | eron +<br>otype<br>=X) | | ıbjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category 1 | Category 2 | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one local solicited adverse event | NA | | | | | | | | | | | | | | |
| At least one systemic solicited adverse event | NA | | | | | | | | | | | | | | |
| At least one unsolicited adverse event | NA | | | | | | | | | | | | | | |
| At least one related<br>unsolicited adverse<br>event | Any Grade | | | | | | | | | | | | | | |
| | Mild (Grade 1) | | | | | | | | | | | | | | |
| | Moderate (Grade 2) | | | | | | | | | | | | | | |
| | Severe (Grade 3) | | | | | | | | | | | | | | |
| At least one severe (Grade 3) unsolicited adverse event | Any relationship | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | |
| | Unrelated | | | | | | | | | | | | | | |
| At least one serious adverse event <sup>b</sup> | Any relationship | | | | | | | | | | | | | | |
| | Related | | | | | | | | | | | | | | |
| | Unrelated | | | | | | | | | | | | | | |

| Subjects <sup>a</sup> with | | Proto<br>(N= | otype<br>=X) | Beta + (N= | Omicron<br>=X) | (2 D | Omicron<br>oses)<br>=X) | Delt<br>Omi<br>(N= | cron | Omi<br>(N= | cron<br>=X) | | eron +<br>otype<br>=X) | All Su<br>(N= | bjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category 1 | Category 2 | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one adverse<br>event leading to early<br>termination <sup>c</sup> | NA | | | | | | | | | | | | | | |
| At least one Adverse<br>Event of Special<br>Interest | NA | | | | | | | | | | | | | | |
| At least one medically attended adverse event | NA | | | | | | | | | | | | | | |
| At least one new onset chronic medical condition | NA | | | | | | | | | | | | | | |

N = Number of subjects in the Safety Population

<sup>a</sup>Subjects are counted once for each category regardless of the number of events.

<sup>b</sup>A listing of Serious Adverse Events is included in Table 483.

<sup>c</sup>As reported on the Adverse Event eCRF.

Table 470: Serious Adverse Events and Non-Serious Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Safety Population

| Preferred Term | MedDRA<br>System Organ<br>Class | | Proto<br>(N= | type<br>X) | Bet | (N= | micron<br>X) | | ta + Oı<br>(2 Dos<br>(N=) | | Delt | ta + Oı<br>(N=X | micron<br>K) | | Omicr<br>(N=X | | | Omicro<br>Protot<br>(N=X | ype | A | All Suk<br>(N=) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Events | | | | | | | | | | | | | | | | | | | | | | |
| All | All | Х | х | X | х | х | X | | | | | | | | | | | | | x | X | X |
| PT1 | SOC1 | х | х | X | Х | х | X | | | | | | | | | | | | | X | X | Х |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | | | | |
| Other (Non-serious) Adv | erse Events | | | | | | | | | | | | | | | | | | | | | |
| All | All | Х | Х | X | X | Х | X | | | | | | | | | | | | | x | X | х |
| PT1 | SOC1 | Х | х | х | Х | х | Х | | | | | | | | | | | | | х | X | Х |
| Etc | Etc | | | | | | | | | | | | | | | | | | | | | |

N = number of subjects in the Safety Population (number of subjects at risk).

n = number of subjects reporting event.

Events = total frequency of events reported.

## 14.3.1.1 Solicited Adverse Events

Table 471: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Post Dose 1

| | | Prote<br>(N: | otype<br>=X) | | Omicron<br>(=X) | | Omicron<br>=X) | | icron<br>=X) | Prot | eron +<br>otype<br>=X) | All St<br>(N | ubjects<br>[=X] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % |
| Any Symptom | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Any Systemic | None | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Fever <sup>a</sup> | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |

| | | Proto<br>(N= | Prototype<br>(N=X) | | Beta + Omicron<br>(N=X) | | Delta + Omicron<br>(N=X) | | icron<br>=X) | Prot | eron +<br>otype<br>=X) | All S<br>(N | ubjects<br>(=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % |
| | Severe | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Any Local Symptom | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | |

| | | Proto<br>(N= | otype<br>=X) | | Omicron<br>=X) | | Omicron<br>=X) | | icron<br>=X) | Prot | eron +<br>otype<br>=X) | All Si<br>(N | ubjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |

Severity is the maximum severity reported over all solicited symptoms post dosing for each subject. N=All subjects receiving vaccination with any solicited event data recorded in the database.

Table 472: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Two Dose Treatment Group

| | | Post I | ron (2 Doses)<br>Dose 2<br>=X) | Beta + Omica<br>Post Eitl<br>(N= | ner Dose |
|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | 0/0 |
| Any Symptom | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Any Systemic Symptom | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Arthralgia | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Fatigue | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Fever <sup>a</sup> | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |

| | | Beta + Omic<br>Post I<br>(N= | Pose 2 | Beta + Omici<br>Post Eith<br>(N= | er Dose |
|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % |
| Feverishness | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Headache | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Myalgia | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Nausea | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Any Local Symptom | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Erythema/Redness | None | | | | |
| | Mild | | | | |

| | | Post I | ron (2 Doses)<br>Dose 2<br>=X) | Post Eit | ron (2 Doses)<br>her Dose<br>=X) |
|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % |
| | Moderate | | | | |
| | Severe | | | | |
| Erythema/Redness | None | | | | |
| Measurement (mm) | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Induration/Swelling | None | | | | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Induration/Swelling | None | | | | |
| Measurement (mm) | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |
| Pain | None | | | _ | |
| | Mild | | | | |
| | Moderate | | | | |
| | Severe | | | | |

Table 473: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Prototype

| | | | -Dose<br>(=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N: | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>(=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N | ny 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N | 7 8+ 1<br>=X) | A<br>Post- | ny<br>Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any<br>Systemic | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |

| | | | Dose<br>=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N: | ny 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N: | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any Local | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| | None | | | | | | | | | | | | | | | | | | | | | | |

| | | | Dose<br>=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N | ay 2<br>=X) | Da<br>(N: | ny 3<br>=X) | | ny 4<br>=X) | Da<br>(N | ıy 5<br>=X) | Da<br>(N | ny 6<br>=X) | | ay 7<br>=X) | Day<br>(N | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose² |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Erythema/Redness | Mild | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |

Notes: N=Number of subjects in the Safety Population.

Severity is the maximum severity reported post dosing for each subject for each day.

1 Day 8+ includes the maximum severity of each symptom reported on or after Day 8 (includes ongoing symptoms)

2 Indicates how many subjects had "None", "Mild", "Moderate", or "Severe" as their maximum severity for any day. A subject may be counted in more than one of these categories.

#### Tables with Similar Format:

Implementation note: For any symptoms or days with missing data, add a "Not Reported" row.

- Table 474: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group Beta + Omicron
- Table 475: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group Delta + Omicron
- Table 476: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group Omicron
- Table 477: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group Omicron + Prototype

Table 478: Summary of Solicited Events by Days Post Treatment, Symptom, and Treatment Group – Beta+Omicron

| | | | -Dose<br>N=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>(=X) | Da<br>(N: | ny 2<br>=X) | Da<br>(N: | ıy 3<br>=X) | Da<br>(N | ay 4<br>(=X) | Da<br>(N: | ıy 5<br>=X) | Da<br>(N: | ıy 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N | 7 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Dose 2 | | | | | | | | | | | | | | | | | | | | | | | |
| Any | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any | None | | | | | | | | | | | | | | | | | | | | | | |
| Systemic<br>Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | | | |

| | | | Dose<br>=X) | | -Dose<br>=X) | D:<br>(N | ay 1<br>=X) | Da<br>(N | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N: | ıy 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N: | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any Local | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |

| | | | -Dose<br>(=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N: | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N | ny 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N: | 7 8+ 1<br>=X) | | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any Dose | | | | | | | | | | | | | | | | | | | | | | | |
| Any | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | 1 | | | | | | | | | | | | | | | | | | | | | |
| | Severe | 1 | | | | | | | | | | | | | | | | | | | | | |
| | None | 1 | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |

| | | | -Dose<br>(=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N: | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N | ny 6<br>=X) | Da<br>(N | ay 7<br>=X) | Day<br>(N: | 8+ 1<br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any<br>Systemic | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Arthralgia | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | | | | | |

| | | | -Dose<br>(=X) | | -Dose<br>=X) | Da<br>(N | ay 1<br>=X) | Da<br>(N: | ny 2<br>=X) | Da<br>(N: | ny 3<br>=X) | Da<br>(N | ay 4<br>=X) | Da<br>(N: | ny 5<br>=X) | Da<br>(N | ıy 6<br>=X) | Da<br>(N | ny 7<br>=X) | Day<br>(N: | 8+ <sup>1</sup><br>=X) | A<br>Post- | ny<br>-Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Any Local | None | | | | | | | | | | | | | | | | | | | | | | |
| Symptom | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Erythema/Redness | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |

| | | | Dose<br>=X) | | -Dose<br>=X) | | ny 1<br>=X) | | ny 2<br>=X) | | ny 3<br>=X) | | ny 4<br>=X) | | ny 5<br>=X) | | ıy 6<br>=X) | | ny 7<br>=X) | Day<br>(N: | 8+ 1<br>=X) | | ny<br>Dose <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Induration/Swelling | None | | | | | | | | | | | | | | | | | | | | | | |
| Measurement (mm) | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |
| Pain | None | | | | | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | | | | | |

Notes: N=Number of subjects in the Safety Population.

Severity is the maximum severity reported post dosing for each subject for each day.

1 Day 8+ includes the maximum severity of each symptom reported on or after Day 8 (includes ongoing symptoms)

<sup>&</sup>lt;sup>2</sup> Indicates how many subjects had "None", "Mild", "Moderate", or "Severe" as their maximum severity for any day. A subject may be counted in more than one of these categories.

 Table 479:
 Summary of Duration of Solicited Symptoms by Treatment Group - All Subjects

| Variable | Statistic | Prototype<br>(N=X) | Beta + Omicron<br>(N=X) | Beta + Omicron<br>(Second Dose)<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Any Symptom | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Any Systemic | n | | | | | | | |
| Symptom | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Arthralgia | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Fatigue | n | | | | | | | |

| Variable | Statistic | Prototype<br>(N=X) | Beta + Omicron<br>(N=X) | Beta + Omicron<br>(Second Dose)<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Fever | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Feverishness | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Headache | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |

| Variable | Statistic | Prototype<br>(N=X) | Beta + Omicron<br>(N=X) | Beta + Omicron<br>(Second Dose)<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Myalgia | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Nausea | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Any Local | n | | | | | | | |
| Symptom | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |

| Variable | Statistic | Prototype<br>(N=X) | Beta + Omicron<br>(N=X) | Beta + Omicron<br>(Second Dose)<br>(N=X) | Delta +<br>Omicron<br>(N=X) | Omicron<br>(N=X) | Omicron +<br>Prototype<br>(N=X) | All Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Erythema/redness | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Induration/swelling | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |
| Pain | n | | | | | | | |
| | Mean | | | | | | | |
| | Standard<br>Deviation | | | | | | | |
| | Median | | | | | | | |
| | Minimum | | | | | | | |
| | Maximum | | | | | | | |

Notes: N=Number of subjects in the Safety Population.

n=Number of solicited adverse events.

## 14.3.1.2 Unsolicited Adverse Events

Table 480: All Adverse Events Cross-Classified by MedDRA System Organ Class, Severity, Relationship to Study Treatment, and Treatment Group

| | | | Rela | ationship to | Vaccination |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| Prototype | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Mild Moderate Severe Severe Mild Moderate Severe Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Beta + Omicron | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Beta + Omicron (Post Second | Any SOC | Mild | | | |
| Dose)<br>(N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Delta + Omicron | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |

| | | | Relationship to Vaccination | | |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Omicron (N=X) | Any SOC | Mild | | | |
| N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| Omicron + Prototype<br>(N=X) | Any SOC | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |
| All Subjects | Any SOC | Mild | | | |
| (N=X) | | Moderate | | | |
| | | Severe | | | |
| | [Repeat for all reported SOC] | Mild | | | |
| | | Moderate | | | |
| | | Severe | | | |

| | | | Rela | Vaccination | |
|---|---|---|---|---|---|
| Treatment Group | MedDRA System Organ Class | Severity | Not Related (n) | Related (n) | Not Yet Determined (n) |
| Notes: N=Number of subjects in the n=Number of events. | Safety Population. | | | | |

Table 481: Summary of All Unsolicited Adverse Events by MedDRA System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group

| | System Organ Class (SOC) | | | Severity | | | Relationship to Study Vaccination | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | | Preferred Term (PT) | Total<br>Events<br>(n) | Mild (n) | Moderate (n) | Severe<br>(n) | Not<br>Related<br>(n) | Related (n) | Not Yet<br>Determined<br>(n) |
| Prototype | Any SOC | Any PT | | | | | | | |
| (N=X) | Gastrointestinal disorders | Any PT | | | | | | | |
| | | Flatulence | | | | | | | |
| | | Vomiting | | | | | | | |
| | [Repeat for all reported | Any PT | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | |
| Beta + Omicron | Any SOC | Any PT | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | |
| Beta + Omicron (Post | Any SOC | Any PT | | | | | | | |
| Second Dose)<br>(N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | |
| , | | [Repeat for all reported PT] | | | | | | | |
| Delta + Omicron | Any SOC | Any PT | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | |
| Omicron | Any SOC | Any PT | | | | | | | |
| (N=X) | | Any PT | | | | | | | |

| | | | | Severity | | | Relationship to Study Vaccination | | |
|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | System Organ Class (SOC) | Preferred Term (PT) | Total<br>Events<br>(n) | Mild<br>(n) | Moderate (n) | Severe (n) | Not<br>Related<br>(n) | Related (n) | Not Yet<br>Determined<br>(n) |
| | [Repeat for all reported SOC] | [Repeat for all reported PT] | | | | | | | |
| Omicron + Prototype | Any SOC | Any PT | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | |
| All Subjects | Any SOC | Any PT | | | | | | | |
| (N=X) | [Repeat for all reported | Any PT | | | | | | | |
| | SOC] | [Repeat for all reported PT] | | | | | | | |

Notes: N=Number of subjects in the Safety Population. n=Number of events.
Table 482: Number and Percentage of Subjects Experiencing Unsolicited Adverse Events by MedDRA® System Organ Class and Preferred Term, Severity, Relationship, and Treatment Group

| | | | | | | | Sev | erity | | | Rel | ationsh<br>Vacci | ip to S<br>nation | tudy |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | A<br>Inci | ny<br>dence | M | Iild | Mod | lerate | Se | vere | | lot<br>ated | Rel | ated |
| Treatment Group | MedDRA System Organ Class | MedDRA Preferred<br>Term | n | % | n | % | n | % | n | % | n | % | n | % |
| Prototype | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |
| Beta + Omicron | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |
| Beta + Omicron (Post | Any SOC | Any PT | | | | | | | | | | | | |
| Second Dose)<br>(N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |
| Delta + Omicron | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |
| Omicron | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |

| | | | | | | | Sev | erity | | | Rel | ationsh<br>Vacci | ip to St<br>nation | tudy |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Aı<br>Incid | | M | lild | Mod | erate | Sev | ere | | lot<br>ated | Rel | ated |
| Treatment Group | MedDRA System Organ Class | MedDRA Preferred<br>Term | n | % | n | % | n | % | n | % | n | % | n | % |
| Omicron + Prototype<br>(N=X) | Any SOC | Any PT | | | | | | | | | | | | |
| | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |
| All Subjects | Any SOC | Any PT | | | | | | | | | | | | |
| (N=X) | [Repeat for all reported SOC] | Any PT | | | | | | | | | | | | |
| | | [Repeat for all reported PT] | | | | | | | | | | | | |

Note: N=Number of subjects in the Safety Population.

n=Number of subjects reporting event with the specified SOC.

This table presents number and percentage of subjects. A subject is only counted once per PT and is summarized according to their highest severity and closest relationship.

# 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

# **Table 483:** Listing of Serious Adverse Events

| Adverse<br>Event | Associated<br>with Dose<br>No. | No. of Days Post Associated Dose (Duration) | No. of Days<br>Post Dose<br>the Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken with Study Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | : , Treatment C | Group: , AE Nu | mber: | | | | | | | | | |
| Comments | • | | | | | | | | | | | |
| Subject ID | : , Treatment C | Group: , AE Nu | mber: | | | | | | | | | |
| Comments | : | | | | | | | | | | | |

#### Table 484: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days<br>Post<br>Associated<br>Dose<br>(Duration) | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Tr | eatment Group: , | AE Number: | | | | | | | | |
| Comments: | | | | | | | | | | |
| Subject ID: , Tr | reatment Group: , | AE Number: | | | | | | | | |
| Comments: | | | | | | | | | | |

#### Table 485: Listing of AESIs, MAAEs and NOCMCs

| Subject ID | Treatment<br>Group | Event<br>Description | Date of Product<br>Administration <sup>a</sup> | Duration of Event | Date of<br>Onset | MedDRA®<br>Sytem Organ<br>Class | MAAEs | NOCMCs | AESI | Relationship <sup>b</sup> | Outcome |
|---|---|---|---|---|---|---|---|---|---|---|---|

# 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

# 14.3.4 Abnormal Laboratory Value Listings (by Subject)

Not Applicable.

# 14.3.5 Displays of Laboratory Results

Not Applicable.

# 14.3.6 Displays of Vital Signs

Not Applicable.

# 14.4 Summary of Concomitant Medications

Table 486: Number and Percentage of Subjects with Prior and Concurrent Medications by WHO Drug Classification and Treatment Group

| WHO<br>Drug<br>Code<br>Level 1,<br>Anatomic<br>Group | WHO Drug<br>Code<br>Level 2,<br>Therapeutic<br>Subgroup | Prototype<br>(N=X) | | Om | Beta +<br>Omicron<br>(N=X) | | nicron omicron (N=X) | | on Omicron | | on (N=X) Prototype | | Omicron +<br>Prototype<br>(N=X) | | Sub | All<br>ojects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | |
| Any Level<br>1 Codes | Any Level 2<br>Codes | X | XX | X | xx | X | XX | X | XX | X | XX | X | xx | х | xx | |
| [ATC<br>Level 1 -<br>1] | Any [ATC 1 – 1] | | | | | | | | | | | | | | | |
| | [ATC 2 - 1] | | | | | | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | | | | | | |
| [ATC<br>Level 1 –<br>2] | [ATC 2 - 1] | | | | | | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | | | | | | |

N = [define the population for this table, e.g., Number of subjects in the Safety Population].

n=Number of subjects reporting taking at least one medication in the specific WHO Drug Class.

# **APPENDIX 2. FIGURE MOCK-UPS**

# LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram | 301 |
|---|---|---|
| Figure 2: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Prototype, Overall – mITT<br>Population | 302 |
| Figure 3: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Prototype, Overall – Per<br>Protocol Population | 303 |
| Figure 4: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Prototype, Younger<br>Cohort – mITT Population | 303 |
| Figure 5: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Prototype, Younger<br>Cohort – Per Protocol Population | 303 |
| Figure 6: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Cohort – mITT Population | 303 |
| Figure 7: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Prototype, Older Cohort –<br>Per Protocol Population | 303 |
| Figure 8: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 303 |
| Figure 9: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 303 |
| Figure 10: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 303 |
| Figure 11: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 303 |
| Figure 12: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 303 |
| Figure 13: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Prototype, Younger<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 303 |

| Figure 14: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 303 |
|---|---|---|
| Figure 15: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 303 |
| Figure 16: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 304 |
| Figure 17: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 304 |
| Figure 18: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 304 |
| Figure 19: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 304 |
| Figure 20: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall – mITT Population | 304 |
| Figure 21: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Overall– Per Protocol Population | 304 |
| Figure 22: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Cohort – mITT Population | 304 |
| Figure 23: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Cohort – Per Protocol Population | 304 |
| Figure 24: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Older Cohort – mITT Population | 304 |
| Figure 25: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Older Cohort – Per Protocol Population | 304 |
| Figure 26: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | |

| Figure 27: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population30 | 04 |
|---|---|---|
| Figure 28: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report) Cohort – mITT Population | 04 |
| Figure 29: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population30 | 05 |
| Figure 30: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population30 | 05 |
| Figure 31: | plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol | 05 |
| Figure 32: | plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – mITT | 05 |
| Figure 33: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 05 |
| Figure 34: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 05 |
| Figure 35: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 05 |
| Figure 36: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population30 | 05 |
| Figure 37: | plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron,<br>Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol | 05 |
| Figure 38: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Geometric Mean by Time Point and Variant, Delta + Omicron, Overall - mITT Population | 05 |

| Figure 39: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron, Overall<br>- Per Protocol Population | 305 |
|---|---|---|
| Figure 40: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron,<br>Younger Cohort – mITT Population | 305 |
| Figure 41: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron,<br>Younger Cohort – Per Protocol Population | 305 |
| Figure 42: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort – mITT Population. | 306 |
| Figure 43: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older<br>Cohort – Per Protocol Population | 306 |
| Figure 44: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron, Infected<br>(by Self-Report or N-protein) Cohort – mITT Population | 306 |
| Figure 45: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron, Infected<br>(by Self-Report or N-protein) Cohort – Per Protocol Population | 306 |
| Figure 46: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron,<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 306 |
| Figure 47: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron,<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 306 |
| Figure 48: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 306 |
| Figure 49: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 306 |
| Figure 50: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 51: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Delta + Omicron, | |

| | Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 306 |
|---|---|---|
| Figure 52: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 306 |
| Figure 53: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 306 |
| Figure 54: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 306 |
| Figure 55: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 307 |
| Figure 56: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron, Overall–mITT<br>Population | 307 |
| Figure 57: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron, Overall – Per<br>Protocol Population | 307 |
| Figure 58: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron, Younger Cohort<br>– mITT Population | 307 |
| Figure 59: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Geometric Mean by Time Point and Variant, Omicron, Younger Cohort — Per Protocol Population | 307 |
| Figure 60: | | |
| Figure 61: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron, Older Cohort –<br>Per Protocol Population | |
| Figure 62: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 63: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |

| Figure 64: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron, Uninfected (by<br>Self-Report or N-protein) Cohort – mITT Population | 307 |
|---|---|---|
| Figure 65: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 307 |
| Figure 66: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 307 |
| Figure 67: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 307 |
| Figure 68: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 307 |
| Figure 69: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 308 |
| Figure 70: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 308 |
| Figure 71: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 308 |
| Figure 72: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 308 |
| Figure 73: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 308 |
| Figure 74: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Overall– mITT Population | 308 |
| Figure 75: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Overall– Per Protocol Population | |
| Figure 76: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Younger Cohort – mITT Population | |

| Figure 77: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Younger Cohort – Per Protocol Population | 308 |
|---|---|---|
| Figure 78: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population | 308 |
| Figure 79: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Older Cohort – Per Protocol Population | 308 |
| Figure 80: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 308 |
| Figure 81: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 308 |
| Figure 82: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 309 |
| Figure 83: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 309 |
| Figure 84: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 309 |
| Figure 85: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 309 |
| Figure 86: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 87: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 309 |
| Figure 88: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 309 |
| Figure 89: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype, | |

| | Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 309 |
|---|---|---|
| Figure 90: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 309 |
| Figure 91: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, Omicron + Prototype,<br>Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 309 |
| Figure 92: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Overall– mITT Population. | 309 |
| Figure 93: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Overall– Per Protocol Population | 309 |
| Figure 94: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Cohort – mITT Population | 309 |
| Figure 95: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Cohort – Per Protocol Population | 310 |
| Figure 96: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Older Cohort – mITT Population | 310 |
| Figure 97: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Older Cohort – Per Protocol Population | 310 |
| Figure 98: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 310 |
| Figure 99: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 310 |
| Figure 100 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 310 |
| Figure 101 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 310 |

| Figure 102: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 310 |
|---|---|---|
| Figure 103: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 310 |
| Figure 104: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – mITT<br>Population | 310 |
| Figure 105: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 310 |
| Figure 106: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 310 |
| Figure 107: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron,<br>Older Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 310 |
| Figure 108: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 311 |
| Figure 109: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 311 |
| Figure 110: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall – mITT Population | 311 |
| Figure 111: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall – Per Protocol Population | 311 |
| Figure 112: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Cohort – mITT Population | 311 |
| Figure 113: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Cohort – Per Protocol Population | 311 |
| Figure 114: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Cohort – mITT Population | 311 |

| Figure 115: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Older Cohort – Per Protocol Population | |
|---|---|
| Figure 116: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – m Population | |
| Figure 117: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 118: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Population | - mITT |
| Figure 119: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Protocol Population | - Per |
| Figure 120: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Younger Infected (by Self-Report or N-protein) ComITT Population | ohort – |
| Figure 121: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Younger Infected (by Self-Report or N-protein) Coper Protocol Population | ohort – |
| Figure 122: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | ) |
| Figure 123: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | ) |
| Figure 124: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Older Infected (by Self-Report or N-protein) CohomITT Population | ort — |
| Figure 125: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Older Infected (by Self-Report or N-protein) Coho Per Protocol Population | ort – |
| Figure 126: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Older Uninfected (by Self-Report or N-protein) ComITT Population | ohort – |
| Figure 127: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Coper Protocol Population | ohort – |
| Figure 128: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Poir Variant 1 Dose Beta + Omicron, Overall - mITT Population | |

| Figure 129: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population | 312 |
|---|---|
| Figure 130: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – mITT Population | 312 |
| Figure 131: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 312 |
| Figure 132: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – mITT Population | 312 |
| Figure 133: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 312 |
| Figure 134: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 312 |
| Figure 135: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 312 |
| Figure 136: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 312 |
| Figure 137: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 312 |
| Figure 138: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 312 |
| Figure 139: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 312 |
| Figure 140: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 312 |
| Figure 141: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 313 |
| Figure 142: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 313 |
| Figure 143: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 313 |

| Figure 144: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 313 |
|---|---|
| Figure 145: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 313 |
| Figure 146: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall– mITT Population | 313 |
| Figure 147: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall – Per Protocol Population | 313 |
| Figure 148: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort – mITT Population | 313 |
| Figure 149: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort – Per Protocol Population | 313 |
| Figure 150: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort – mITT Population | 313 |
| Figure 151: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort – Per Protocol Population | 313 |
| Figure 152: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 313 |
| Figure 153: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 313 |
| Figure 154: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 313 |
| Figure 155: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 313 |
| Figure 156: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 313 |
| Figure 157: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 314 |
| Figure 158: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |

| Figure 159: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 314 |
|---|---|
| Figure 160: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 314 |
| Figure 161: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 314 |
| Figure 162: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 314 |
| Figure 163: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 314 |
| Figure 164: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Overall– mITT Population | 314 |
| Figure 165: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Overall – Per Protocol Population | 314 |
| Figure 166: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Cohort – mITT Population | 314 |
| Figure 167: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Cohort – Per Protocol Population | 314 |
| Figure 168: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort – mITT Population | 314 |
| Figure 169: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort – Per Protocol Population | 314 |
| Figure 170: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 314 |
| Figure 171: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 314 |
| Figure 172: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 314 |
| Figure 173: Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 315 |

| Figure 174: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | .315 |
|---|---|---|
| Figure 175: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .315 |
| Figure 176: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .315 |
| Figure 177: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .315 |
| Figure 178: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | .315 |
| Figure 179: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .315 |
| Figure 180: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .315 |
| Figure 181: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .315 |
| Figure 182: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall – mITT Population | .315 |
| Figure 183: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall – Per Protocol Population | .315 |
| Figure 184: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort – mITT Population | .315 |
| Figure 185: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort – Per Protocol Population | .315 |
| Figure 186: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population | .315 |
| Figure 187: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort – Per Protocol Population | .315 |
| Figure 188: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population. | .315 |

| Figure 189: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 315 |
|---|---|---|
| Figure 190: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 316 |
| Figure 191: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 316 |
| Figure 192: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 316 |
| Figure 193: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 316 |
| Figure 194: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 316 |
| Figure 195: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 316 |
| Figure 196: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 316 |
| Figure 197: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 316 |
| | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 199: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 200: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population | |
| Figure 201: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population | 316 |
| Figure 202: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant. 2 Dose Beta + Omicron, Younger Cohort – mITT Population | 316 |

| Figure 203: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 316 |
|---|---|---|
| Figure 204: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population | 316 |
| Figure 205: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 316 |
| Figure 206: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population. | 317 |
| Figure 207: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 317 |
| Figure 208: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 317 |
| Figure 209: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 317 |
| Figure 210: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 317 |
| Figure 211: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 317 |
| Figure 212: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 317 |
| Figure 213: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 317 |
| Figure 214: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 317 |
| Figure 215: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 317 |
| Figure 216: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 317 |

| Figure 217: | Pseudovirus Neutralization Assay ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 317 |
|---|---|---|
| Figure 218: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall–mITT Population | 317 |
| Figure 219: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall– Per Protocol Population | 318 |
| Figure 220: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Cohort – mITT Population | 318 |
| Figure 221: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Cohort – Per Protocol Population | 318 |
| Figure 222: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Cohort – mITT Population | 318 |
| Figure 223: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Cohort – Per Protocol Population | 318 |
| Figure 224: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 318 |
| Figure 225: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 318 |
| Figure 226: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 318 |
| Figure 227: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 318 |
| Figure 228: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 318 |
| Figure 229: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 318 |
| Figure 230: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 318 |
| Figure 231: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 318 |

| | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 318 |
|---|---|---|
| | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 318 |
| Figure 234: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 318 |
| Figure 235: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 318 |
| Figure 236: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall – mITT Population | 319 |
| Figure 237: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall – Per Protocol Population | 319 |
| Figure 238: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – mITT Population | 319 |
| Figure 239: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 319 |
| Figure 240: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – mITT Population | 319 |
| Figure 241: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 319 |
| Figure 242: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 319 |
| Figure 243: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 244: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 245: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | |

| Figure 246: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 319 |
|---|---|---|
| Figure 247: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 319 |
| Figure 248: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 319 |
| Figure 249: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 319 |
| Figure 250: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 319 |
| Figure 251: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 320 |
| Figure 252: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 320 |
| Figure 253: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 320 |
| Figure 254: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall – mITT Population | 320 |
| Figure 255: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall – Per Protocol Population | 320 |
| Figure 256: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort – mITT Population | 320 |
| Figure 257: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort – Per Protocol Population | 320 |
| Figure 258: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort – mITT Population | 320 |
| Figure 259: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort – Per Protocol Population | 320 |
| Figure 260: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population. | 320 |

| Figure 261: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tin and Variant, Delta + Omicron, Infected (by Self-Report or N-prot – Per Protocol Population | ein) Cohort |
|---|---|
| Figure 262: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tinand Variant, Delta + Omicron, Uninfected (by Self-Report or N-p Cohort – mITT Population | orotein) |
| Figure 263: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tinand Variant, Delta + Omicron, Uninfected (by Self-Report or N-p Cohort – Per Protocol Population | orotein) |
| Figure 264: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tin and Variant, Delta + Omicron, Younger Infected (by Self-Report protein) Cohort – mITT Population | or N- |
| Figure 265: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tinand Variant, Delta + Omicron, Younger Infected (by Self-Report protein) Cohort – Per Protocol Population | or N- |
| Figure 266: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tinand Variant, Delta + Omicron, Younger Uninfected (by Self-Repoprotein) Cohort – mITT Population | ort or N- |
| Figure 267: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tin and Variant, Delta + Omicron, Younger Uninfected (by Self-Repoprotein) Cohort – Per Protocol Population | ort or N- |
| Figure 268: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tinand Variant, Delta + Omicron, Older Infected (by Self-Report or Cohort – mITT Population | N-protein) |
| Figure 269: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tin and Variant, Delta + Omicron, Older Infected (by Self-Report or Cohort – Per Protocol Population | N-protein) |
| Figure 270: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tin and Variant, Delta + Omicron, Older Uninfected (by Self-Report protein) Cohort – mITT Population | or N- |
| Figure 271: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tin and Variant, Delta + Omicron, Older Uninfected (by Self-Report protein) Cohort – Per Protocol Population | or N- |
| Figure 272: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tinand Variant, Omicron, Overall – mITT Population | |
| Figure 273: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tin and Variant, Omicron, Overall – Per Protocol Population | |
| Figure 274: Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Tinand Variant, Omicron, Younger Cohort – mITT Population | |

| Figure 275: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Cohort – Per Protocol Population | 321 |
|---|---|---|
| Figure 276: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort – mITT Population | 321 |
| Figure 277: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort – Per Protocol Population | 321 |
| Figure 278: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 321 |
| Figure 279: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 321 |
| Figure 280: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 321 |
| Figure 281: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 321 |
| Figure 282: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 321 |
| Figure 283: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 322 |
| Figure 284: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 322 |
| Figure 285: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 322 |
| Figure 286: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 322 |
| Figure 287: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 288: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) | 322 |

| Figure 289: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 322 |
|---|---|---|
| Figure 290: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall – mITT Population | 322 |
| Figure 291: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall – Per Protocol Population | 322 |
| Figure 292: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort – mITT Population | 322 |
| Figure 293: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort – Per Protocol Population | 322 |
| Figure 294: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population | 322 |
| Figure 295: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort – Per Protocol Population | 322 |
| Figure 296: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 322 |
| Figure 297: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 322 |
| Figure 298: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 322 |
| Figure 299: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 323 |
| Figure 300: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 323 |
| Figure 301: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 323 |
| Figure 302: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 323 |
| Figure 303: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 323 |

| Figure 304: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 323 |
|---|---|---|
| Figure 305: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 323 |
| Figure 306: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 323 |
| Figure 307: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 323 |
| Figure 308: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population | 323 |
| Figure 309: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population | 323 |
| Figure 310: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population | 323 |
| Figure 311: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 323 |
| Figure 312: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population | 323 |
| Figure 313: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 323 |
| Figure 314: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 324 |
| Figure 315: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 316: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 317: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | |

| Figure 318: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 324 |
|---|---|---|
| Figure 319: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 324 |
| Figure 320: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 324 |
| Figure 321: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 324 |
| Figure 322: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 324 |
| Figure 323: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 324 |
| Figure 324: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 325: | Focus Reduction Neutralization Test ID <sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 324 |
| Figure 326: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Overall – mITT<br>Population | |
| | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Overall – Per<br>Protocol Population | 325 |
| Figure 328: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Younger Cohort –<br>mITT Population | |
| Figure 329: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Younger Cohort –<br>Per Protocol Population | |
| Figure 330: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Older Cohort – mITT Population. | 325 |

| Figure 331 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Older Cohort – Per<br>Protocol Population | 326 |
|---|---|---|
| Figure 332 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Infected (by Self-<br>Report or N-protein) Cohort – mITT Population | 326 |
| Figure 333 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Infected (by Self-<br>Report or N-protein) Cohort – Per Protocol Population | 326 |
| Figure 334 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Uninfected (by Self-<br>Report or N-protein) Cohort – mITT Population | 326 |
| Figure 335 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Uninfected (by Self-<br>Report or N-protein) Cohort – Per Protocol Population | 326 |
| Figure 336 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Younger Infected<br>(by Self-Report or N-protein) Cohort – mITT Population | 326 |
| Figure 337 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Younger Infected<br>(by Self-Report or N-protein) Cohort – Per Protocol Population | 326 |
| Figure 338 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Younger Uninfected<br>(by Self-Report or N-protein) Cohort – mITT Population | 326 |
| Figure 339 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Younger Uninfected<br>(by Self-Report or N-protein) Cohort – Per Protocol Population | 326 |
| Figure 340 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Older Infected (by<br>Self-Report or N-protein) Cohort – mITT Population | 326 |
| Figure 341 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Older Infected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population | 326 |
| Figure 342 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Older Uninfected<br>(by Self-Report or N-protein) Cohort – mITT Population | 326 |
| Figure 343 | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Prototype, Older Uninfected<br>(by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 344: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Overall – mITT Population | 327 |
|---|---|---|
| Figure 345: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Overall– Per Protocol Population | 327 |
| Figure 346: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Cohort – mITT Population. | 327 |
| Figure 347: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Cohort – Per Protocol Population | 327 |
| Figure 348: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older<br>Cohort – mITT Population | 327 |
| Figure 349: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older<br>Cohort – Per Protocol Population | 327 |
| Figure 350: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 327 |
| Figure 351: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 327 |
| Figure 352: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 327 |
| Figure 353: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 327 |
| Figure 354: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 327 |
| Figure 355: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 327 |
| Figure 356: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – mITT<br>Population | 327 |
| | 1 Openanon | ا ہے د |

| Figure 357: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron,<br>Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol<br>Population | 328 |
|---|---|---|
| Figure 358: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 328 |
| Figure 359: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 328 |
| Figure 360: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 328 |
| Figure 361: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 328 |
| Figure 362: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Overall –<br>mITT Population | 328 |
| Figure 363: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Overall – Per<br>Protocol Population | 328 |
| Figure 364: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Younger<br>Cohort – mITT Population | 328 |
| Figure 365: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Younger<br>Cohort – Per Protocol Population | 328 |
| Figure 366: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Older Cohort<br>– mITT Population | 328 |
| Figure 367: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Older Cohort<br>- Per Protocol Population | 328 |
| Figure 368: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Infected (by<br>Self-Report or N-protein) Cohort – mITT Population | 328 |
| Figure 369: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Infected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population | 328 |

| Figure 370: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Uninfected<br>(by Self-Report or N-protein) Cohort – mITT Population | 328 |
|---|---|---|
| Figure 371: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Uninfected<br>(by Self-Report or N-protein) Cohort – Per Protocol Population | 329 |
| Figure 372: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Younger<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 329 |
| Figure 373: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Younger<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 329 |
| Figure 374: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 329 |
| Figure 375: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 329 |
| Figure 376: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Older<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 329 |
| Figure 377: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Older<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 329 |
| Figure 378: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 329 |
| Figure 379: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Delta + Omicron, Older<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 329 |
| Figure 380: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Overall—mITT<br>Population | 329 |
| Figure 381: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Overall – Per<br>Protocol Population | 329 |
| Figure 382: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Younger Cohort –<br>mITT Population | |

| Figure 383: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Younger Cohort –<br>Per Protocol Population | 329 |
|---|---|---|
| Figure 384: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Older Cohort –<br>mITT Population | 329 |
| Figure 385: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Older Cohort – Per<br>Protocol Population | 329 |
| Figure 386: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Infected (by Self-<br>Report or N-protein) Cohort – mITT Population | 330 |
| Figure 387: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Infected (by Self-<br>Report or N-protein) Cohort – Per Protocol Population | 330 |
| Figure 388: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 330 |
| Figure 389: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Uninfected (by Self-<br>Report or N-protein) Cohort – Per Protocol Population | 330 |
| Figure 390: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Younger Infected (by<br>Self-Report or N-protein) Cohort – mITT Population | 330 |
| Figure 391: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 330 |
| Figure 393: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 330 |
| Figure 394: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Older Infected (by<br>Self-Report or N-protein) Cohort – mITT Population | 330 |
| Figure 395: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Older Infected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population | 330 |

| Figure 396: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Older Uninfected (by<br>Self-Report or N-protein) Cohort – mITT Population | 330 |
|---|---|---|
| Figure 397: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron, Older Uninfected (by<br>Self-Report or N-protein) Cohort – Per Protocol Population | 330 |
| Figure 398: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Overall—<br>mITT Population | 330 |
| Figure 399: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Overall–<br>Per Protocol Population | 331 |
| Figure 400: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Younger<br>Cohort – mITT Population | 331 |
| Figure 401: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Younger<br>Cohort – Per Protocol Population | 331 |
| Figure 402: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Older<br>Cohort – mITT Population | 331 |
| Figure 403: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Older<br>Cohort – Per Protocol Population | |
| Figure 404: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Infected<br>(by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 405: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Infected<br>(by Self-Report or N-protein) Cohort – Per Protocol Population | 331 |
| Figure 406: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype,<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 331 |
| Figure 407: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype,<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 331 |
| Figure 408: | : Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Younger<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 331 |

| ] | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Younger<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 331 |
|---|---|---|
| 1 | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 331 |
| 1 | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Younger<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 331 |
| ] | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Older<br>Infected (by Self-Report or N-protein) Cohort – mITT Population | 332 |
| 1 | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Older<br>Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 332 |
| 1 | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Older<br>Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 332 |
| 1 | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, Omicron + Prototype, Older<br>Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 332 |
| ] | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron,<br>Overall– mITT Population | 332 |
| Figure 417: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron,<br>Overall– Per Protocol Population | 332 |
| Figure 418: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Cohort – mITT Population | 332 |
| Figure 419: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron,<br>Younger Cohort – Per Protocol Population | |
| Figure 420: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older<br>Cohort – mITT Population | |
| Figure 421: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population | |

| Figure 422: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-<br>plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron,<br>Infected (by Self-Report or N-protein) Cohort – mITT Population |
|---|---|
| Figure 423: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population332 |
| Figure 424: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population332 |
| Figure 425: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population333 |
| Figure 426: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population333 |
| Figure 427: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population |
| Figure 428: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population |
| Figure 429: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10- plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population |
| Figure 430: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population |
| Figure 431: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population333 |
| Figure 432: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population333 |
| Figure 433: | Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population333 |
| Figure 434: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Overall – mITT Population |

| Figure 435: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Overall – Per Protocol Population | 333 |
|---|---|---|
| Figure 436: | : Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Cohort – mITT Population | 333 |
| Figure 437: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Cohort – Per Protocol Population | 333 |
| Figure 438: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Cohort – mITT Population | 333 |
| Figure 439: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Cohort – Per Protocol Population | 333 |
| Figure 440: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 334 |
| Figure 441: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 334 |
| Figure 442: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 334 |
| Figure 443: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 334 |
| Figure 444: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 334 |
| Figure 445: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 334 |
| Figure 446: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 334 |
| Figure 447: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 334 |
| Figure 448: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 334 |
| Figure 449: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 334 |

| Figure 450: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 334 |
|---|---|
| Figure 451: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 334 |
| Figure 452: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall– mITT Population | 334 |
| Figure 453: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population | 334 |
| Figure 454: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – mITT Population | 334 |
| Figure 455: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 334 |
| Figure 456: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – mITT Population | 334 |
| Figure 457: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 335 |
| Figure 458: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 335 |
| Figure 459: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 335 |
| Figure 460: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 335 |
| Figure 461: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 335 |
| Figure 462: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 335 |
| Figure 463: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 335 |
| Figure 464: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 335 |

| Figure 465: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 335 |
|---|---|
| Figure 466: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 335 |
| Figure 467: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 335 |
| Figure 468: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 335 |
| Figure 469: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 335 |
| Figure 470: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall– mITT Population | 335 |
| Figure 471: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall – Per Protocol Population | 335 |
| Figure 472: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort – mITT Population | 335 |
| Figure 473: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort – Per Protocol Population | 336 |
| Figure 474: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort – mITT Population | 336 |
| Figure 475: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort – Per Protocol Population | 336 |
| Figure 476: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 336 |
| Figure 477: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 336 |
| Figure 478: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 336 |
| Figure 479: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 336 |

| Figure 480: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 336 |
|---|---|---|
| Figure 481: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 336 |
| Figure 482: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 336 |
| Figure 483: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 336 |
| Figure 484: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 336 |
| Figure 485: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 336 |
| Figure 486: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 336 |
| Figure 487: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 336 |
| Figure 488: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall– mITT Population | |
| Figure 489: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall – Per Protocol Population | |
| Figure 490: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort – mITT Population | 336 |
| Figure 491: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort – Per Protocol Population | 337 |
| Figure 492: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort – mITT Population | 337 |
| Figure 493: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort – Per Protocol Population | 337 |
| Figure 494: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 337 |

| Figure 495: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 337 |
|---|---|---|
| Figure 496: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 337 |
| Figure 497: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 337 |
| Figure 498: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population. | 337 |
| Figure 499: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 337 |
| Figure 500: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 337 |
| Figure 501: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 337 |
| Figure 502: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 337 |
| Figure 503: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 337 |
| | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |
| Figure 505: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 506: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall – mITT Population | |
| Figure 507: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall – Per Protocol Population | 337 |
| Figure 508: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort – mITT Population | 337 |

| Figure 509: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort – Per Protocol Population | 338 |
|---|---|---|
| Figure 510: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population | 338 |
| Figure 511: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort – Per Protocol Population | 338 |
| Figure 512: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 338 |
| Figure 513: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 338 |
| Figure 514: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 338 |
| Figure 515: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 338 |
| Figure 516: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 338 |
| Figure 517: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 338 |
| Figure 518: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 338 |
| Figure 519: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 338 |
| Figure 520: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 338 |
| Figure 521: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 522: | Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | |

| Figure 523: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 338 |
|---|---|
| Figure 524: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population | 338 |
| Figure 525: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population | 338 |
| Figure 526: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population | 339 |
| Figure 527: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 339 |
| Figure 528: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population | 339 |
| Figure 529: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 339 |
| Figure 530: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 339 |
| Figure 531: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 339 |
| Figure 532: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 339 |
| Figure 533: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 339 |
| Figure 534: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 339 |
| Figure 535: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 339 |
| Figure 536: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 339 |
| Figure 537: Pseudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 339 |

| Var | rudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and riant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or Ntein) Cohort – mITT Population | 339 |
|---|---|---|
| Var | rudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and riant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or Ntein) Cohort – Per Protocol Population | 339 |
| Var | rudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and riant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or Ntein) Cohort – mITT Population | 339 |
| Var | rudovirus Neutralization Assay ID <sub>50</sub> Distribution by Time Point and riant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or Ntein) Cohort – Per Protocol Population | 339 |
| _ | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Overall– mITT Population | 340 |
| _ | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Overall– Per Protocol Population | 340 |
| _ | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Younger Cohort – mITT Population | 340 |
| _ | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Younger Cohort – Per Protocol Population | 340 |
| _ | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Older Cohort – mITT Population | 340 |
| _ | eus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Older Cohort – Per Protocol Population | 340 |
| Var | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Infected (by Self-Report or N-protein) Cohort – mITT bulation | 340 |
| Var | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Infected (by Self-Report or N-protein) Cohort – Per tocol Population | 340 |
| Var | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT bulation | 340 |
| Var | eus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per tocol Population | 340 |
| Figure 552: Foc<br>Var | cus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and riant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – | 340 |

| • | ID <sub>50</sub> Distribution by Time Point and<br>(by Self-Report or N-protein) Cohort – |
|---|---|
| Figure 554: Focus Reduction Neutralization Test<br>Variant, Prototype, Younger Uninfec<br>Cohort – mITT Population | · |
| Figure 555: Focus Reduction Neutralization Test<br>Variant, Prototype, Younger Uninfect<br>Cohort – Per Protocol Population | · |
| Figure 556: Focus Reduction Neutralization Test<br>Variant, Prototype, Older Infected (b<br>mITT Population | • |
| Figure 557: Focus Reduction Neutralization Test<br>Variant, Prototype, Older Infected (b<br>Per Protocol Population | · |
| | ID <sub>50</sub> Distribution by Time Point and<br>(by Self-Report or N-protein) Cohort – |
| | ID <sub>50</sub> Distribution by Time Point and (by Self-Report or N-protein) Cohort – |
| Figure 560: Focus Reduction Neutralization Test<br>Variant, 1 Dose Beta + Omicron, Ov | ID <sub>50</sub> Distribution by Time Point and erall – mITT Population341 |
| Figure 561: Focus Reduction Neutralization Test<br>Variant, 1 Dose Beta + Omicron, Ov | ID <sub>50</sub> Distribution by Time Point and erall – Per Protocol Population341 |
| Figure 562: Focus Reduction Neutralization Test<br>Variant, 1 Dose Beta + Omicron, Yo | ID <sub>50</sub> Distribution by Time Point and unger Cohort – mITT Population341 |
| Figure 563: Focus Reduction Neutralization Test<br>Variant, 1 Dose Beta + Omicron, Yo | ID <sub>50</sub> Distribution by Time Point and unger Cohort – Per Protocol Population341 |
| Figure 564: Focus Reduction Neutralization Test<br>Variant, 1 Dose Beta + Omicron, Old | ID <sub>50</sub> Distribution by Time Point and ler Cohort – mITT Population341 |
| Figure 565: Focus Reduction Neutralization Test<br>Variant, 1 Dose Beta + Omicron, Old | ID <sub>50</sub> Distribution by Time Point and ler Cohort – Per Protocol Population341 |
| Figure 566: Focus Reduction Neutralization Test Variant, 1 Dose Beta + Omicron, Info Cohort – mITT Population | · |
| Figure 567: Focus Reduction Neutralization Test Variant, 1 Dose Beta + Omicron, Info Cohort - Per Protocol Population | ID <sub>50</sub> Distribution by Time Point and |

| Figure 568: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 341 |
|---|---|
| Figure 569: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 341 |
| Figure 570: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 341 |
| Figure 571: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 341 |
| Figure 572: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 341 |
| Figure 573: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 341 |
| Figure 574: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 341 |
| Figure 575: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 342 |
| Figure 576: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 342 |
| Figure 577: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 342 |
| Figure 578: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall – mITT Population | 342 |
| Figure 579: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall – Per Protocol Population | 342 |
| Figure 580: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort – mITT Population | 342 |
| Figure 581: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort – Per Protocol Population | |
| Figure 582: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort – mITT Population | |

| Figure 583: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort – Per Protocol Population | 342 |
|---|---|
| Figure 584: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 342 |
| Figure 585: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 342 |
| Figure 586: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 342 |
| Figure 587: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 342 |
| Figure 588: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 342 |
| Figure 589: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 342 |
| Figure 590: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 342 |
| Figure 591: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 342 |
| Figure 592: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 343 |
| Figure 593: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 343 |
| Figure 594: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 343 |
| Figure 595: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | |
| Figure 596: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall – mITT Population | |

| Figure 597: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall – Per Protocol Population | .343 |
|---|---|---|
| Figure 598: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort – mITT Population | .343 |
| Figure 599: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort – Per Protocol Population | .343 |
| Figure 600: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort – mITT Population | .343 |
| Figure 601: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort – Per Protocol Population | .343 |
| Figure 602: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | .343 |
| Figure 603: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .343 |
| Figure 604: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .343 |
| Figure 605: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .343 |
| Figure 606: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | .343 |
| Figure 607: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .343 |
| Figure 608: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | .343 |
| Figure 609: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | .344 |
| Figure 610: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | .344 |
| Figure 611: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | .344 |

| Figure 612: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population. | 344 |
|---|---|
| Figure 613: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 344 |
| Figure 614: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall – mITT Population | 344 |
| Figure 615: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall – Per Protocol Population | 344 |
| Figure 616: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort – mITT Population | 344 |
| Figure 617: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort – Per Protocol Population | 344 |
| Figure 618: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population | 344 |
| Figure 619: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort – Per Protocol Population | 344 |
| Figure 620: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population | 344 |
| Figure 621: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 344 |
| Figure 622: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 344 |
| Figure 623: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 344 |
| Figure 624: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 344 |
| Figure 625: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 345 |
| Figure 626: Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 345 |

| Figure 627: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 345 |
|---|---|---|
| Figure 628: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 345 |
| Figure 629: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 345 |
| Figure 630: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 345 |
| Figure 631: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 345 |
| Figure 632: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population | 345 |
| Figure 633: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population | 345 |
| Figure 634: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population | 345 |
| Figure 635: | : Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population | 345 |
| Figure 636: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population | 345 |
| Figure 637: | : Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population | 345 |
| Figure 638: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population | 345 |
| Figure 639: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 345 |
| Figure 640: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 345 |
| Figure 641: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 346 |

| Figure 642: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population | 346 |
|---|---|---|
| Figure 643: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 346 |
| Figure 644: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 346 |
| Figure 645: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 346 |
| Figure 646: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population | 346 |
| Figure 647: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population | 346 |
| Figure 648: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population | 346 |
| Figure 649: | Focus Reduction Neutralization Test ID <sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population | 346 |
| Figure 650: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Overall - mITT Population | 347 |
| Figure 651: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Overall - Per Protocol Population | 347 |
| Figure 652: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Overall - mITT Population | 347 |
| Figure 653: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Overall - Per Protocol Population | 347 |
| Figure 654: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Overall - mITT Population | 347 |
| Figure 655: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Overall - Per Protocol Population | 347 |
| Figure 656: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Overall - mITT Population | 347 |

| Figure 657: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Overall - Per Protocol Population | 347 |
|---|---|---|
| Figure 658: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Overall - mITT Population | 348 |
| Figure 659: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Overall - Per Protocol Population | 348 |
| Figure 660: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Overall - mITT Population | 348 |
| Figure 661: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Overall - Per Protocol Population | 348 |
| Figure 662: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Younger Cohort - mITT Population | 348 |
| Figure 663: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Younger Cohort - Per Protocol Population | 348 |
| Figure 664: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool,<br>Younger Cohort - mITT Population | 348 |
| Figure 665: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool,<br>Younger Cohort - Per Protocol Population | 348 |
| Figure 666: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Younger Cohort - mITT Population | 348 |
| Figure 667: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Younger Cohort - Per Protocol Population | 348 |
| Figure 668: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool,<br>Younger Cohort - mITT Population | 348 |
| Figure 669: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool,<br>Younger Cohort - Per Protocol Population | 348 |
| Figure 670: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Cohort - mITT Population | 348 |
| Figure 671: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Cohort - Per Protocol Population | 348 |
| Figure 672: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Cohort - mITT Population | 348 |
| Figure 673: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Cohort - Per Protocol Population | 348 |
| Figure 674: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Cohort - mITT Population | |
| Figure 675: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Cohort - Per Protocol Population | |

| Figure 676: | : Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Cohort - mITT Population | 348 |
|---|---|---|
| Figure 677: | : Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Cohort - Per Protocol Population | 349 |
| Figure 678: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Cohort - mITT Population | 349 |
| Figure 679: | : Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Cohort - Per Protocol Population | 349 |
| Figure 680: | : Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Cohort - mITT Population | 349 |
| Figure 681: | : Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Cohort - Per Protocol Population | 349 |
| Figure 682: | : Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older<br>Cohort - mITT Population | 349 |
| Figure 683: | : Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Cohort - Per Protocol Population | 349 |
| Figure 684: | : Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Cohort - mITT Population | 349 |
| Figure 685: | : Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Cohort - Per Protocol Population | 349 |
| Figure 686: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - mITT Population | 349 |
| Figure 687: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Infected (by Self-Report and N-protein) Cohort - Per Protocol Population | 349 |
| Figure 688: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - mITT Population | 349 |
| Figure 689: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool,<br>Infected (by Self-Report and N-protein) Cohort - Per Protocol Population | 349 |
| Figure 690: | : Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Infected (by Self-Report and N-protein) Cohort - mITT Population | 349 |
| Figure 691: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Infected (by Self-Report and N-protein) Cohort - Per Protocol Population | 349 |
| Figure 692: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - mITT Population | 349 |
| Figure 693: | : Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - Per Protocol Population | 349 |
| Figure 694: | : Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - mITT Population | |

| _ | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - Per Protocol Population349 |
|---|---|
| _ | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - mITT Population350 |
| _ | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort - Per Protocol Population350 |
| | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - mITT Population350 |
| _ | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population350 |
| _ | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - mITT Population350 |
| _ | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population350 |
| _ | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - mITT Population350 |
| | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population350 |
| _ | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - mITT Population350 |
| _ | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population350 |
| | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - mITT Population350 |
| | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population350 |
| | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - mITT Population350 |
| _ | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool,<br>Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population350 |
| _ | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Younger Infected (by Self-Report and N-protein) Cohort - mITT Population350 |
| | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort - mITT Population350 |

| Figure 713: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort - Per Protocol Population |
|---|---|
| Figure 714: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Younger Infected (by Self-Report and N-protein) Cohort - mITT Population350 |
| Figure 715: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Younger Infected (by Self-Report and N-protein) Cohort - Per Protocol<br>Population |
| Figure 716: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool,<br>Younger Infected (by Self-Report and N-protein) Cohort - mITT Population351 |
| Figure 717: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool,<br>Younger Infected (by Self-Report and N-protein) Cohort - Per Protocol<br>Population |
| Figure 718: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort - mITT Population351 |
| Figure 719: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort - Per Protocol Population351 |
| Figure 720: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort - mITT Population351 |
| Figure 721: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort - Per Protocol Population351 |
| Figure 722: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Older Infected (by Self-Report and N-protein) Cohort - mITT Population351 |
| Figure 723: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - mITT Population351 |
| Figure 725: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| Figure 726: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Older Infected (by Self-Report and N-protein) Cohort - mITT Population351 |
| Figure 727: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| Figure 728: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - mITT Population |

| Figure 729: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - Per Protocol Population | 51 |
|---|---|---|
| Figure 730: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - mITT Population | 51 |
| Figure 731: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - Per Protocol Population3 | 51 |
| Figure 732: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - mITT Population | 51 |
| Figure 733: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort - Per Protocol Population3 | 51 |
| Figure 734: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool,<br>Younger Uninfected (by Self-Report and N-protein) Cohort - mITT<br>Population | 52 |
| Figure 735: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population | 52 |
| Figure 736: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - mITT Population | 52 |
| Figure 737: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population | 52 |
| Figure 738: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - mITT Population | 52 |
| Figure 739: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population | 52 |
| Figure 740: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - mITT Population | 52 |
| Figure 741: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population | 52 |
| Figure 742: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - mITT Population3 | 52 |
| Figure 743: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population3 | 52 |

| Figure 744: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - mITT Population352 |
|---|---|
| Figure 745: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population352 |
| Figure 746: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - mITT Population352 |
| Figure 747: | Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| Figure 748: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool,<br>Older Uninfected (by Self-Report and N-protein) Cohort - mITT Population352 |
| Figure 749: | Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| Figure 750: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool,<br>Older Uninfected (by Self-Report and N-protein) Cohort - mITT Population352 |
| Figure 751: | Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| Figure 752: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool,<br>Older Uninfected (by Self-Report and N-protein) Cohort - mITT Population352 |
| Figure 753: | Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population |
| Figure 754: | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - mITT Population353 |
| | Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population353 |
| Figure 756: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - mITT Population353 |
| Figure 757: | Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort - Per Protocol Population353 |
| Figure 758: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Overall - mITT Population354 |
| Figure 759: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Overall – Per Protocol Population354 |
| Figure 760: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Overall – mITT Population |

| Figure 761 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Overall – Per Protocol Population | 354 |
|---|---|---|
| Figure 762 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Overall – mITT Population | 354 |
| Figure 763 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Overall – Per Protocol Population | 354 |
| Figure 764 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Overall – mITT Population | 354 |
| Figure 765 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Overall – Per Protocol Population | 354 |
| Figure 766 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Overall – mITT Population | 354 |
| Figure 767 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Beta by timepoint and Vaccination arm, Overall – Per Protocol Population | 354 |
| Figure 768 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Overall – mITT Population | 354 |
| Figure 769 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Overall – Per Protocol<br>Population | 355 |
| Figure 770 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Overall – mITT Population | 355 |
| Figure 771 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Overall – Per Protocol Population | 355 |
| Figure 772 | : Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Overall – mITT Population | 355 |
| Figure 773 | : Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Overall – Per Protocol Population | 355 |
| Figure 774 | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Overall – mITT Population | 355 |
| Figure 775 | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Overall – Per Protocol Population | 355 |
| Figure 776 | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Overall – mITT Population | 355 |
| Figure 777 | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Overall – Per Protocol Population | 355 |
| Figure 778 | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm. Overall – mITT Population | 355 |

| Figure 779: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Overall – Per Protocol Population355 |
|---|---|
| Figure 780: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Overall – mITT Population |
| Figure 781: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Overall – Per Protocol Population |
| Figure 782: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Overall – mITT Population |
| Figure 783: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Overall – Per Protocol Population |
| Figure 784: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Overall – mITT Population |
| Figure 785: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Overall – Per Protocol Population355 |
| Figure 786: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Cohort - mITT Population355 |
| Figure 787: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population355 |
| Figure 788: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Cohort – mITT Population356 |
| Figure 789: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population356 |
| Figure 790: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Cohort – mITT Population356 |
| Figure 791: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population |
| Figure 792: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Cohort – mITT Population356 |
| Figure 793: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population |
| Figure 794: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Cohort – mITT Population356 |
| Figure 795: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population. |

| Figure 796: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Younger Cohort – mITT<br>Population | 356 |
|---|---|---|
| Figure 797: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Younger Cohort – Per<br>Protocol Population | 356 |
| Figure 798: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Younger Cohort – mITT<br>Population | 356 |
| Figure 799: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Younger Cohort – Per Protocol<br>Population | 356 |
| Figure 800: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Cohort – mITT Population | 356 |
| Figure 801: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population | 356 |
| Figure 802: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Cohort – mITT Population | 356 |
| Figure 803: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population | 356 |
| Figure 804: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Cohort – mITT Population | 356 |
| Figure 805: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population | 356 |
| Figure 806: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Cohort – mITT Population | 356 |
| Figure 807: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population | 357 |
| Figure 808: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Cohort – mITT Population | 357 |
| Figure 809: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population | 357 |
| Figure 810: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Cohort – mITT Population | 357 |
| Figure 811: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Cohort – Per Protocol Population | 357 |
| Figure 812: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Cohort – mITT Population | 357 |

| _ | istribution of Percent of IgG B-cells expressing RBD Delta-Beta by mepoint and Vaccination arm, Younger Cohort – Per Protocol Population357 |
|---|---|
| | istribution of Percent of IgG B-cells expressing RBD Prototype-Beta by mepoint and Vaccination arm, Older Cohort - mITT Population357 |
| _ | istribution of Percent of IgG B-cells expressing RBD Prototype-Beta by mepoint and Vaccination arm, Older Cohort – Per Protocol Population357 |
| | istribution of Percent of IgG B-cells expressing RBD Prototype-Delta by mepoint and Vaccination arm, Older Cohort – mITT Population357 |
| | istribution of Percent of IgG B-cells expressing RBD Prototype-Delta by mepoint and Vaccination arm, Older Cohort – Per Protocol Population357 |
| _ | istribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta vimepoint and Vaccination arm, Older Cohort – mITT Population357 |
| _ | istribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta timepoint and Vaccination arm, Older Cohort – Per Protocol Population357 |
| _ | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicron timepoint and Vaccination arm, Older Cohort – mITT Population357 |
| | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicron timepoint and Vaccination arm, Older Cohort – Per Protocol Population357 |
| _ | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicroneta by timepoint and Vaccination arm, Older Cohort – mITT Population357 |
| Ве | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicroneta by timepoint and Vaccination arm, Older Cohort – Per Protocol opulation |
| De | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>elta-Beta by timepoint and Vaccination arm, Older Cohort – mITT<br>opulation |
| De | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>elta-Beta by timepoint and Vaccination arm, Older Cohort – Per Protocol<br>opulation |
| _ | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicronelta by timepoint and Vaccination arm, Older Cohort – mITT Population358 |
| De | istribution of Percent of IgG B-cells expressing RBD Prototype-Omicronelta by timepoint and Vaccination arm, Older Cohort – Per Protocol opulation |
| _ | istribution of Percent of IgG B-cells expressing RBD Omicron by mepoint and Vaccination arm, Older Cohort – mITT Population358 |
| _ | istribution of Percent of IgG B-cells expressing RBD Omicron by mepoint and Vaccination arm, Older Cohort – Per Protocol Population358 |

| Figure 830: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Cohort – mITT Population | 358 |
|---|---|---|
| Figure 831: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population | 358 |
| Figure 832: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Cohort – mITT Population | 358 |
| Figure 833: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population | 358 |
| Figure 834: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Cohort – mITT Population | 358 |
| Figure 835: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population | 358 |
| Figure 836: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Cohort – mITT Population | 358 |
| Figure 837: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population | 358 |
| Figure 838: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Cohort – mITT Population | 358 |
| Figure 839: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population | 358 |
| Figure 840: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Cohort – mITT Population | 358 |
| Figure 841: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population | 358 |
| Figure 842: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort - mITT Population | 358 |
| Figure 843: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 358 |
| Figure 844: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 359 |
| Figure 845: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 359 |
| Figure 846: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | |

| Figure 847: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 359 |
|---|---|---|
| Figure 848: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 359 |
| Figure 849: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 359 |
| Figure 850: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 359 |
| Figure 851: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 359 |
| Figure 852: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 359 |
| Figure 853: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 359 |
| Figure 854: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 855: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-<br>protein) Cohort – Per Protocol Population | |
| Figure 856: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 359 |
| Figure 857: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 359 |
| Figure 858: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 859: | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | |

| Figure 860: | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 360 |
|---|---|---|
| Figure 861: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 360 |
| Figure 862: | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 360 |
| Figure 863: | : Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 360 |
| Figure 864: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 360 |
| Figure 865: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 360 |
| Figure 866: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 360 |
| Figure 867: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 360 |
| Figure 868: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – mITT Population | 360 |
| Figure 869: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 360 |
| Figure 870: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort - mITT Population | 360 |
| Figure 871: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 360 |
| Figure 872: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |

| Figure 873: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 360 |
|---|---|---|
| Figure 874: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 361 |
| Figure 875: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 361 |
| Figure 876: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 361 |
| Figure 877: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 361 |
| Figure 878: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 361 |
| Figure 879: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 361 |
| Figure 880: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report<br>and N-protein) Cohort – mITT Population | 361 |
| Figure 881: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report<br>and N-protein) Cohort – Per Protocol Population | |
| Figure 882: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 361 |
| Figure 883: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-<br>protein) Cohort – Per Protocol Population | 361 |
| Figure 884: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 885: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 886: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 361 |
|---|---|---|
| Figure 887: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 361 |
| Figure 888: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 362 |
| Figure 889: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 362 |
| Figure 890: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 362 |
| Figure 891: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 362 |
| Figure 892: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 362 |
| Figure 893: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 362 |
| Figure 894: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 362 |
| Figure 895: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 362 |
| Figure 896: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 897: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 898: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort - mITT Population | |

| Figure 899: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 362 |
|---|---|---|
| Figure 900: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 362 |
| Figure 901: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 362 |
| Figure 902: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 362 |
| Figure 903: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 363 |
| Figure 904 | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 363 |
| Figure 905 | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 363 |
| Figure 906 | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 363 |
| Figure 907: | : Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 363 |
| Figure 908: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 363 |
| Figure 909 | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 363 |
| Figure 910: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 911: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | |

| Figure 912: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 363 |
|---|---|---|
| Figure 913: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 363 |
| Figure 914: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 363 |
| Figure 915: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 363 |
| Figure 916: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 364 |
| Figure 917: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 364 |
| Figure 918: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 364 |
| Figure 919: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 364 |
| Figure 920: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 921: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 364 |
| Figure 922: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | 364 |
| Figure 923: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 924: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – mITT Population | |

| Figure 925: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 364 |
|---|---|---|
| Figure 926: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort - mITT Population | 364 |
| Figure 927: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 364 |
| Figure 928: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 364 |
| Figure 929: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 364 |
| Figure 930: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 365 |
| Figure 931: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 932: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 933: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 365 |
| Figure 935: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 365 |
| Figure 936: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 937: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 365 |

| Figure 938: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 365 |
|---|---|---|
| Figure 939: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 365 |
| Figure 940: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 365 |
| Figure 941: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 365 |
| Figure 942: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 365 |
| Figure 943: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 366 |
| Figure 944: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 366 |
| Figure 945: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 946: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 366 |
| Figure 948: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 366 |
| Figure 949: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 950: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population. | 366 |

| Figure 951: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 366 |
|---|---|---|
| Figure 952: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 366 |
| Figure 953: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 366 |
| Figure 954: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort - mITT Population | 366 |
| Figure 955: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 366 |
| Figure 956: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 366 |
| Figure 957: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 958: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 959: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 367 |
| Figure 961: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 367 |
| Figure 962: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 963: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 367 |

| Figure 964: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 367 |
|---|---|---|
| Figure 965: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-<br>Report and N-protein) Cohort – Per Protocol Population | 367 |
| Figure 966: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 367 |
| Figure 967: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 367 |
| Figure 968: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 367 |
| Figure 969: | Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 367 |
| Figure 970: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 971: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 972: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 368 |
| | Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 368 |
| Figure 974: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 368 |
| Figure 975: | Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 368 |
| Figure 976: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population. | 368 |

| Figure 977: | Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort — Per Protocol Population | 368 |
|---|---|---|
| Figure 978: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 368 |
| Figure 979: | Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 368 |
| Figure 980: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – mITT Population | 368 |
| Figure 981: | Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort – Per Protocol Population | 368 |
| Figure 982: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort - mITT Population | 368 |
| Figure 983: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 368 |
| Figure 984: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 985: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 369 |
| | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 369 |
| Figure 987: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 988: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 989: | Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |

| Figure 990: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 369 |
|---|---|
| Figure 991: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 369 |
| Figure 992: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-<br>Report and N-protein) Cohort – mITT Population | 369 |
| Figure 993: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-<br>Report and N-protein) Cohort – Per Protocol Population | 369 |
| Figure 994: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-<br>Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report<br>and N-protein) Cohort – mITT Population | 369 |
| Figure 995: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 369 |
| Figure 996: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 369 |
| Figure 997: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 369 |
| Figure 998: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | |
| Figure 999: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | |
| Figure 1000: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-<br>Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report<br>and N-protein) Cohort – mITT Population | |
| Figure 1001: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-<br>Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report<br>and N-protein) Cohort – Per Protocol Population | |
| Figure 1002: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | y |

| Figure 1003: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 370 |
|---|---|
| Figure 1004: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 370 |
| Figure 1005: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 370 |
| Figure 1006: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 370 |
| Figure 1007: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 370 |
| Figure 1008: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – mITT Population | 370 |
| Figure 1009: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort – Per Protocol Population | 370 |
| Figure 1010: Time to Infection Kaplan-Meier Curve by Vaccination Group, Overall - mITT Population | 371 |
| Figure 1011: Time to Infection Kaplan-Meier Curve by Vaccination Group, Younger Cohort- mITT Population | 371 |
| Figure 1012: Time to Infection Kaplan-Meier Curve by Vaccination Group, Older Cohort - mITT Population | 371 |
| Figure 1013: Time to Infection Kaplan-Meier Curve by Vaccination Group, Infected Cohort (By Self-report or N-protein)- mITT Population | 371 |
| Figure 1014: Time to Infection Kaplan-Meier Curve by Vaccination Group, Uninfected Cohort (By Self-report or N-protein) - mITT Population | 371 |
| Figure 1015: Time to Infection Kaplan-Meier Curve by Vaccination Group, Younger Infected Cohort (By Self-report or N-protein) - mITT Population | 371 |
| Figure 1016: Time to Infection Kaplan-Meier Curve by Vaccination Group, Younger Uninfected Cohort (By Self-report or N-protein) - mITT Population | 371 |
| Figure 1017: Time to Infection Kaplan-Meier Curve by Vaccination Group, Older Infected Cohort (By Self-report or N-protein) - mITT Population | 372 |
| Figure 1018: Time to Infection Kaplan-Meier Curve by Vaccination Group, Older Uninfected Cohort (By Self-report or N-protein) - mITT Population | 372 |

| Figure 1019: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Prototype – Safety Population | 373 |
|---|---|
| Figure 1020: Summary of Breakthrough Infections by PANGO Call and Treatment Group, 1 Dose Beta + Omicron – Safety Population | 373 |
| Figure 1021: Summary of Breakthrough Infections by PANGO Call and Treatment Group, 2 Dose Beta + Omicron – Safety Population | 373 |
| Figure 1022: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Delta + Omicron – Safety Population | 373 |
| Figure 1023: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Omicron – Safety Population | 373 |
| Figure 1024: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Omicron + Prototype – Safety Population | 373 |
| Figure 1025: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 1 | 374 |
| Figure 1026: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 2 | 374 |
| Figure 1027: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 1 | 375 |
| Figure 1028: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 2 | 375 |
| Figure 1029: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Dose 1 | 376 |
| Figure 1030: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Dose 2 | 377 |
| Figure 1031: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Dose 1 | 377 |
| Figure 1032: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Dose 2 | 377 |
| Figure 1033: Solicited Symptoms by Days Post Vaccination and Treatment Group— Arthralgia | 378 |
| Figure 1034: Solicited Symptoms by Days Post Vaccination and Treatment Group—Chills | 379 |
| Figure 1035: Solicited Symptoms by Days Post Vaccination and Treatment Group— Erythema | 379 |
| Figure 1036: Solicited Symptoms by Days Post Vaccination and Treatment Group— Erythema (mm) | 379 |
| Figure 1037: Solicited Symptoms by Days Post Vaccination and Treatment Group— | 379 |

| _ | Solicited Symptoms by Days Post Vaccination and Treatment Group- | |
|---|---|---|
| Fe | ever | 379 |
| _ | Solicited Symptoms by Days Post Vaccination and Treatment Group—eadache | 379 |
| _ | Solicited Symptoms by Days Post Vaccination and Treatment Group—duration | 379 |
| _ | Solicited Symptoms by Days Post Vaccination and Treatment Group—duration (mm) | 379 |
| _ | Solicited Symptoms by Days Post Vaccination and Treatment Group—yalgia | 379 |
| _ | Solicited Symptoms by Days Post Vaccination and Treatment Group—ausea | 379 |
| _ | Solicited Symptoms by Days Post Vaccination and Treatment Group— | 379 |
| • | Frequency of Adverse Events by MedDRA System Organ Class and everity | 380 |
| | Incidence of Adverse Events by MedDRA® System Organ Class and aximum Severity | 381 |

## 10.1 Disposition of Subjects

Figure 1: CONSORT Flow Diagram



## 14.2.2 Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point

Figure 2: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Overall – mITT Population

[Implementation Note: Below is an example figure. Lines will be shown for each variant. Y-axis label will say Area Under the Curve  $(Log_{10})$ .]



## Figures with Similar Format:

- Figure 3: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Overall Per Protocol Population
- Figure 4: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Figure 5: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Cohort – Per Protocol Population
- Figure 6: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Cohort mITT Population
- Figure 7: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Cohort – Per Protocol Population
- Figure 8: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 9: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 10: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 11: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 12: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 13: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 14: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 15: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 16: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 17: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 18: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 19: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 20: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall mITT Population
- Figure 21: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population
- Figure 22: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort mITT Population
- Figure 23: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort –
  Per Protocol Population
- Figure 24: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort mITT Population
- Figure 25: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population
- Figure 26: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 27: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 28: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report) Cohort mITT Population

- Figure 29: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 30: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 31: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 32: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 33: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 34: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 35: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 36: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected
  (by Self-Report or N-protein) Cohort mITT Population
- Figure 37: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 38: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Overall mITT Population
- Figure 39: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Figure 40: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort – mITT Population
- Figure 41: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort – Per Protocol Population

- Figure 42: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Figure 43: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort – Per Protocol Population
- Figure 44: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 45: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 46: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 47: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 48: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 49: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 50: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 51: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 52: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 53: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 54: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 55: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 56: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Overall–mITT Population
- Figure 57: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Overall Per Protocol Population
- Figure 58: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Cohort mITT Population
- Figure 59: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Cohort – Per Protocol Population
- Figure 60: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Cohort mITT Population
- Figure 61: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Cohort – Per Protocol Population
- Figure 62: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 63: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 64: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 65: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 66: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 67: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 68: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 69: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 70: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 71: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 72: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 73: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 74: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall– mITT Population
- Figure 75: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall- Per Protocol Population
- Figure 76: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort – mITT Population
- Figure 77: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort – Per Protocol Population
- Figure 78: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort – mITT Population
- Figure 79: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort – Per Protocol Population
- Figure 80: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 81: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 82: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 83: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 84: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 85: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 86: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 87: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected
  (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 88: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 89: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 90: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 91: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 92: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall–mITT Population
- Figure 93: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall– Per Protocol Population
- Figure 94: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population

- Figure 95: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population
- Figure 96: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort mITT Population
- Figure 97: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population
- Figure 98: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 99: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 100: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 101: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 102: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 103: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 104: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 105: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 106: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 107: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population

- Figure 108: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 109: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 110: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall mITT Population
- Figure 111: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall Per Protocol Population
- Figure 112: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Figure 113: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- Figure 114: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Cohort mITT Population
- Figure 115: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Cohort Per Protocol Population
- Figure 116: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 117: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 118: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 119: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 120: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 121: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 122: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 123: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 124: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population

- Figure 125: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 126: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 127: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 128: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall– mITT Population
- Figure 129: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population
- Figure 130: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – mITT Population
- Figure 131: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – Per Protocol Population
- Figure 132: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – mITT Population
- Figure 133: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population
- Figure 134: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 135: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 136: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 137: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Figure 138: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 139: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 140: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT
  Population

- Figure 141: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 142: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 143: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 144: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 145: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 146: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall– mITT Population
- Figure 147: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Figure 148: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort mITT Population
- Figure 149: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort Per Protocol Population
- Figure 150: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Figure 151: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol Population
- Figure 152: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 153: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 154: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 155: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 156: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population

- Figure 157: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant,
  Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Figure 158: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 159: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 160: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 161: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 162: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 163: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant,
  Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Figure 164: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Overall–mITT Population
- Figure 165: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Overall Per Protocol Population
- Figure 166: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Cohort mITT Population
- Figure 167: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- Figure 168: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort mITT Population
- Figure 169: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort Per Protocol Population
- Figure 170: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 171: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 172: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 173: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 174: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 175: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 176: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 177: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 178: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 179: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 180: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 181: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 182: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall mITT Population
- Figure 183: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall Per Protocol Population
- Figure 184: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT Population
- Figure 185: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort Per Protocol Population
- Figure 186: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort mITT Population
- Figure 187: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- Figure 188: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 189: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 190: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 191: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 192: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 193: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 194: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 195: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant,
  Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 196: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 197: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 198: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 199: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 200: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT PopulationFigure 201: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population
- Figure 202: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population
- Figure 203: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population
- Figure 204: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population
- Figure 205: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2

- Dose Beta + Omicron, Older Cohort Per Protocol Population
- Figure 206: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 207: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 208: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 209: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Figure 210: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 211: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 212: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 213: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 214: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 215: Pseudovirus Neutralization Assay ID50 Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 216: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 217: Pseudovirus Neutralization Assay ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 218: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall–mITT Population

- Figure 219: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Overall– Per Protocol Population
- Figure 220: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Figure 221: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- Figure 222: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Cohort mITT Population
- Figure 223: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Cohort Per Protocol Population
- Figure 224: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 225: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 226: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 227: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 228: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 229: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 230: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 231: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 232: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 233: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 234: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 235: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 236: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall – mITT Population
- Figure 237: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Overall – Per Protocol Population
- Figure 238: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – mITT Population
- Figure 239: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort – Per Protocol Population
- Figure 240: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – mITT Population
- Figure 241: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort – Per Protocol Population
- Figure 242: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 243: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Figure 244: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 245: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol
  Population
- Figure 246: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 247: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 248: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 249: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 250: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT
  Population

- Figure 251: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1
  Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 252: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 253: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 254: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall mITT Population
- Figure 255: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Figure 256: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort mITT Population
- Figure 257: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Cohort Per Protocol Population
- Figure 258: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Figure 259: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol Population
- Figure 260: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 261: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 262: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 263: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 264: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 265: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 266: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 267: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 268: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 269: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 270: Focus Reduction Neutralization Test ID50 Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 271: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 272: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Overall mITT Population
- Figure 273: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Overall Per Protocol Population
- Figure 274: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Cohort mITT Population
- Figure 275: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- Figure 276: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort mITT Population
- Figure 277: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Cohort Per Protocol Population
- Figure 278: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 279: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 280: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 281: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 282: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population

- Figure 283: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 284: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 285: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 286: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 287: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 288: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 289: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 290: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall mITT Population
- Figure 291: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Overall Per Protocol Population
- Figure 292: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT Population
- Figure 293: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Cohort Per Protocol Population
- Figure 294: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort mITT Population
- Figure 295: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- Figure 296: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 297: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 298: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 299: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 300: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 301: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 302: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 303: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 304: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 305: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 306: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 307: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 308: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – mITT Population
- Figure 309: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Overall – Per Protocol Population
- Figure 310: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – mITT Population
- Figure 311: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort – Per Protocol Population
- Figure 312: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – mITT Population
- Figure 313: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort – Per Protocol Population

- Figure 314: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 315: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 316: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 317: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 318: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 319: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 320: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 321: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 322: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 323: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 324: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2
  Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 325: Focus Reduction Neutralization Test ID<sub>50</sub> Geometric Mean by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
Figure 326: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Overall – mITT Population

[Implementation Note: Below is an example figure. Group boxplots by variant instead of by treatment arm as in the example figure. Y-axis label will say Area Under the Curve (Log<sub>10</sub>). Include lines to connect points between each box plot over time (the lines will connect the points for a subject).]



Figures with Similar Format:

- Figure 327: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Overall Per Protocol Population
- Figure 328: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Figure 329: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- Figure 330: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Older Cohort mITT Population

- Figure 331: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Older Cohort Per Protocol Population
- Figure 332: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 333: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 334: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 335: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 336: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 337: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 338: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 339: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 340: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 341: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 342: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 343: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 344: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall mITT Population
- Figure 345: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population
- Figure 346: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort mITT Population
- Figure 347: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort Per
  Protocol Population
- Figure 348: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort mITT
  Population
- Figure 349: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Figure 350: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 351: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 352: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 353: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 354: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 355: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 356: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 357: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 358: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 359: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 360: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 361: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 362: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Overall mITT Population
- Figure 363: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Figure 364: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort mITT
  Population
- Figure 365: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort Per
  Protocol Population
- Figure 366: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Figure 367: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol
  Population
- Figure 368: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or Nprotein) Cohort mITT Population
- Figure 369: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or Nprotein) Cohort Per Protocol Population
- Figure 370: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 371: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 372: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 373: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 374: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 375: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 376: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 377: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 378: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 379: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 380: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Overall—mITT Population
- Figure 381: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Overall Per Protocol Population
- Figure 382: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Cohort mITT Population
- Figure 383: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- Figure 384: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Older Cohort mITT Population
- Figure 385: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Older Cohort Per Protocol Population

- Figure 386: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein)
  Cohort mITT Population
- Figure 387: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein)
  Cohort Per Protocol Population
- Figure 388: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 389: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 390: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 391: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 392: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 393: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 394: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 395: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 396: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 397: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 398: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Overall–mITT Population

- Figure 399: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Overall– Per Protocol Population
- Figure 400: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT
  Population
- Figure 401: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort Per
  Protocol Population
- Figure 402: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort mITT
  Population
- Figure 403: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- Figure 404: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 405: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 406: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 407: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 408: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 409: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 410: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 411: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 412: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 413: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 414: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 415: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 416: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall–mITT Population
- Figure 417: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall– Per Protocol
  Population
- Figure 418: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort mITT Population
- Figure 419: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort Per
  Protocol Population
- Figure 420: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort mITT Population
- Figure 421: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Figure 422: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 423: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 424: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 425: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 426: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 427: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 428: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 429: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 430: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex
  Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 431: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 432: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 433: Serum IgG Binding Assay Area Under the Curve Measured by ECLIA 10-plex Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 434: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Overall mITT Population
- Figure 435: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Overall Per Protocol Population
- Figure 436: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Figure 437: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- Figure 438: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Cohort mITT Population
- Figure 439: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Cohort Per Protocol Population

- Figure 440: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 441: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 442: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 443: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 444: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 445: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 446: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 447: Pseudovirus Neutralization Assay ID50 Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 448: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 449: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 450: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 451: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 452: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall– mITT Population
- Figure 453: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall– Per Protocol Population
- Figure 454: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort mITT Population
- Figure 455: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Figure 456: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort mITT Population

- Figure 457: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Figure 458: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 459: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 460: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 461: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 462: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 463: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 464: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 465: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 466: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 467: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 468: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 469: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 470: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall– mITT Population
- Figure 471: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Figure 472: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort mITT Population

- Figure 473: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort Per Protocol Population
- Figure 474: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Figure 475: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol Population
- Figure 476: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 477: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 478: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 479: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 480: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 481: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 482: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 483: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 484: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 485: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 486: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 487: Pseudovirus Neutralization Assay ID50 Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 488: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall– mITT Population
- Figure 489: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall Per Protocol Population
- Figure 490: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort mITT Population

- Figure 491: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- Figure 492: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort mITT Population
- Figure 493: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort Per Protocol Population
- Figure 494: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 495: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 496: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 497: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 498: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 499: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 500: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 501: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 502: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 503: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 504: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 505: Pseudovirus Neutralization Assay ID50 Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 506: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall mITT Population
- Figure 507: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall Per Protocol Population
- Figure 508: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT Population

- Figure 509: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort Per Protocol Population
- Figure 510: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort mITT Population
- Figure 511: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- Figure 512: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 513: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 514: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 515: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 516: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 517: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 518: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 519: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 520: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 521: Pseudovirus Neutralization Assay ID50 Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 522: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 523: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 524: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall mITT PopulationFigure 525: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall Per Protocol Population

- Figure 526: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort mITT Population
- Figure 527: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Figure 528: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort mITT Population
- Figure 529: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Figure 530: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 531: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 532: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 533: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 534: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 535: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 536: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 537: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 538: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 539: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 540: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 541: Pseudovirus Neutralization Assay ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 542: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Overall–mITT Population
- Figure 543: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Overall– Per Protocol Population
- Figure 544: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Cohort mITT Population
- Figure 545: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Cohort Per Protocol Population
- Figure 546: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Cohort mITT Population
- Figure 547: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Cohort Per Protocol Population
- Figure 548: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 549: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 550: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 551: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 552: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 553: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 554: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 555: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 556: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 557: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 558: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 559: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 560: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall mITT Population
- Figure 561: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Overall Per Protocol Population
- Figure 562: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort mITT Population
- Figure 563: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Figure 564: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort mITT Population
- Figure 565: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Figure 566: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 567: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 568: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 569: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 570: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 571: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 572: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 573: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 574: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population

- Figure 575: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 576: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 577: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 1 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 578: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall mITT Population
- Figure 579: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Overall Per Protocol Population
- Figure 580: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort mITT Population
- Figure 581: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Cohort Per Protocol Population
- Figure 582: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort mITT Population
- Figure 583: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Cohort Per Protocol Population
- Figure 584: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 585: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 586: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 587: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 588: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 589: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 590: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 591: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population

- Figure 592: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 593: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 594: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 595: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Delta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 596: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall mITT Population
- Figure 597: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Overall Per Protocol Population
- Figure 598: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort mITT Population
- Figure 599: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Cohort Per Protocol Population
- Figure 600: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort mITT Population
- Figure 601: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Cohort Per Protocol Population
- Figure 602: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 603: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 604: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 605: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 606: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 607: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 608: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 609: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 610: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 611: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 612: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 613: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 614: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall mITT Population
- Figure 615: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Overall Per Protocol Population
- Figure 616: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort mITT Population
- Figure 617: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Cohort Per Protocol Population
- Figure 618: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort mITT Population
- Figure 619: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Cohort Per Protocol Population
- Figure 620: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort – mITT Population
- Figure 621: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 622: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 623: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 624: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort – mITT Population

- Figure 625: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant,
  Omicron + Prototype, Younger Infected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 626: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant,
  Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort mITT
  Population
- Figure 627: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Younger Uninfected (by Self-Report or N-protein) Cohort – Per Protocol Population
- Figure 628: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 629: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, Omicron + Prototype, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 630: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 631: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant,
  Omicron + Prototype, Older Uninfected (by Self-Report or N-protein) Cohort Per
  Protocol Population
- Figure 632: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall mITT Population
- Figure 633: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Overall Per Protocol Population
- Figure 634: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort mITT Population
- Figure 635: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Cohort Per Protocol Population
- Figure 636: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort mITT Population
- Figure 637: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Cohort Per Protocol Population
- Figure 638: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 639: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 640: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort mITT Population

- Figure 641: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 642: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 643: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 644: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 645: Focus Reduction Neutralization Test ID50 Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Younger Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 646: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort mITT Population
- Figure 647: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Infected (by Self-Report or N-protein) Cohort Per Protocol Population
- Figure 648: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort mITT Population
- Figure 649: Focus Reduction Neutralization Test ID<sub>50</sub> Distribution by Time Point and Variant, 2 Dose Beta + Omicron, Older Uninfected (by Self-Report or N-protein) Cohort Per Protocol Population



Figure 650: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Overall - mITT Population

## Implementation Note:

Figure shown is an example. Have one plot for each of the 6 treatment arms. Along the x-axis should be each of the study days (Days 1, 15, 91, 181, and 271 for 1 dose treatment arms and Days 1, 15, 57, 71, 147, 237, and 327 for 2 dose treatment arms).

Figures with Similar Format:

- Figure 651: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Overall Per Protocol Population
- Figure 652: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Overall mITT Population
- Figure 653: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Overall Per Protocol Population
- Figure 654: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Overall mITT Population
- Figure 655: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Overall Per Protocol Population
- Figure 656: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Overall mITT Population
- Figure 657: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Overall Per Protocol Population

- Figure 658: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Overall mITT Population
- Figure 659: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Overall Per Protocol Population
- Figure 660: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Overall mITT Population
- Figure 661: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Overall Per Protocol Population
- Figure 662: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Cohort-mITT Population
- Figure 663: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Cohort-Per Protocol Population
- Figure 664: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Cohort mITT Population
- Figure 665: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Cohort Per Protocol Population
- Figure 666: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Cohort mITT Population
- Figure 667: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Cohort Per Protocol Population
- Figure 668: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Cohort-mITT Population
- Figure 669: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Cohort Per Protocol Population
- Figure 670: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Cohort mITT Population
- Figure 671: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Cohort Per Protocol Population
- Figure 672: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Cohort mITT Population
- Figure 673: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Cohort Per Protocol Population
- Figure 674: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Cohort mITT Population
- Figure 675: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Cohort Per Protocol Population
- Figure 676: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Cohort mITT Population

- Figure 677: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Cohort Per Protocol Population
- Figure 678: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Cohort mITT Population
- Figure 679: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Cohort Per Protocol Population
- Figure 680: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Cohort mITT Population
- Figure 681: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Cohort Per Protocol Population
- Figure 682: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Cohort mITT Population
- Figure 683: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Cohort Per Protocol Population
- Figure 684: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Cohort mITT Population
- Figure 685: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Cohort Per Protocol Population
- Figure 686: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 687: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 688: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 689: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 690: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 691: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 692: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 693: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 694: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 695: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Infected (by Self-Report and N-protein) Cohort Per Protocol Population

- Figure 696: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 697: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 698: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 699: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 700: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 701: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 702: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 703: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 704: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 705: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 706: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 707: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 708: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 709: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 710: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 711: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 712: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 713: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 714: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort mITT Population

- Figure 715: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 716: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 717: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 718: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 719: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 720: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 721: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 722: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 723: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 724: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 725: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 726: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 727: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 728: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 729: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 730: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 731: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 732: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 733: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population

- Figure 734: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 735: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 736: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 737: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 738: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 739: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 740: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 741: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 742: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 743: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 744: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 745: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 746: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 747: Percentages of CD4 T Cells Expressing Th1 Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 748: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 749: Percentages of CD4 T Cells Expressing Th2 Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 750: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 751: Percentages of CD4 T Cells Expressing Th1 Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 752: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population

- Figure 753: Percentages of CD4 T Cells Expressing Th2 Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 754: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 755: Percentages of CD8 T Cells Expressing Cytokines S1 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 756: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 757: Percentages of CD8 T Cells Expressing Cytokines S2 Peptide Pool, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population

Figure 758: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Overall - mITT Population



Figures with similar format:

- Figure 759: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 760: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Overall mITT Population
- Figure 761: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 762: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Overall mITT Population
- Figure 763: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 764: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Overall mITT Population
- Figure 765: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 766: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Overall mITT Population
- Figure 767: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 768: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Overall mITT Population

- Figure 769: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 770: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Overall mITT Population
- Figure 771: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 772: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Overall mITT Population
- Figure 773: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 774: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Overall mITT Population
- Figure 775: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 776: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Overall mITT Population
- Figure 777: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 778: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Overall mITT Population
- Figure 779: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 780: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Overall mITT Population
- Figure 781: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 782: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Overall mITT Population
- Figure 783: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 784: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Overall mITT Population
- Figure 785: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Overall Per Protocol Population
- Figure 786: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 787: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population

- Figure 788: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 789: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 790: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 791: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 792: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 793: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 794: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 795: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 796: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 797: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 798: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 799: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 800: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 801: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 802: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 803: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 804: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 805: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 806: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Cohort mITT Population

- Figure 807: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 808: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 809: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 810: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 811: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 812: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Cohort mITT Population
- Figure 813: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Cohort Per Protocol Population
- Figure 814: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Cohort mITT Population
- Figure 815: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Cohort Per Protocol Population
- Figure 816: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Cohort mITT Population
- Figure 817: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Cohort Per Protocol Population
- Figure 818: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Cohort mITT Population
- Figure 819: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Cohort Per Protocol Population
- Figure 820: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Cohort mITT Population
- Figure 821: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Cohort Per Protocol Population
- Figure 822: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Cohort mITT Population
- Figure 823: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Cohort Per Protocol Population
- Figure 824: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Older Cohort mITT Population

**Figure 842:** 

Figure 843:

Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by **Figure 825:** timepoint and Vaccination arm, Older Cohort - Per Protocol Population Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by Figure 826: timepoint and Vaccination arm, Older Cohort – mITT Population Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by **Figure 827:** timepoint and Vaccination arm, Older Cohort - Per Protocol Population Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Figure 828: Vaccination arm, Older Cohort – mITT Population Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Figure 829: Vaccination arm, Older Cohort – Per Protocol Population Figure 830: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Cohort - mITT Population Figure 831: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint **Figure 832:** and Vaccination arm, Older Cohort - mITT Population Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint Figure 833: and Vaccination arm, Older Cohort - Per Protocol Population Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Figure 834: Vaccination arm, Older Cohort – mITT Population **Figure 835:** Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population Figure 836: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Cohort - mITT Population Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination **Figure 837:** arm, Older Cohort - Per Protocol Population Figure 838: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Cohort – mITT Population Figure 839: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Figure 840: Vaccination arm, Older Cohort – mITT Population Figure 841: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Cohort – Per Protocol Population Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and

Vaccination arm, Infected (by Self-Report and N-protein) Cohort - mITT Population

## **Population**

- Figure 844: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 845: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 846: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 847: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 848: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 849: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 850: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 851: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 852: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 853: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 854: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 855: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 856: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 857: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population

- Figure 858: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 859: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 860: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 861: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 862: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 863: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 864: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 865: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 866: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 867: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 868: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 869: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 870: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 871: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 872: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 873: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol
#### **Population**

- Figure 874: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 875: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 876: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 877: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 878: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 879: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 880: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 881: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 882: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 883: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 884: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 885: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 886: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 887: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population

- Figure 888: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 889: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 890: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 891: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 892: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 893: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 894: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 895: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 896: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 897: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 898: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 899: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 900: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 901: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 902: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT

#### **Population**

- Figure 903: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 904: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 905: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 906: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 907: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 908: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 909: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 910: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 911: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 912: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 913: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 914: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 915: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population

- Figure 916: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 917: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 918: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 919: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 920: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 921: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 922: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 923: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 924: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 925: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 926: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 927: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 928: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 929: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population

- Figure 930: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 931: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 932: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 933: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 934: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 935: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 936: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein)

  Cohort mITT Population
- Figure 937: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein)

  Cohort Per Protocol Population
- Figure 938: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 939: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 940: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 941: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 942: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population

- Figure 943: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 944: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 945: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 946: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 947: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 948: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 949: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 950: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 951: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 952: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 953: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Younger Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 954: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 955: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 956: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population

- Figure 957: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 958: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 959: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 960: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 961: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 962: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 963: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 964: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 965: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 966: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 967: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 968: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 969: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 970: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT

#### **Population**

- Figure 971: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 972: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 973: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 974: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 975: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 976: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 977: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 978: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 979: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 980: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort mITT Population
- Figure 981: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Infected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 982: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 983: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 984: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population

- Figure 985: Distribution of Percent of IgG B-cells expressing RBD Prototype-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 986: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 987: Distribution of Percent of IgG B-cells expressing RBD Prototype-Beta-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 988: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 989: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 990: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 991: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 992: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 993: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 994: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 995: Distribution of Percent of IgG B-cells expressing RBD Prototype-Omicron-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 996: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 997: Distribution of Percent of IgG B-cells expressing RBD Omicron by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population

- Figure 998: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 999: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 1000: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 1001: Distribution of Percent of IgG B-cells expressing RBD Omicron-Beta-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 1002: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 1003: Distribution of Percent of IgG B-cells expressing RBD Omicron-Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 1004: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 1005: Distribution of Percent of IgG B-cells expressing RBD Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 1006: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 1007: Distribution of Percent of IgG B-cells expressing RBD Delta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population
- Figure 1008: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort mITT Population
- Figure 1009: Distribution of Percent of IgG B-cells expressing RBD Delta-Beta by timepoint and Vaccination arm, Older Uninfected (by Self-Report and N-protein) Cohort Per Protocol Population



Figure 1010: Time to Infection Kaplan-Meier Curve by Vaccination Group, Overall - mITT Population

Implementation Note: A separate curve will be shown for each vaccination group.

Figures with Similar Format:

- Figure 1011: Time to Infection Kaplan-Meier Curve by Vaccination Group, Younger Cohort- mITT Population
- Figure 1012: Time to Infection Kaplan-Meier Curve by Vaccination Group, Older Cohort mITT Population
- Figure 1013: Time to Infection Kaplan-Meier Curve by Vaccination Group, Infected Cohort (By Self-report or N-protein)- mITT Population
- Figure 1014: Time to Infection Kaplan-Meier Curve by Vaccination Group, Uninfected Cohort (By Self-report or N-protein) mITT Population
- Figure 1015: Time to Infection Kaplan-Meier Curve by Vaccination Group, Younger Infected Cohort (By Self-report or N-protein) mITT Population
- Figure 1016: Time to Infection Kaplan-Meier Curve by Vaccination Group, Younger Uninfected Cohort (By Self-report or N-protein) mITT Population

- Figure 1017: Time to Infection Kaplan-Meier Curve by Vaccination Group, Older Infected Cohort (By Self-report or N-protein) mITT Population
- Figure 1018: Time to Infection Kaplan-Meier Curve by Vaccination Group, Older Uninfected Cohort (By Self-report or N-protein) mITT Population

Figure 1019: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Prototype – Safety Population

[Implementation Note: Figure will be color coded by PANGO Call.]



Figures with Similar Format:

- Figure 1020: Summary of Breakthrough Infections by PANGO Call and Treatment Group, 1 Dose Beta + Omicron Safety Population
- Figure 1021: Summary of Breakthrough Infections by PANGO Call and Treatment Group, 2 Dose Beta + Omicron Safety Population
- Figure 1022: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Delta + Omicron Safety Population
- Figure 1023: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Omicron Safety Population
- Figure 1024: Summary of Breakthrough Infections by PANGO Call and Treatment Group, Omicron + Prototype Safety Population

#### 14.3.1.1 Solicited Adverse Events

Figure 1025: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 1



Figure with Similar Format:

Figure 1026: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 2

Figure 1027: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 1



Figure with Similar Format:

Figure 1028: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Vaccination and Treatment Group – Dose 2

Figure 1029: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Dose 1

[Implementation Note: Have a panel for each treatment group.]



#### Figures with Similar Format:

Figure 1030: Onset of Solicited Systemic Symptoms by Days Post Vaccination and Treatment Group – Dose 2

Figure 1031: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Dose 1

Figure 1032: Onset of Solicited Local Symptoms by Days Post Vaccination and Treatment Group – Dose 2

Figure 1033: Solicited Symptoms by Days Post Vaccination and Treatment Group-Arthralgia



#### Figures with Similar Format:

| Figure 1034: | Calinitad C | rymntome by | Dove I | Doct Va | agination | and Tr | ootmont | Croun | Chille |
|---|---|---|---|---|---|---|---|---|---|
| rigure 1034: | Solicited S | ovindionis dv | v Davs r | OSL VZ | iccination : | anu ii | eaument ' | Group- | CIIIIS |

Figure 1035: Solicited Symptoms by Days Post Vaccination and Treatment Group-Erythema

Figure 1036: Solicited Symptoms by Days Post Vaccination and Treatment Group-Erythema (mm)

Figure 1037: Solicited Symptoms by Days Post Vaccination and Treatment Group-Fatigue

Figure 1038: Solicited Symptoms by Days Post Vaccination and Treatment Group-Fever

Figure 1039: Solicited Symptoms by Days Post Vaccination and Treatment Group-Headache

Figure 1040: Solicited Symptoms by Days Post Vaccination and Treatment Group-Induration

Figure 1041: Solicited Symptoms by Days Post Vaccination and Treatment Group-Induration (mm)

Figure 1042: Solicited Symptoms by Days Post Vaccination and Treatment Group-Myalgia

Figure 1043: Solicited Symptoms by Days Post Vaccination and Treatment Group-Nausea

Figure 1044: Solicited Symptoms by Days Post Vaccination and Treatment Group-Pain

#### 14.3.1.2 Unsolicited Adverse Events

Figure 1045: Frequency of Adverse Events by MedDRA System Organ Class and Severity

[Implementation Note: Have a panel for each treatment group for Dose 1 and a seventh panel for Dose 2.]



Figure 1046: Incidence of Adverse Events by MedDRA® System Organ Class and Maximum Severity

[Implementation Note: Have a panel for each treatment group for Dose 1 and a seventh panel for Dose 2]



# 14.3.5 Displays of Laboratory Results

Not Applicable.

# APPENDIX 3. LISTINGS MOCK-UPS

# LISTINGS

| Listing 1: | 16.1.6: Listing of Subjects Receiving Investigational Product | 385 |
|---|---|---|
| Listing 2: | 16.2.1: Early Terminations or Discontinued Subjects | 386 |
| Listing 3: | 16.2.2.1: Subject-Specific Protocol Deviations | 387 |
| Listing 4: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | 388 |
| Listing 5: | 16.2.3: Subjects Excluded from Analysis Populations | 389 |
| Listing 6: | 16.2.4.1: Demographic Data | 390 |
| Listing 7: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 391 |
| Listing 8: | 16.2.6: Individual Immunogenicity Response Data | 393 |
| Listing 9: | 16.2.6: Individual T-cell Response Data | 393 |
| Listing 10: | 16.2.7.1: Solicited Events – Systemic Symptoms | 395 |
| Listing 11: | 16.2.7.2: Solicited Events – Local Symptoms | 396 |
| Listing 12: | 16.2.7.3: Unsolicited Adverse Events | 397 |
| Listing 13: | 16.2.9.1: Vital Signs | 399 |
| Listing 14: | 16.2.9.2: Physical Exam Findings | 400 |
| Listing 15: | 16.2.10: Concomitant Medications | 401 |
| Listing 16: | 16.2.11.1: Pregnancy Reports – Maternal Information | 402 |
| Listing 17: | 16.2.11.2: Pregnancy Reports – Gravida and Para | 402 |
| Listing 18: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | 403 |
| Listing 19: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | 403 |
| Listing 20: | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 403 |

### Listing 1: 16.1.6: Listing of Subjects Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

### 16.2 Database Listings by Subject

## **16.2.1 Discontinued Subjects**

### **Listing 2:** 16.2.1: Early Terminations or Discontinued Subjects

| Vaccination Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

#### **16.2.2 Protocol Deviations**

## **Listing 3:** 16.2.2.1: Subject-Specific Protocol Deviations

| Vaccination<br>Group | Subject ID | DV Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted<br>in Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

### Listing 4: 16.2.2.2: Non-Subject-Specific Protocol Deviations

| Site | Start Date | Deviation | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.3 Subjects Excluded from the Efficacy Analysis

### **Listing 5:** 16.2.3: Subjects Excluded from Analysis Populations

| Vaccination Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

### 16.2.4 Demographic Data

# Listing 6: 16.2.4.1: Demographic Data

| Vaccination<br>Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race | BMI | Time Between<br>First and<br>Second<br>Booster (Days) | Time Between<br>Covid<br>Infection and<br>Second<br>Booster (Days) | Time Between<br>Covid<br>Infection or<br>First Booster<br>and Second<br>Booster (Days) |
|---|---|---|---|---|---|---|---|---|---|

### Listing 7: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

| Vaccination<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

### 16.2.5 Compliance and/or Drug Concentration Data (if available)

Not Applicable.

#### 16.2.6 Individual Immunogenicity Response Data

Listing 8: 16.2.6: Individual Immunogenicity Response Data

| Vaccination<br>Group | Subject ID | Planned Time Point | Actual Study Day | Assay | Units | Results |
|---|---|---|---|---|---|---|

# **Listing 9:** 16.2.6: Individual T-cell Response Data

| Vaccination<br>Group | Subject ID | Planned Time Point | Actual Study Day | T-Cell | Peptide Pool | Cytokine | Adjusted Percent | Responder (Y/N) |
|---|---|---|---|---|---|---|---|---|

### **Listing 10:** 16.2.6: Individual B-cell Response Data

| Vaccination Group | Subject ID | Planned Time Point | Actual Study Day | Probe | Percent |
|---|---|---|---|---|---|

# Listing 11: 16.2.6: Individual Sequencing Data

| Vaccination Group | Subject ID | Planned Time Point | Actual Study Day | PANGO |
|---|---|---|---|---|

#### 16.2.7 Adverse Events

**Listing 12:** 16.2.7.1: Solicited Events – Systemic Symptoms

| Vaccination<br>Group | Subject ID | Dose Number | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

**Listing 13:** 16.2.7.2: Solicited Events – Local Symptoms

| Treatment Group | Subject ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity |
|---|---|---|---|---|---|---|
| | | | | MA | | |
| | | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

#### Listing 14: 16.2.7.3: Unsolicited Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | <u> </u> | <u> </u> | | <u> </u> | 1 | | <u> </u> | | | <u> </u> | |
| Treatment ( | <br>Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | ı | ı | ı | 1 | 1 | | 1 | 1 | | 1 | |
| Note: For ac | dditional details | about SAEs, se | ee Figure: xx. | | | | | | | | |

# 16.2.8 Individual Laboratory Measurements

Not Applicable.

### 16.2.9 Vital Signs and Physical Exam Findings

Listing 15: 16.2.9.1: Vital Signs

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate (beats/min) | Respiratory Rate (breaths/min) | Weight (kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|---|

### Listing 16: 16.2.9.2: Physical Exam Findings

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|

#### **16.2.10** Concomitant Medications

## **Listing 17: 16.2.10: Concomitant Medications**

| Treatment<br>Group | Subject ID | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an AE?<br>(AE Description;<br>Number) | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.11 Pregnancy Reports

#### **Listing 18:** 16.2.11.1: Pregnancy Reports – Maternal Information

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco,<br>Alcohol, or<br>Drug Use<br>During<br>Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

#### Listing 19: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

#### **Listing 20:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

#### **Listing 21:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

### **Listing 22:** 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|